## Official Title of Study:

A Phase 2, Fast Real-time Assessment of Combination Therapies in Immuno-ONcology Study in Participants With Advanced Gastric Cancer (FRACTION-Gastric Cancer)

PROTOCOL CA018-003

NCT Number: NCT02935634

Document Date (Date in which document was last revised): August 13, 2021

Page: 1

Protocol Number: CA018003 IND Number: 131,283

EUDRACT Number: 2016-002807-24

Date: 12-Aug-2016

Revised Date: 13-Aug-2021

#### **CLINICAL PROTOCOL CA018003**

A Phase 2, <u>Fast Real-time Assessment of Combination Therapies in Immuno-ON</u>cology Study in Participants with Advanced Gastric Cancer (FRACTION-Gastric Cancer)

## Protocol Amendment Number: 06 Incorporates Administrative Letters 03 and 04

Clinical Trial Physician - Medical Monitor Bristol Myers Squibb Company 3401 Princeton Pike Lawrenceville, NJ 08648 Phone email: Clinical Scientist
Bristol Myers Squibb Company
3401 Princeton Pike Lawrenceville, NJ 08648
Phone
email:

24-hr Emergency Telephone Number

USA: International:

### **Bristol-Myers Squibb Research and Development**

Route 206 & Province Line Road Lawrenceville, NJ 08543 Avenue de Finlande 4 B-1420 Braine-l'Alleud, Belgium

This document is the confidential and proprietary information of Bristol-Myers Squibb Company and its global affiliates (BMS). By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis within your organization or to your independent ethics committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (eg, amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to return it to BMS or promptly destroy it. All other rights reserved. References to BMS in this protocol may apply to partners to which BMS has transferred obligations, eg, a Contract Research Organization (CRO).

# **DOCUMENT HISTORY**

| Document | Date of Issue | Summary of Change |
|---|---|---|
| Protocol<br>Amendment 06 | 13-Aug-2021 | Due to early closure of the trial for reasons unrelated to safety, the study schedule was adjusted to remove retreatment/re-randomization options, Response Follow-up, and Survival Follow-up periods for all parts of the study. No changes were made to the Treatment period or Safety Follow-up period. |
| Administrative<br>Letter 04 | 30-Sep-2020 | Updates to staff/contact information for the Medical Monitor |
| Administrative<br>Letter 03 | 12-Dec-2019 | Updates to staff/contact information for the Medical Monitor |
| Revised Protocol<br>05 | 13-Sep-2019 | The nivolumab management algorithms (Appendix 6) were updated to include the myocarditis adverse event management algorithm. Esophagus Cancer Subscale (ECS) from the Functional Assessment of Cancer Therapy-Esophageal (FACT-E) patient-reported outcome assessment was added. Medical Monitor/Study Direction information was updated. |
| Revised Protocol<br>04 | 03-May-2019 | Collection timing and assessment of pretreatment tumor biopsy was clarified. Additional approval information for pembrolizumab was added. Option to utilize a local pathologist for tumor biopsy assessments was removed. Language was updated to indicate that vaccines containing live/attenuated viruses are prohibited. Processing of tumor biopsies was updated. Language describing participants who are imprisoned and Appendix 02 (Study Governance Considerations) were updated to align with the current BMS Protocol Model Document. |
| Administrative<br>Letter 02 | 05-Mar-2019 | Screening biopsy requirement was corrected. |
| Revised Protocol 03 | 05-Feb-2019 | The FRACTION-Gastric Master Protocol was revised to expand indication to esophageal cancer based on the results of CheckMate-032 clinical study. Added clarification on timing and eligibility for efficacy assessment scans at FU1 and FU3. |
| Administrative<br>Letter 01 | 24-Jul-2018 | Change in Medical Monitor Information |
| Revised Protocol<br>02 | 14-Dec-2017 | Revised to allow participants to continue on study treatment for up to 2 years, and re-treatment is not permitted. Stratification by PD-L1 is no longer a factor. Typographical errors were corrected. |
| Revised Protocol | 15-Sep-2016 | Incorporates Amendment 01 |
| Amendment 01 | 15-Sep-2016 | Typographical errors were corrected, and clarifications were made for consistency. |
| Original Protocol | 12-Aug-2016 | Not applicable |

Protocol Amendment No.: 06

## **OVERALL RATIONALE FOR PROTOCOL AMENDMENT 06:**

Due to early closure of the trial for reasons unrelated to safety, the study schedule was adjusted to remove retreatment/re-randomization options, Response Follow-up, and Survival Follow-up periods for all parts of the study. No changes were made to the Treatment period or Safety Follow-up period.

| SUMMARY OF KI | EY CHANGES FOR PROTOCOL AMENDME | NT 06 |
|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Title page | Updated medical monitor and clinical scientist information. | Administrative update. |
| Synopsis | Removed follow-up text from study design. | These changes were made to clarify the removal of the option for treatment beyond progression. |
| Section 2, Schedule of Activities | <ol> <li>Removed Response/Survival Follow-up column in Table 2-3.</li> <li>Footnote "b" in Table 2-3 is no longer applicable as of Protocol Amendment 06.</li> <li>Added text in footnote "c" in Table 2-3 about monitoring safety.</li> </ol> | These changes were made to clarify the removal of the retreatment/re-randomization option, Response Follow-up, and Survival Follow-up periods for the study. |
| Section 3.3,<br>Benefit/Risk<br>Assessment | Added language on the risk assessment of non-live COVID-19 vaccination. | This change was made to address unknown effects of newly available COVID-19 vaccines. |
| Section 5.1.1,<br>FRACTION-Gastric<br>Cancer Tracks 1 and 2<br>Design | <ol> <li>Updated FRACTION-Gastric Cancer Tracks 1 and 2 design follow-up description.</li> <li>Removed Response/Survival Follow-up Phase text from footnote "c" in Figure 5.1.1-1, and marked footnotes "d", "e", and "f" as not applicable as of Protocol Amendment 06.</li> </ol> | These changes were made to clarify the removal of the retreatment/re-randomization option, Response Follow-up, and Survival Follow-up periods for the study. |
| Section 5.1.3, Study<br>Phases | <ol> <li>Updated the number of phases of the study from 4 to 3 phases.</li> <li>Removed Response and Survival Follow up text.</li> <li>Removed reference to subject treatment beyond progression.</li> <li>Added text about discontinuing the collection of biological samples for reasons other than safety monitoring.</li> <li>Added text to allow stopping Survival Follow ups as of Protocol Amendment 06.</li> </ol> | These changes were made to clarify the removal of Response Follow-up, Survival Follow-up periods, and collection of biological samples (nonsafety) for the study. |
| Section 7.4.2,<br>Treatment Beyond<br>Disease Progression | Removed treatment beyond disease progression text and replaced with "Not applicable per Protocol Amendment 06." | These changes were made to clarify the removal of the option for treatment beyond progression. |

Protocol Amendment No.: 06

| SUMMARY OF KEY CHANGES FOR PROTOCOL AMENDMENT 06 | | |
|---|---|---|
| Section Number<br>& Title | Description of Change | Brief Rationale |
| Section 7.7.3, Permitted Therapy | Added text permitting non-live COVID-19 vaccination. | This change was made to adopt the BMS guidance allowing the use of COVID-19 vaccination and clarifying that the safety of such vaccines in study participants receiving investigational agents is unknown. |
| Section 8.1.3, Post<br>Study Treatment<br>Follow-up | Specified that participants will continue to be followed for safety and removed text about Survival Follow up. | These changes were made to clarify the removal of Survival Follow up for the study. |
| Section 9, Study<br>Assessments and<br>Procedures | <ol> <li>Updated text in Section 9.1 to clarify discontinuation of efficacy assessments.</li> <li>Added text in Section 9.5 about discontinuing on-treatment and post-treatment PK sample collection.</li> <li>Added text in Section 9.6 about discontinuing on-treatment and post-treatment pharmacodynamic assessment collection.</li> <li>Added text in Section 9.8 about discontinuing on-treatment and post-treatment biomarker assessment collection.</li> </ol> | These changes were made to clarify the removal of collection of biological samples (nonsafety) for the study. |
| Appendix 2, Study<br>Governance<br>Considerations | <ol> <li>Added text about remote monitoring.</li> <li>Added text on the dissemination of clinical study data.</li> </ol> | <ol> <li>To clarify conditions where remote monitoring can be considered.</li> <li>To clarify disclosure of study data in compliance with national and international standards.</li> </ol> |
| Throughout Document | Updated "subject" terminology to "participant" throughout the document, where applicable. | This update was made to ensure alignment and consistency regarding terminology throughout the document. |

Protocol Amendment No.: 06

Date: 13-Aug-2021 4

# TABLE OF CONTENTS

| TITLE PAGE | |
|----------------------------------------------------------------|-----|
| DOCUMENT HISTORY | ••• |
| OVERALL RATIONALE FOR PROTOCOL AMENDMENT 06: | ••• |
| SUMMARY OF KEY CHANGES FOR PROTOCOL AMENDMENT 06 | |
| TABLE OF CONTENT | ••• |
| 1 SYNOPSIS | |
| 2 SCHEDULE OF ACTIVITIES | |
| 3 INTRODUCTION | |
| 3.1 Study Rationale | ••• |
| 3.1.1 FRACTION Program | |
| 3.1.1.1 Rationale for the FRACTION Program | |
| 3.1.1.2 Specific Attributes of the FRACTION Program Design | |
| 3.1.1.3 Rationale for Biomarker Assessments | |
| 3.2 Background | |
| 3.2.1 FRACTION-Gastric Cancer | |
| 3.3 Benefit/Risk Assessment | |
| 3.3.1 Safety Monitoring on Study Treatment | |
| 4 OBJECTIVES AND ENDPOINTS | |
| 5 STUDY DESIGN | |
| 5.1 Overall Design | |
| 5.1.1 FRACTION-Gastric Cancer Tracks 1 and 2 Design | |
| 5.1.2 Safety Monitoring Board and Other External Committees | |
| 5.1.3 Study Phases | |
| 5.1.3.1 Screening | |
| 5.1.3.2 Treatment | ••• |
| 5.1.3.3 Follow-up | ••• |
| 5.2 Number of Participants | |
| 5.3 End of Study Definition | ••• |
| 5.4 Scientific Rationale for Study Design | |
| 5.4.1 Rationale for Duration of Therapy | |
| 5.5 Justification for Dose | |
| 6 STUDY POPULATION | |
| 6.1 Inclusion Criteria | |
| 6.2 Exclusion Criteria | |
| 6.3 Lifestyle Restrictions | |
| 6.4 Screen Failures | |
| 6.4.1 Retesting During Screening | |
| 7 TREATMENT | ••• |
| 7.1 Treatments Administered | ••• |
| 7.2 Method of Treatment Assignment | |
| 7.3 Blinding | |
| 7.4 Dosage Modification | |
| 7.4.1 Dose Reductions and Delays and Criteria to Resume Dosing | |
| 7.4.2 Treatment Beyond Disease Progression | |

Protocol Amendment No.: 06 Date: 13-Aug-2021

| 7.4.3 Management Algorithms for IO and Oncology Agents | 49 |
|---|---|
| 7.4.4 Treatment of Treatment-related Infusion Reactions | |
| 7.5 Preparation/Handling/Storage/Accountability | |
| 7.5.1 Retained Samples for Bioavailability / Bioequivalence / Biocomparabil | |
| 7.3.1 Retained Samples for Bioavailability / Bioequivalence / Biocomparabil | 50 |
| 7.6 Treatment Compliance | |
| 7.7 Concomitant Therapy | _ |
| 7.7.1 Prohibited and/or Restricted Treatments | |
| 7.7.2 Other Restrictions and Precautions | |
| 7.7.2.1 Imaging Restriction and Precautions | |
| 7.7.3 Permitted Therapy | |
| 7.7.4 Palliative Local Therapy | 52 |
| 7.7.5 Supportive Care Management | |
| 7.8 Treatment After the End of the Study | |
| 8 DISCONTINUATION CRITERIA | |
| 8.1 Discontinuation from Study Treatment | |
| 8.1.1 Permanent Discontinuation | |
| 8.1.2 Study Treatment Combination Arm Discontinuation Criteria | _ |
| 8.1.3 Post Study Treatment Study Follow-up | |
| 8.2 Discontinuation from the Study | |
| 8.3 Lost to Follow-up | |
| 9 STUDY ASSESSMENTS AND PROCEDURES. | |
| 9.1 Efficacy Assessments | |
| 9.1.1 Imaging Assessment for the Study | 11 |
| 9.2 Adverse Events | |
| 9.2.1 Time Period and Frequency for Collecting AE and SAE Information | |
| 9.2.2 Method of Detecting AEs and SAEs | |
| 9.2.3 Follow-up of AEs and SAEs | |
| 9.2.4 Regulatory Reporting Requirements for SAEs | |
| 9.2.5 Pregnancy | |
| 9.2.6 Laboratory Test Result Abnormalities | |
| 9.2.7 Potential Drug Induced Liver Injury | |
| 9.2.8 Other Safety Considerations | 62 |
| 9.3 Overdose | 62 |
| 9.4 Safety | 62 |
| 9.4.1 Clinical Safety Laboratory Assessments | |
| 9.4.2 Imaging Safety Assessment | 64 |
| 9.5 Pharmacokinetic | 64 |
| 9.6 Pharmacodynamics | 64 |
| 9.7 Pharmacogenomics | |
| 9.8 Biomarkers | 64 |

7

| 9.8.5 Immunogenicity Assessments |
|-------------------------------------------------------------------------|
| 9.0.3 Immunogenicity Assessments |
| 9.8.10 Other Assessments |
| 9.9 Medical Resource Utilization and Health Economics |
| 9.9.1 Patient-reported Outcomes |
| 10 STATISTICAL CONSIDERATIONS |
| 10.1 Sample Size Determination |
| 10.1.1 Track 1 - Anti-PD-1, Anti-PD-L1, and Anti-CTLA-4 Treatment-naïve |
| Participants |
| 10.1.2 Track 2 - Anti-PD-1, Anti-PD-L1, or Anti-CTLA-4 Treatment- |
| experienced Participants |
| 10.2 Populations for Analyses |
| 10.3 Statistical Analyses |
| 10.3.1 Efficacy Analyses |
| 10.3.2 Safety Analyses |
| 10.3.3 Other Analyses |
| 10.3.3.1 Pharmacokinetic Analyses |
| 10.3.3.2 Immunogenicity Analyses |
| 10.3.3.3 Exploratory Biomarker Analyses |
| 10.3.3.4 Outcomes Research Analyses |
| 10.5.4 Intertin Analyses |
| 12 APPENDICES |
| APPENDIX 1 ABBREVIATIONS AND TRADEMARKS |
| APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS |
| APPENDIX 3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: |
| DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, |
| FOLLOW UP AND REPORTING |
| APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND |
| METHODS OF CONTRACEPTION |
| APPENDIX 5 RECIST V1.1 |
| APPENDIX 6 NIVOLUMAB MANAGEMENT ALGORITHMS |
| APPENDIX 7 ECOG PERFORMANCE STATUS |
| APPENDIX 8 COUNTRY SPECIFIC REQUIREMENTS |

APPENDIX 9 REVISED PROTOCOL SUMMARY OF CHANGE HISTORY .......

129

8

Protocol Amendment No.: 06 Date: 13-Aug-2021

#### 1 SYNOPSIS

**Protocol Title:** A Phase 2, <u>Fast Real-time Assessment of Combination Therapies in Immuno-ON</u>cology Study in Participants with Advanced Gastric Cancer (FRACTION-Gastric Cancer)

Study Phase: Phase 2

#### **Rationale:**

To determine which combinations show the most clinical promise and thus should be prioritized for registrational studies; Bristol-Myers Squibb Company (BMS) has initiated the Fast Real-time Assessment of Combination Therapy in Immuno-ONcology (FRACTION) Program (globally listed under the descriptor BMS-986217). The FRACTION Program will employ repeat core biopsies and serial assessments with different treatment options. Novel study treatment combinations and/or additional controls will be appended as FRACTION-Gastric Cancer Sub-Protocols. These FRACTION-Gastric Cancer Sub-Protocols will evaluate the safety profile, tolerability, preliminary efficacy, pharmacokinetic (PK), and pharmacodynamics of novel study treatment combinations in participants with advanced gastric cancer (GC).

### **Study Population:**

Male and female participants, aged 18 years and older, with inoperable, advanced, or metastatic esophageal cancer (EC), gastric cancer (GC) or gastroesophageal junction (GEJ) carcinoma and have histologically confirmed predominant adenocarcinoma and/or squamous carcinoma, may be eligible for the study. The documentation of GEJ involvement can include biopsy, endoscopy, or imaging.

Track-specific eligibility criteria are as follows:

- Track 1: anti-programmed death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), and anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) treatment-naïve participants
  - Participants must not have received any anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment prior to this study. Participants previously treated with agents other than anti-PD-1, anti-PD-L1, or anti-CTLA-4 are eligible for Track 1.
  - Participants may have been offered platinum-based chemotherapy for progressive or recurrent disease.
    - ♦ The platinum-based chemotherapy may have been in the adjuvant, neoadjuvant, or recurrent setting.
  - Participants will be required to submit a fresh tumor biopsy.
- Track 2: anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment-experienced participants
  - Participants must have had progressive or recurrent disease during or after anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment. (Participants treated with any study treatment targeting PD-1, PD-L1, or CTLA-4 will be considered anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment experienced, respectively.)

- Participants may have been offered platinum-based chemotherapy for progressive or recurrent disease.
  - ♦ The platinum-based chemotherapy may have been in the adjuvant, neoadjuvant, or recurrent setting.
- Participants who have had prior treatment with any 1 of the agents (or any other agent targeting PD-1, PD-L1, or CTLA-4) in monotherapy or in any combination regimen in a FRACTION-Gastric Cancer Sub-Protocol are eligible for treatment on Track 2.
- Participants who have had prior combination treatment with the same immuno-oncology (IO) combination agents (or IO agents directed against the same targets) as 1 of the combination regimens in a FRACTION-Gastric Cancer Sub-Protocol are eligible for study treatment on Track 2 but must be randomized to another combination regimen.
- Participants will be required to submit a fresh tumor biopsy.

## **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the efficacy (ORR, DOR, and PFSR at 24 weeks) of each FRACTION-Gastric Cancer study treatment combination (relative to nivolumab in combination with ipilimumab, when applicable) in participants with advanced GC and/or EC | ORR defined as the proportion of all treated participants with a BOR of CR or PR as assessed per RECIST v1.1 by investigator, median DOR, and PFSR at 24 weeks |
| Secondary | |
| To investigate additional safety and tolerability of each<br>FRACTION-Gastric Cancer study treatment combination<br>in participants with advanced GC and/or EC | Incidence of AEs, SAEs, AEs leading to<br>discontinuation, deaths, and clinical<br>laboratory test abnormalities |
| Tertiary/Exploratory | |
| To assess the pharmacodynamic effects as a function of exposure, by evaluation of select biomarkers | Summary measures of change (or % change) from baseline or baseline level biomarker measurements |
| To explore potential associations between anti-tumor activity or safety and select biomarker measures | Correlation (or similar appropriate measure of association) of biomarker measure with |
| To evaluate the PK of each IP component | parameters of interest |
| • To evaluate the immunogenicity of each IP, when applicable | Summary measures of PK parameters from serum concentration |
| To assess the OS in treated participants | Incidence of ADAs |
| <ul> <li>To evaluate disease-related symptom improvement, as measured by the GaCS of the FACT-Ga and the ECS of the FACT-E in treated participants</li> <li>To evaluate general health, functional status, and utility</li> </ul> | <ul> <li>OS rate at certain time points</li> <li>Summary measures of EQ-5D-3L index and<br/>VAS scores, GaCS scores, and/or ECS scores,<br/>and corresponding change form baselines for</li> </ul> |
| for health using the EQ-5D-3L in treated participants | each score |

Abbreviations: ADA = anti-dug antibody; AE = adverse event; BOR = best overall response; CR = complete response; DOR = duration of response; EQ 5D-3L = 3-level version of EQ-5D self-report questionnaire; EC =

esophageal cancer; ECS = Esophagus Cancer Subscale; FACT-E = Functional Assessment of Cancer Therapy-Esophageal; FACT-Ga = Functional Assessment of Cancer Therapy-Gastric; GaCS = Gastric Cancer Subscale; GC=gastric cancer; IP = investigational product; ORR = objective response rate; OS = overall survival; PFSR = progression-free survival rate; PK = pharmacokinetic; PR = partial response; RECIST = Response Evaluation Criteria in Solid Tumors; SAE = serious adverse event; VAS = visual analog scale

### **Overall Design:**

This is a rolling, Phase 2, adaptive study that will evaluate the preliminary efficacy, safety, tolerability, PK, and pharmacodynamics of novel FRACTION-Gastric Cancer study treatment combinations in participants with advanced GC and/or EC. The details pertaining to the specific study treatment regimens are provided in each FRACTION-Gastric Cancer Sub-Protocol.

Participants will be enrolled in 1 of the 2 tracks. Participants who are anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment naïve will be enrolled for Track 1. Participants who have had prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment will be assigned to Track 2.

Participants on Tracks 1 and 2 will begin on the Treatment Phase (with a total duration of approximately 2 years). Tumor assessments will be conducted according to the timing described in each FRACTION-Gastric Cancer Sub-Protocol.

Participants in Tracks 1 and 2 will be treated until completion of the Treatment Phase, progression, toxicity, or protocol-specified discontinuation.

### **Number of Participants:**

For Sub-Protocols utilizing a Simon-2 stage (optimal) design, up to 54 anti-PD-1/PD-L1 or anti-CTLA-4 treatment-naive participants will be treated per study treatment combination in Track 1. In Track 2, up to 41 participants will be treated per study treatment combination.

For Sub-Protocols not utilizing a Simon-2 stage (optimal) design, a different sample size may be used depending on the statistical considerations for those treatment combinations. In those cases, sample size will be discussed within the individual Sub-Protocols.

### **Treatment Arms and Duration and Study Treatments:**

Specific dosing and treatment regimens for each FRACTION-Gastric Cancer study treatment combination are outlined in each FRACTION-Gastric Cancer Sub-Protocol.

### 2 SCHEDULE OF ACTIVITIES

Study assessments and procedures are presented in Table 2-1 (Screening Procedural Outline), Table 2-2 (Baseline for Re-randomization Procedural Outline), and Table 2-3 (Follow-up Procedural Outline). The On-treatment Procedural Outline(s) and exceptions for study treatment combination arms are included in each Fast Real-time Assessment of Combination Therapy in Immuno-ONcology (FRACTION)-Gastric Cancer Sub-Protocol.

 Table 2-1:
 Screening Procedural Outline

| Procedure | Screening<br>Visit <sup>a</sup> | Notes |
|---|---|---|
| Eligibility Assessments | • | |
| Informed Consent | X | A participant is considered enrolled only when a protocol-specific informed consent is signed. Obtain patient identification number via IRT after signing of the written informed consent. |
| Utilize IRT | X | Obtain patient identification number. After completing all screening procedures, utilize IRT to either screen fail or obtain randomization information, as applicable. Randomization can occur up to 7 days prior to first dose. In limited circumstances, if patients cannot be treated within 7 days of randomization due to a study-related test, the duration can be extended after discussion with the medical monitor. |
| Inclusion/Exclusion Criteria | X | All inclusion/exclusion criteria should be assessed at screening and confirmed prior to first dose. |
| Medical History | X | Includes prior conditions and any toxicities or allergies related to previous treatments |
| Collect Data on Prior Anti-PD-1,<br>Anti-PD-L1, or Anti-CTLA-4 Treatment<br>Exposure | X | Prior to screening for the protocol, investigative sites are required to determine the participant's exposure to anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment. Those data will be collected as part of the Screening Phase. Toxicities from prior immunotherapies with details on timing, treatment, and resolution, if applicable, should be captured. |
| Prior Therapy | X | Radiotherapy/surgery/systemic therapy administered for the treatment of gastric cancer |
| Safety Assessments | | |
| | | If the screening physical examination is performed within 24 hours prior to dosing on Day 1, then a single examination may count as both the screening and predose evaluation. |
| Oxygen Saturation | X | Record at rest and after mild to moderate exertion via pulse oximetry to establish baseline. If participant has oxygen saturation $\leq 90\%$ , consult the BMS Medical Monitor (or designee) prior to enrollment. |
| Physical Measurements | X | Include height and weight |
| Vital Signs | X | Include body temperature, seated blood pressure, and heart rate |
| ECOG Performance Status | X | |

Protocol Amendment No.: 06

Date: 13-Aug-2021

Approved v8.0

930104678 8.0

 Table 2-1:
 Screening Procedural Outline

| Procedure | Screening<br>Visit <sup>a</sup> | Notes |
|---|---|---|
| 12-lead ECG X | | ECGs should be recorded after the participant has been supine for at least 5 minutes. Record QTcF. If ECG abnormality is noted, a repeat ECG must be performed. |
| Chest X-ray | X* | *Optional |
| Concomitant Medication Collection | X | Includes medications taken within 14 days prior to assigned study treatment |
| Assessment of Baseline Signs and<br>Symptoms | X | Assess within 14 days prior to first dose of study treatment. |
| <b>Laboratory Tests</b> | | Include blood and urine samples |
| Hematology | X | Includes CBC with differential including platelets |
| Serum Chemistry <sup>b</sup> | X | See Section 9.4.1. |
| Thyroid Function Panel <sup>b</sup> X | | If TSH is abnormal, then obtain free T3 and T4. |
| Serology X | | Perform testing for Hepatitis A IgM and IgG antibodies, HBsAg, hepatitis C antibody (if hepatitis C antibody is positive, reflex to hepatitis C RNA), or hepatitis C RNA. (Note: Testing for HIV-1 and HIV-2 must be performed at sites where mandated by local requirements. For sites in Germany, see Appendix 8.) |
| Pregnancy Serum or Urine Test | For WOCBP only. Serum or urine, within 24 hours prior to first dose of assi treatment. An extension of up to 72 hours prior to start of study treatment is situations where results cannot be obtained within the standard 24-hour wind | |
| Follicle Stimulating Hormone X | | For women only. Refer to Appendix 4. |
| Mandatory Pretreatment Tumor Biopsy X | | Biopsy must be performed during the Screening Phase in all participants prior to randomization. Tumor tissue must be obtained from a primary or metastatic site. Adequacy of tumor tissue must be confirmed by central laboratory prior to randomization. (Note: Fine needle aspiration and bone metastases samples are not acceptable for submission.) |
| | | An archival, formalin-fixed, paraffin-embedded tumor tissue block (preferred) or a minimum of 20 slides of samples from a primary or metastatic site should be provided by all participants, if available. |

930104678 8.0

Approved v8.0

Protocol Amendment No.: 06

15

Table 2-1: Screening Procedural Outline

| Procedure | Screening<br>Visit <sup>a</sup> | Notes |
|---|---|---|
| Efficacy Assessment | | |
| Baseline Tumor Assessment | X | Assessed by RECIST v1.1 criteria (see Appendix 5) |
| | | Disease assessment with contrast-enhanced CT/MRI scans acquired on dedicated CT/MRI |
| | | equipment is preferred for this study. CT or MRI of the chest, abdomen, pelvis, and all known |
| | | sites of disease should be performed within 28 days prior to first dose of study treatment. Assessment must include other anatomic regions, as indicated based on the participant's tumor type and/or disease history. |
| | | Participants with a history of brain metastasis should have an MRI (preferred) or CT of the brain. |
| | | Participants with a history of bone metastasis should have a bone scan. |
| AE Reporting | | |
| SAEs | X | All SAEs must be collected from the date of the participant's written consent until 100 days post-discontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. All SAEs and AEs will be assessed using NCI CTCAE Version 4.03. |

<sup>&</sup>lt;sup>a</sup> Within 28 days of first dose of assigned study treatment unless specified in notes section.

Abbreviations: AE = adverse event; BMS = Bristol-Myers Squibb Company; CBC = complete blood count; CT = computed tomography; CTCAE = Common Terminology Criteria for Adverse Events; CTLA-4 = cytotoxic T-lymphocyte antigen 4; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; HBsAg = hepatitis B surface antigen; HIV = human immunodeficiency virus; IgG = immunoglobin G; IgM = immunoglobin M; IRT = Interactive Response Technology; MRI = magnetic resonance imaging; NCI = National Cancer Institute; PD-1 = programmed death-1; PD-L1 = programmed death-ligand 1; QTcF = QT interval corrected with Fridericia's formula; RECIST = Response Evaluation Criteria in Solid Tumors; RNA = ribonucleic acid; SAE = serious adverse event; T3 = triiodothyronine; T4 = thyroxine; TSH = thyroid-stimulating hormone; WOCBP = women of child-bearing potential.

Protocol Amendment No.: 06

b If a participant is screened and begins study treatment within 3 days, the laboratory assessments for the Screening Phase can be used for Day 1 of the On-treatment Procedural Outline in each FRACTION-Gastric Cancer Sub-Protocol as well.

 Table 2-2:
 Baseline for Re-randomization Procedural Outline

| Procedure | Days -1<br>to -28 <sup>a</sup> | Notes |
|---|---|---|
| Eligibility Assessments | X X | Participants must continue to meet eligibility criteria. All inclusion/exclusion criteria should be assessed at the retreatment/re-randomization baseline visit and confirmed prior to first dose. |
| Informed Consent | X | Participants must sign informed consent for retreatment/re-randomization. |
| Participant Registration for Retreatment/Rerandomization | X | Ensure participant continues to meet eligibility for study treatment. |
| Safety Assessments | - | |
| Physical Examination | X | If the retreatment/re-randomization baseline physical examination is performed within 24 hours prior to dosing on Day 1, then a single examination may count as both the retreatment/re-randomization baseline and predose evaluation. |
| Physical Measurements | X | Include weight |
| Vital Signs X Include body temperature, seated blood pr | | Include body temperature, seated blood pressure, and heart rate |
| ECOG Performance Status | X | |
| 12-lead ECG | X | ECGs should be recorded after the participant has been supine for at least 5 minutes. Record QTcF. If ECG abnormality is noted, a repeat ECG must be performed. |
| Concomitant Medication Collection | X | Includes medications taken within 14 days prior to study treatment |
| Oxygen Saturation | X | Record at rest and after mild to moderate exertion via pulse oximetry to establish baseline. If participant has oxygen saturation ≤ 90%, consult BMS Medical Monitor (or designee) prior to entering retreatment/re-randomization. |
| Assessment of Baseline Signs and Symptoms | X | If re-baseline or re-randomization occurs > 100 days after the last dose, signs and symptoms that occur up to 14 days prior to the next dose of study treatment should be recorded. |
| Laboratory Tests | • | Include blood and urine samples |
| Hematology | X | Includes CBC with differential including platelets |
| Serum Chemistry <sup>b</sup> | X | See Section 9.4.1. |

Protocol Amendment No.: 06

 Table 2-2:
 Baseline for Re-randomization Procedural Outline

| Procedure | Days -1<br>to -28 <sup>a</sup> | Notes |
|---|---|---|
| Thyroid Function Panel <sup>b</sup> | X | If TSH is abnormal, then obtain free T3 and T4. |
| Serology | X | Serology must be collected if > 6 months has passed since the previous assessment. Perform testing for Hepatitis A IgM and IgG antibodies, HBsAg, hepatitis C antibody (if hepatitis C antibody is positive, reflex to hepatitis C RNA), or hepatitis C RNA. (Note: Testing for HIV-1 and HIV-2 must be performed at sites where mandated by local requirements.) |
| Pregnancy Serum or Urine Test | X For WOCBP only. Serum or urine, within 24 hours prior to first dose of as study treatment. An extension of up to 72 hours prior to start of study treat permissible in situations where results cannot be obtained within the stand hour window. | |
| Follicle Stimulating Hormone | X | For women only. Refer to Appendix 4. |
| Mandatory Pretreatment Tumor Biopsy | X | A mandatory pretreatment fresh tumor biopsy must be performed if a progression biopsy from the current study is not available. Sufficient tumor tissue must be obtained before start of study treatment from a primary or metastatic site. Tumor tissue samples must be shipped from site to central laboratory prior to retreatment/re-randomization. (Note: Fine needle aspiration and bone metastases samples are not acceptable for submission.) |
| Efficacy Assessments | | |
| Baseline Tumor Assessment | X | Assessed by RECIST v1.1 criteria (see Appendix 5) |
| | | Disease assessment with contrast-enhanced CT/MRI scans acquired on dedicated CT/MRI equipment is preferred for this study. CT or MRI of the chest, abdomen, pelvis, and all known sites of disease should be done within 28 days prior to first dose of study treatment. Assessment must include other anatomic regions, as indicated based on the participant's tumor type and/or disease history. |
| | | Participants with a history of brain metastasis should have an MRI (preferred) or CT of the brain, or if clinically indicated. |
| | | Participants with a history of bone metastasis should have a bone scan, or if clinically indicated. |

Protocol Amendment No.: 06

Date: 13-Aug-2021

Approved v8.0

930104678 8.0

Table 2-2: Baseline for Re-randomization Procedural Outline

| Procedure | Days -1<br>to -28 <sup>a</sup> | Notes |
|---|---|---|
| AE Reporting | | |
| SAEs | X | All SAEs must be collected from the date of the participant's written consent until 100 days postdiscontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. All SAEs and AEs will be assessed using NCI CTCAE Version 4.03. |

<sup>&</sup>lt;sup>a</sup> Within 28 days of first dose of assigned study treatment unless otherwise specified in notes section.

Abbreviations: AE = adverse event; BMS = Bristol-Myers Squibb Company; CBC = complete blood count; CT = computed tomography; CTCAE = Common Terminology Criteria for Adverse Events; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; HBsAg = hepatitis B surface antigen; HIV = human immunodeficiency virus; IgG = immunoglobin G; IgM = immunoglobin M; MRI = magnetic resonance imaging; NCI = National Cancer Institute; PK = pharmacokinetic; QTcF = QT interval corrected with Fridericia's formula; RECIST = Response Evaluation Criteria in Solid Tumors; RNA = ribonucleic acid; SAE = serious adverse event; T3 = triiodothyronine; T4 = thyroxine; TSH = thyroid-stimulating hormone; WOCBP = women of child-bearing potential.

Protocol Amendment No.: 06

b If a participant is screened and begins study treatment within 3 days, the laboratory assessments for the Screening Phase can be used for Day 1 of the On treatment- Procedural Outline in each FRACTION-Gastric Cancer Sub-Protocol as well.

Note: On-treatment Procedural Outlines are in the relevant FRACTION-Gastric Cancer Sub-Protocol

Table 2-3: Follow-up Procedural Outline

| | Safety Follow-up <sup>a</sup> | | | |
|---|---|---|---|---|
| Procedure | FU 1<br>30 Days<br>(± 7 Days) | FU 2<br>60 Days<br>(± 7 Days) | FU 3<br>100 Days<br>(± 7 Days) | Notes |
| Safety Assessments | | | | |
| Physical Examination | X | X | X | |
| Oxygen Saturation | X | As clinically indicated | | Record at rest and after mild to moderate exertion via pulse oximetry. |
| Vital Signs and Weight | X | X | X | Includes body temperature, seated blood pressure, and heart rate |
| ECOG Performance Status | X | X | X | |
| Review of Concomitant<br>Medications | X | X | X | |
| <b>Laboratory Tests</b> | | | | |
| Hematology and Serum<br>Chemistry | X | | X | |
| PK Samples <sup>c</sup> | X | | | Details are provided in each FRACTION-Gastric Cancer Sub-Protocol. |
| Anti-drug Antibody Samples <sup>c</sup> | X | | | Details are provided in each FRACTION-Gastric Cancer Sub-Protocol. |
| AE Reporting | | | | |
| Monitor for Nonserious AEs | X | X | X | Nonserious AEs must be collected from first dose until 100 days following the last dose of study treatment. All SAEs and AEs will be assessed using NCI CTCAE Version 4.03. |

Protocol Amendment No.: 06

Date: 13-Aug-2021

Approved v8.0 930104678 8.0

 Table 2-3:
 Follow-up Procedural Outline

| | Safety Follow-up <sup>a</sup> | | | |
|---|---|---|---|---|
| Procedure | FU 1<br>30 Days<br>(± 7 Days) | FU 2<br>60 Days<br>(± 7 Days) | FU 3<br>100 Days<br>(± 7 Days) | Notes |
| Monitor for SAEs | X | X | X | All SAEs must be collected from the date of the participant's written consent until 100 days postdiscontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. All SAEs and AEs will be assessed using NCI CTCAE Version 4.03. |
| Efficacy Assessments | 1 | | 1 | |
| Tumor Response<br>Assessment <sup>c</sup> | X | | X | Assessed by RECIST v1.1 criteria (see Appendix 5). Participants with a history of brain metastasis should have an MRI (preferred) or CT of the brain, if clinically indicated. Participants with a history of bone metastasis should have a bone scan, if clinically indicated. All participants should receive scans at FU1 except for participants who started subsequent therapy or participants with PD who have already been treated beyond progression. Scans at FU3 and every 12 weeks (±14 days) will only be collected for participants with CR, PR, SD, or NE at treatment discontinuation. |

Protocol Amendment No.: 06

Date: 13-Aug-2021

Approved v 8.0 930104678 8.0

| | Safety Follow-up <sup>a</sup> | | | |
|---|---|---|---|---|
| Procedure | FU 1<br>30 Days<br>(± 7 Days) | FU 2<br>60 Days<br>(± 7 Days) | FU 3<br>100 Days<br>(± 7 Days) | Notes |
| Patient-reported Outcomes<br>Assessment <sup>c</sup> | X | X | X | EQ-5D-3L and GaCS and/or ECS Can be collected by telephone at regularly scheduled times |
| Collection of Survival Status<br>and Subsequent Treatment<br>Information <sup>c</sup> | Х | X | X | Safety follow-up visits must occur in the office. Response (and survival) follow-up visits may be performed by telephone contact or clinic visit. |

<sup>&</sup>lt;sup>a</sup> FU visits at 30, 60, and 100 days (± 7 days) should occur after the last dose of study treatment or coinciding with the date of discontinuation ± 7 days, if the date of discontinuation is greater than 30 days after the last dose, to monitor for AEs.

Abbreviations: AE = adverse event; BMS = Bristol-Myers Squibb Company; CR = complete response; CT = computed tomography; CTCAE = Common Terminology Criteria for Adverse Events; ECOG = Eastern Cooperative Oncology Group; ECS = Esophagus Cancer Subscale; EQ-5D-3L = 3-level version of EQ-5D self-report questionnaire; FU = follow-up; GaCS = Gastric Cancer Subscale; MRI = magnetic resonance imaging; NCI = National Cancer Institute; PD = progressive disease; PK = pharmacokinetic; PR = partial response; RECIST = Response Evaluation Criteria in Solid Tumors; SAE = serious adverse event; SD = stable disease.

Protocol Amendment No.: 06

b Not applicable as of Protocol Amendment 06: Additional survival follow-up will be collected every 6 months for 3 additional years (2 years of response follow-up + 3 years of survival follow-up = total of 5 years of follow-up). BMS may request that survival data be collected on all treated/randomized participants outside of the protocol-defined window. At the time of this request, each participant will be contacted to determine their survival status unless the participant has withdrawn consent for all contacts or is lost to follow-up. Withdrawal of consent must be clearly documented. See Section 5.1.3.3 for details.

As of Protocol Amendment 06: Assessments necessary for monitoring safety (eg, safety labs, oxygen saturation, vital signs, physical exams, review of concomitant medications, AE/ SAE reporting, etc) will continue per sub-protocol until the FU 3 visit. Tumor Scans, survival status follow-ups, and collection of subsequent treatment information will end once the participant has disease progression, or treatment discontinuation for any reason, whichever occurs first. Collection of samples for PK, ADA, biomarkers, as well as collection of data for patient-reported outcomes should be discontinued. The intent is to minimize the burden on study participants and site staff.

In the event that multiple procedures are required at a single time point, the following is a list of procedures from highest priority to lowest:

- Safety (clinical laboratory examinations)
- Safety (electrocardiogram [ECG])
- Biomarker sampling
- Pharmacokinetic (PK) and anti-drug antibody (ADA) sampling

Protocol Amendment No.: 06

#### 3 INTRODUCTION

Traditional or conventional treatment options for patients with advanced cancer include surgery, radiation, chemotherapy, and hormonal therapy. Despite advances in these therapies, the majority of patients with metastatic disease die from progressive disease (PD). Immunotherapeutic approaches have demonstrated clinical efficacy and have been approved in multiple countries worldwide and in several solid tumor malignancies, including melanoma, renal cell, lung, and hormone-refractory prostate cancers. Tumors may modulate and evade the host immune response through a number of mechanisms, including downregulation of tumor-specific antigen expression and presentation, secretion of anti-inflammatory cytokines, and upregulation of inhibitory ligands. T-cell checkpoint regulators such as cytotoxic T-lymphocyte-antigen 4 (CTLA-4; see Appendix 1) and programmed death-1 (PD-1, cluster of differentiation [CD] 279) are cell surface molecules that, when engaged by their cognate ligands, induce signaling cascades that downregulate T-cell activation and proliferation. One proposed model by which therapeutic T-cell checkpoint inhibitors derive anti-tumor activity is through breaking of immune tolerance to tumor cell antigens by T-cell activation and proliferation.

Following on the success of anti-CTLA-4 and anti-PD-1 pathway-targeted agents in several cancers, the field of tumor immunotherapy is rapidly expanding. In addition to blocking these and other co-inhibitory pathways such as lymphocyte activation gene 3 (LAG-3), activating co-stimulatory pathways to potentiate anti-tumor immune responses is being evaluated as a promising approach.<sup>3</sup> Members of the tumor necrosis factor receptor super family (TNFRsf) include several co-stimulatory proteins with key roles in B- and T-cell development, survival, immune activation, and anti-tumor immune responses.<sup>4</sup> Preclinical data have provided the basis for clinical studies of agonist antibodies to such TNFRsf co-stimulatory receptors such as 4-1BB, <sup>5,6</sup> OX40, <sup>7,8</sup> glucocorticoid-induced tumor necrosis factor receptor-related (GITR) gene, <sup>9,10</sup> and CD27, <sup>11,12</sup> along with a growing list of immuno-oncology (IO) targets that modulate other immunomodulatory mechanisms as potential therapies for patients with cancer. Overall, enhancement of the magnitude and potency of tumor antigen-specific adaptive cellular responses by CD8 and CD4 T cells is now considered a major goal in cancer immunotherapy.

With emerging clinical data showing significant activity of single agent immunotherapies, it is possible, and indeed likely, that- combination therapies could potentially lead to a greater depth of response and an increase in overall survival (OS), as has been noted with the combination of anti-PD-1 and anti-CTLA-4 in participants with advanced melanoma and renal cell carcinoma. <sup>13,14,15,16</sup> This raises the possibility that combining agents with a broader range of relevant targets (eg, checkpoint blocking antibodies with agonist antibodies to T-cell co-stimulatory molecules and immunomodulatory agents) is likely to lead to durable, long-term responses and possibly even cures in this high unmet medical need population of patients with metastatic or refractory tumors. Preclinical data from evaluation of combinations in mouse tumor models indicate that treatment with the combination of IO agents may lead to enhanced anti-tumor activity above that from each agent alone. <sup>17</sup> Thus, the combination of IO agents has the potential to provide clinical benefit to such patients with high unmet medical needs.

## 3.1 Study Rationale

## 3.1.1 FRACTION Program

## 3.1.1.1 Rationale for the FRACTION Program

Bristol-Myers Squibb Company (BMS) has an extensive portfolio of novel agents that span a variety of targets. Within the immune system, these include T-cell checkpoint inhibitors, co-stimulatory molecules acting on T cells, regulatory T cell- and natural killer (NK) cell targeted- agents, treatments that alter the tumor microenvironment to favor a tumor inhibitory milieu, and treatments that target myeloid-derived suppressor cells or tumor-associated- macrophages. In addition to agents that target the immune system, BMS has a portfolio of agents that directly target tumor cells. These include antibody drug conjugates and both biologic and small molecule inhibitors of key signaling pathways. In fact, the number of compounds to be evaluated has grown so large that it is no longer possible or efficient to test all possible combinations in a standard clinical Phase 1 or Phase 2 setting.

To determine which combinations show the most clinical promise and thus should be prioritized for registrational studies, BMS has initiated the FRACTION Program (globally listed under the descriptor, BMS-986217). The FRACTION Program will employ repeat core biopsies and serial assessments with different treatment options. These approaches are supported by the National Cancer Institute (NCI) Biomarker-integrated Approaches of Targeted Therapy for Lung Cancer Elimination (BATTLE) program, <sup>18</sup> the Investigation of Serial Studies to Predict Your Therapeutic Response with Imaging And moLecular Analysis (I-SPY 1/2 TRIAL), <sup>19</sup> the Lung-MAP: S1400 Biomarker-targeted Second-line Therapy in Treating Patients With Recurrent Stage IIIB-IV Squamous Cell Lung Cancer (NCT02154490), <sup>20</sup> the NCI Molecular Analyses for Therapy Choice (NCT02465060), and the American Society of Clinical Oncology's Targeted Agent and Profiling Utilization Registry. <sup>21</sup> These studies use innovative trial designs to quickly assess new agents in participants with the goal of reducing the time and number of participants required to bring these therapies to those who will benefit from them.

The FRACTION Program will consist of several FRACTION studies, each in a specific tumor type and with a well-defined participant population. Each FRACTION study will have a Master Protocol, which will apply to all study treatment combinations selected for evaluation under that tumor-specific FRACTION study and any control treatments. For the FRACTION Program, it is intended that combination agents will be IO agents within the BMS pipeline or IO agents already approved; however, they may also include small molecule agents or other modalities for which there is scientific rationale for combining with an IO agent in a given disease. All novel FRACTION combinations will be selected based on sound scientific rationale, supported whenever possible and appropriate by in vivo model systems, to demonstrate anti-cancer activity and preliminary assessments of clinical tolerability.

Specific study treatment combinations and/or control treatments will be introduced in FRACTION Sub-Protocols for each FRACTION study; these Sub-Protocols will be appended to the Master

Protocol for that study and will include information appropriate to the study treatment combinations and/or control treatments being added to the study, including the preclinical rationale, preclinical toxicology, and clinical safety data, as well as PK and pharmacodynamic information (PD), as available. The minimum preclinical safety information provided in each Sub-Protocol will include the definitive studies that were used to support the health authorities and review for each individual agent, along with any additional preclinical safety studies that were conducted subsequent to the original applications. In addition, the toxicology rationale to support each combination will be discussed. For each agent, the established monotherapy and relevant combination clinical safety package from studies done outside of FRACTION will be included. Participants within the FRACTION Program will not be the first to be exposed to any treatment.

Thus, for the FRACTION Program, study treatment combinations that have high potential to produce transformational anti-tumor activity compared to the control will be selected based on both preclinical and early clinical trials data. The first study in the FRACTION Program, Study CA018001, "Phase 2, Fast Real-time Assessment of Combination Therapies in Immuno-ONcology Study in Subjects with Advanced Non-small Cell Lung Cancer (FRACTION-Lung)," is ongoing. FRACTION-Renal Cell Carcinoma (RCC) is also ongoing.

## 3.1.1.2 Specific Attributes of the FRACTION Program Design

The specific attributes of the FRACTION Program include the following:

- An innovative study design providing participants with advanced cancer the possibility of expeditious access to innovative therapies, including combinations with approved treatments like nivolumab. In addition, it will provide an ongoing treatment option for participants across the spectrum of their disease as they progress through the FRACTION Program, as participants can enter into different treatment "Tracks" based upon their treatment exposure and response.
- A streamlined decision-making process allowing for more rapid and efficient selection of promising treatment options in BMS's evolving portfolio of oncology assets. This extensive pipeline of novel targets and/or agents could result in an excess of 100 individual monotherapy and doublet combinations in need of study. The challenges to study all possible combinations in a traditional clinical program are daunting, especially since animal models and/or biomarker data still cannot effectively predict participant responses. This means that clinical exploration in participants is required if it is to be truly informative and would ultimately lead to participant's benefit. Thus, FRACTION is designed as a way to explore and compare multiple IO combinations against each other and against a control treatment.
- A Master Protocol, in conjunction with appended FRACTION Sub-Protocols, allowing for operational efficiencies for the rapid and efficient opening of new study treatment combination arms and closing of other study treatment combination arms that have demonstrated unacceptable toxicity or futility
- A continuous throughput design allowing data to be available sooner to support either closure of study treatment combination arms (initial signal-seeking arms) or adaptively increasing sample size for further investigation with additional eligibility criteria and statistical considerations in a new sub-protocol if promising efficacy is seen with a treatment combination. This will drive and improve selection and acceleration of optimal combinations to help patients with cancer in dire need of new effective treatment options.

#### 3.1.1.3 Rationale for Biomarker Assessments

that will apply to all novel FRACTION Program study combinations so that comparisons of such data can be made across different study treatments. The goals of the biomarker assessments proposed in the FRACTION Program are to 1) identify predictive biomarkers for both safety and efficacy of a given combination, 2) define the mechanism of action for a particular combination (pharmacodynamic assessment), and 3) determine the mechanisms of resistance to a particular combination. In addition, there will be biomarker assessments that are applied specifically for a given combination as dictated by the biology of the combination.





## 3.2 Background

#### 3.2.1 FRACTION-Gastric Cancer

Gastric and esophageal cancers are among the leading causes of mortality worldwide and are responsible for a combined total of 1,407,000 new cases and 1,123,000 deaths every year. These, therefore, represent the most prevalent subtypes of GI malignancies worldwide, with an alarming increase in esophageal adenocarcinoma in many Western populations in recent decades. Gastric cancer (GC) is the 5th leading cancer and the 3rd leading cause of cancer-related deaths worldwide. The incidence varies with different geographic regions, with over 70% of GCs occurring in developing countries. While esophageal cancer (EC) has a lower incidence (8th most common cancer), overall mortality of EC is high. Moreover, adenocarcinoma of from gastric cardia, GEJ and distal esophagus is increasing in the West. GC and EC often present as advanced disease upon diagnosis.

Locally advanced unresectable and metastatic esophagagogastric carcinomas are not curable and highly lethal. While etiologic, epidemiologic, and biologic heterogeneity among esophagogastric carcinomas are well recognized, similar chemotherapy regimens are used in treatment of metastatic disease. Platinum compounds (oxaliplatin and cisplatin) and fluoropyrimidines (5-fluorouracil, capecitabine, and tegafur/gimeracil/oteracil potassium) are generally considered as standard-of-care treatment options in metastatic EC, GC and GEJ cancer across geographic regions. <sup>25,26,27</sup> Targeted agents that have shown benefit are trastuzumab (for HER-2 positive tumors) and ramucirumab for esophagogastric adenocarcinoma. <sup>28,29,30</sup> The different biologic characteristics and treatment approaches among regions result in different survival outcomes, with median OS durations of 12 to 14 months in Asian countries and 8 to 11 months in the US and Europe. <sup>31,32,33</sup>

Immunotherapeutic approaches have demonstrated clinical efficacy in several advanced solid tumor cancers, including esophagogastric cancer, melanoma, non-small cell lung cancer (NSCLC), renal cell carcinoma, classical Hodgkin lymphoma, recurrent or metastatic squamous cell carcinoma of the head and neck, locally advanced or metastatic urothelial carcinoma, hepatocellular carcinoma, and microsatellite instability-high or mismatch repair deficient metastatic colorectal cancer. 34,35,36,37,38 Nivolumab (BMS-936558), a PD-1 antibody, and ipilimumab (BMS-734016), a CTLA-4 antibody, are such immunotherapies that have been approved in the US, Europe, Japan, and other countries. 38,39,40,41

Preclinical data indicate that the combination of PD-1 and CTLA-4 receptor blockade may further improve anti-tumor activity. <sup>42</sup> In vitro combinations of nivolumab plus ipilimumab increased IFNy

production 2- to 7-fold over either agent alone in a mixed lymphocyte reaction. In a murine melanoma vaccine model, blockade with either CTLA-4 or PD-1 antibodies increased the proportion of CTLA-4- and PD-1-expressing CD4/CD8 tumor-infiltrating T-effector cells, and dual blockade increased tumor infiltration of T-effector cells and decreased intratumoral T regulatory cells, as compared to either agent alone. 42

In patients with esophagogastric cancer, tumors with programmed death-ligand 1 (PD-L1) expression have been reported to be associated with depth of muscle invasion, tumor size, and lymph node metastasis. The survival of patients with PD-L1- or programmed death-ligand 2 (PD-L2)-expressing tumors is significantly worse than for those patients without PD-L1/PD-L2-expressing tumors. PD-L1 or PD-L2-expressing tumors have been reported in approximately 22% to 40% of GC, and PD-L1 has been suggested as a prognostic marker for both GC and EC. <sup>43,44</sup> Thus, blockage of PD-1/PD-L1/PD-L2 might improve the survival of GC patients. To that end, anti-PD-1 and PD-L1 inhibitors (eg, nivolumab, pembrolizumab, and avelumab) have been investigated in GC treatment and have demonstrated anti-tumor activity. 45,46,47 Nivolumab showed an improvement in response rate, progression free survival, and OS compared to placebo in Japanese patients with GC treated with 2 or more lines of chemotherapy, irrespective of PD-L1 status. 48 Anti-PD-1 antibody pembrolizumab was approved in patients with recurrent locally advanced or metastatic, gastric, or GEJ adenocarcinoma whose tumors express PD-L1, as determined by an FDA-approved test and patients must have had disease progression on or after 2 or more prior systemic therapies, including fluoropyrimidine- and platinum-containing chemotherapy and, if appropriate, human epidermal growth factor receptor 2 (HER2)/neu-targeted therapy. <sup>49,50</sup> Pembrolizumab is also approved (accelerated approval) for the treatment of patients with MSI-H (microsatellite instability-high)/dMMR (mismatch repair deficient) cancers with no satisfactory alternative treatment options.

Combining immunotherapeutic agents with different mechanisms of action offers the possibility of further benefit, as noted with the combination of nivolumab and ipilimumab now approved in the US for the treatment of patients with metastatic melanoma. In Study CA209032 ("A Phase 1/2, Open-label Study of Nivolumab Monotherapy or Nivolumab combined with Ipilimumab in Subjects with Advanced or Metastatic Solid Tumors," NCT01928394), participants with GC or GEJ were treated with nivolumab 1 mg/kg in combination with ipilimumab 3 mg/kg or nivolumab monotherapy. Participants treated with nivolumab 1 mg/kg in combination with ipilimumab 3 mg/kg had an objective response rate (ORR) of 24% and 12-month progression-free survival rate (PFSR) of 17%. This was greater than the ORR and 12-month PFSR in participants treated with nivolumab monotherapy, who had an ORR of 12% and a PFSR of 8%. This study treatment combination regimen has also been chosen for use in a Phase 3 registration study in first-line GC. Hence, nivolumab 1 mg/kg in combination with ipilimumab 3 mg/kg has been chosen as the control treatment in FRACTION-Gastric Cancer Sub-Protocol A. (Further details are described in the FRACTION-Gastric Cancer Sub-Protocol A). These data also suggest the potential for other combinations to bring additional benefit to participants with GC and GEJ.

This document will serve as the Master Protocol for the FRACTION-Gastric Cancer study (FRACTION-Gastric Cancer; CA018003). As described above, novel study treatment combinations and/or additional controls will be appended as FRACTION-Gastric Cancer Sub-Protocols. These FRACTION-Gastric Cancer Sub Protocols- will evaluate the safety profile, tolerability, preliminary efficacy, PK, and pharmacodynamics of novel study treatment combinations in participants with advanced GC. The initial control treatment in the FRACTION-Gastric Cancer study will be nivolumab in combination with ipilimumab followed by nivolumab monotherapy, similar to what has been administered in Study CA209032 as described above.

#### 3.3 Benefit/Risk Assessment

An overall risk/benefit assessment for each novel FRACTION-Gastric Cancer study treatment combination will be provided in each FRACTION-Gastric Cancer Sub-Protocol.

Non-live coronavirus disease 2019 (COVID-19) vaccination is considered a simple concomitant medication within the study. However, the efficacy and safety of non-live vaccines (including non-live COVID-19 vaccines) in participants receiving investigational agents is unknown.

# 3.3.1 Safety Monitoring on Study Treatment

Frequent safety assessments will be carried out by the Sponsor/BMS Medical Monitor (or designee) and investigators throughout the study to determine whether dose modification, additional safety measures, or termination of the study treatment combination arm is required at any time. In addition, AEs and serious adverse events (SAEs) will be reviewed regularly by the BMS Medical Monitor (or designee) and the Pharmacovigilance group to look for trends and potential safety signals. Treatment of AEs will follow institutional guidelines and recommended management algorithms, as listed in the Investigator's Brochure (IB) and prescribing information, as applicable, for each combination agent and control comparator, and provided as appendices to this protocol. Specific algorithms for the management of immune-related AEs are provided in Appendix 6 and are applicable to immune-related AEs for all FRACTION-Gastric Cancer study treatment combinations.

#### 4 OBJECTIVES AND ENDPOINTS

The overall FRACTION-Gastric Cancer study-wide objectives are presented in the following sections. Any changes to these objectives for specific study treatments are specified in each FRACTION-Gastric Cancer Sub-Protocol.

Protocol Amendment No.: 06

Table 4-1: Objectives and Endpoints

| | Objectives | Endpoints | |
|---|---|---|---|
| Pri | mary | | |
| • | To assess the efficacy (ORR, DOR, and PFSR at 24 weeks) of each FRACTION-Gastric Cancer study treatment combination (relative to nivolumab in combination with ipilimumab, when applicable) in participants with advanced GC and/or EC | • | ORR, defined as the proportion of all treated participants with a BOR of CR or PR as assessed per RECIST v1.1 by investigator, median DOR, and PFSR at 24 weeks |
| Sec | ondary | | |
| • | To investigate additional safety and tolerability of each FRACTION-Gastric Cancer study treatment combination in participants with advanced GC and/or EC | • | Incidence of AEs, SAEs, and AEs leading to discontinuation, deaths, and clinical laboratory test abnormalities |
| Tei | tiary/Exploratory | | |
| • | To evaluate the PK of each IP component To evaluate the immunogenicity of each IP, when applicable To evaluate disease-related symptom improvement, as measured by the GaCS of the FACT-Ga and the ECS of the FACT-E in treated participants To evaluate general health, functional status, and utility for health using the EQ-5D-3L in treated | • | Summary measures of change (or % change) from baseline or baseline level biomarker measurements Correlation (or similar appropriate measure of association) of biomarker measure Summary measures of PK parameters from serum concentration Incidence of ADAs OS rate at certain time points Summary measures of EQ-5D-3L index and VAS scores, GaCS scores, and/or ECS scores, and corresponding change form baselines for each score |
| A 1 1 | participants | | The population of |

Abbreviations: CR = complete response; BOR = best overall response; DOR = duration of response; EQ-5D-3L = 3-level version of EQ-5D self-report questionnaire; EC = esophageal cancer; ECS = Esophagus Cancer Subscale; FACT-E = Functional Assessment of Cancer Therapy-Esophageal; FACT-Ga = Functional Assessment of Cancer Therapy-Gastric; GaCS = Gastric Cancer Subscale; GC = gastric cancer; IP = investigational product; RECIST = Response Evaluation Criteria in Solid Tumors; VAS = visual analog scale.

AEs and laboratory values will be graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

#### 5 STUDY DESIGN

## 5.1 Overall Design

This is a rolling, Phase 2, adaptive study that will evaluate the preliminary efficacy, safety, tolerability, PK, and pharmacodynamics of novel FRACTION-Gastric Cancer study treatment combinations in participants with advanced GC and/or EC. The details pertaining to the specific study treatment regimens are provided in each FRACTION-Gastric Cancer Sub-Protocol.

Protocol Amendment No.: 06

Participants will be enrolled in 1 of the 2 tracks. Participants who are anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment naïve will be enrolled for Track 1. Participants who have had prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment will be assigned to Track 2, as outlined in Figure 5.1-1 and described in Section 5.1.1.

Participants on Tracks 1 and 2 will begin on the Treatment Phase (with a total duration of approximately 2 years). Tumor assessments will be conducted according to the timing described in each FRACTION-Gastric Cancer Sub-Protocol.

Participants in Tracks 1 and 2 will be treated until completion of the Treatment Phase, progression, toxicity, or protocol-specified discontinuation (see Section 8.1). The decision to continue treatment beyond investigator-assessed progression is possible (for up to completion of that Treatment Phase) and should be discussed with the BMS Medical Monitor (or designee) and documented in the study records (see Section 7.4.2). In addition, a participant with PD has the option to enter into Track 2, assuming that he/she continues to fulfill all eligibility criteria at each new randomization point, including a life expectancy of  $\geq 3$  months (see Section 5.1.1).

A Simon 2-stage (optimal) design will be used in both Tracks 1 and 2 to evaluate the possibility of terminating an arm early and/or moving promising combinations into the next phase of treatment development (see Section 10.1). The number of participants planned for enrollment may vary by track and is described in Section 10.1. Enrollment will be continued after reaching the indicated number of participants at Stage 1 while the initial efficacy evaluation is ongoing. This will allow additional participants to enroll to account for unexpected trial impact, such as response nonevaluable participants due to early dropout, design parameter change (eg, historical rate update), etc. Participants who continue to fulfill eligibility criteria may move from Track 1 into Track 2 or re-enter Track 2, as described in Section 5.1.1.

The study design schematic is presented in Figure 5.1-1.



Figure 5.1-1: Study Design Schematic

Note: Participants treated with any study treatment targeting PD-1, PD-L1, or CTLA-4 will be considered anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment experienced, respectively.

Physical examinations, vital sign measurements, local 12-lead ECG, and clinical laboratory evaluations will be performed at selected times throughout treatment on all tracks (see Section 2 and the On-treatment Procedural Outline[s] specific to each FRACTION-Gastric Cancer Sub-Protocol). Participants will be closely monitored for AEs and SAEs throughout the study. Blood and tumor tissue will be collected at specified times before and after study treatment administration for PK, ADA, and pharmacodynamic analyses. Participants may withdraw or discontinue at any time based on criteria in Section 8.1.

## 5.1.1 FRACTION-Gastric Cancer Tracks 1 and 2 Design

A detailed study schematic for both Tracks 1 and 2 is presented in Figure 5.1.1-1.

Participants who are naïve to anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment will be enrolled in Track 1, and they will be randomized to nivolumab in combination with ipilimumab or to one of the FRACTION-Gastric Cancer study treatment combinations. These participants will receive their assigned study treatment in Track 1 until completion of the Treatment Phase.

Participants who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment will be enrolled in Track 2 and randomized to nivolumab in combination with ipilimumab, or to one of

the FRACTION-Gastric Cancer study treatment combinations. In addition, participants with PD who were treated in Track 1 or 2 and continue to fulfill all entry criteria may be enrolled in Track 2 and re-randomized to a new combination other than that previously received, if applicable. These participants will receive their assigned study treatment in Track 2 until completion of the Treatment Phase. The number of participants who initially enroll in Track 2 and those who enroll in Track 2 after treatment on Tracks 1 or 2 is described in Section 10.1.

- Participants with complete response (CR), PR, or SD at the end of 2 years on Track 1 or 2 Treatment Phase will:
  - Enter safety follow-up and complete FU1, FU2, and FU3 visits
- Participants with PD during the Track 1 or 2 Treatment Phase will:
  - Enter safety follow-up and complete FU1, FU2, and FU3 visits
- Participants with CR, PR, or SD who enter study follow-up and subsequently progress will:
  - Enter safety follow-up and complete FU1, FU2, and FU3 visits

Figure 5.1.1-1: Tracks 1 and 2 Study Design Schematic



Note: This diagram presents the protocol-mandated treatment flow for Tracks 1 and 2, including re-entry into Track 2.

Abbreviations: CR = complete response; RECIST = Response Evaluation Criteria in Solid Tumors.

Protocol Amendment No.: 06

Participants naïve to anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment will be enrolled in Track 1; participants with prior exposure to anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment will be enrolled in Track 2. Following track assignment, participants will be randomized.

b CR, PR, SD, and PD, as defined by RECIST v1.1. Assessments of PR and CR must be confirmed at least 4 weeks later following initial assessment.

<sup>&</sup>lt;sup>c</sup> Safety Follow-up Phase.

d Not applicable as of Protocol Amendment 06: If participants are eligible and if a new study treatment combination is available, they can enroll/re-randomize to a new combination.

e Not applicable as of Protocol Amendment 06: Each individual participant may receive multiple study treatments, including initial treatment, treatment beyond investigator-assessed progression, and/or entry into Track 2, assuming that the participant continues to fulfill all eligibility criteria at each new randomization point (see Section 5.1.3.2 for details).

Not applicable as of Protocol Amendment 06: Participants with PD during treatment may continue treatment beyond progression up to 2 years if criteria in Section 7.4.2 are met.

## 5.1.2 Safety Monitoring Board and Other External Committees

Two independent committees may be utilized: a Safety Monitoring Board (SMB) and an Independent Review Committee (IRC).

The SMB will be established to provide safety monitoring and to provide advice to the Sponsor regarding actions the committee deems necessary for the continuing protection of participants enrolled in the study. The SMB will meet at least twice per year concurrent with BMS internal continuous safety assessments. If needed, additional ad hoc SMB meetings may be convened. Safety-related data summaries and listings (by study track and study treatment arm, as appropriate) will be provided to SMB to facilitate safety monitoring. The SMB will act in an advisory capacity to BMS and will monitor participant safety throughout the study. Additional details are provided in the SMB Charter.

The IRC may be established at the discretion of the Sponsor. The IRC may review all available tumor assessment scans to determine response (Response Evaluation Criteria in Solid Tumors [RECIST] v1.1 criteria). IRC-determined response may be used in the analyses of ORR, PFSR, and duration of response (DOR).

### 5.1.3 Study Phases

Participants will complete up to 3 phases of the study: Screening, Treatment, and Safety Follow-up.

### 5.1.3.1 Screening

Prior to screening for the protocol, investigative sites are required to determine if a participant has previously received anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment through their institutional database, participant medical history, or institutional prescreening process. Once determined, treatment experience is considered source data for this FRACTION-Gastric Cancer study. The participant must be provided with the FRACTION-Gastric Cancer study Institutional Review Board (IRB)-approved written consent. Once the consent is signed, the participant is then considered to have entered screening. The treatment status must be entered into the enrollment management system, and participants will be required to submit a fresh tumor biopsy. An adequate baseline tumor biopsy (as determined by a central laboratory pathologist) must be obtained prior to randomization.

The Screening Phase for each track will last for up to 28 days. Participants will be enrolled using Interactive Response Technology (IRT).

If a participant surpasses the 28-day window during the Screening Phase due to a study-related procedure (eg, scheduling of a tumor biopsy or waiting time for a study-related laboratory value), the participant must be re-consented but does not need to be assigned a new participant identification number. To reduce any undue burden of procedure in this participant population in this situation, the amount of repeat procedures from the initial screening will be minimized, while maintaining safety and eligibility under the discretion of the BMS Medical Monitor (or designee) and investigator.

Enrollment in all study treatment arms in each track will be competitive.

Protocol Amendment No.: 06
## 5.1.3.2 Treatment

The details of the Treatment Phase duration are provided in Section 5.1. Further details of the study treatment administration are in each FRACTION-Gastric Cancer Sub-Protocol. Study assessments are to be collected as outlined in the On-treatment Procedural Outline(s) in each FRACTION-Gastric Cancer Sub-Protocol.

Assessment of response will be outlined for each combination therapy in the specific FRACTION-Gastric Cancer Sub-Protocol. Assessments of PR and CR must be confirmed at least 4 weeks later following initial assessment. Tumor progression or response endpoints will be assessed using RECIST v1.1 criteria for solid tumors (see Appendix 5).

Participants will generally be allowed to continue study treatment until the first occurrence of one of the following: 1) completion of 2 years of study treatment, 2) PD, 3) clinical deterioration suggesting that no further benefit from study treatment is likely, 4) intolerable toxicity, and 5) meeting of criteria for discontinuation of study treatment, as outlined in Section 8.1. Individual participants with confirmed CR will be given the option to discontinue study treatment, on a case-by-case basis, after specific consultation and agreement between the investigator and the BMS Medical Monitor (or designee) in settings where the benefit/risk ratio justifies discontinuation of study treatment.

All participants will be treated as per Section 5.1, unless criteria for study treatment discontinuation are met earlier (see Section 8.1 in this FRACTION-Gastric Master Protocol and Section 8.1 in the FRACTION-Gastric Cancer Sub-Protocol). Upon completion of the Treatment Phase, all participants will enter the Safety Follow-up Phase (see Section 5.1.3.3 and Table 2-3).

As of Protocol Amendment 06, collection of blood or other biological samples for reasons other than safety monitoring (eg, PK, ADA, biomarkers, etc) should be discontinued. Please refer to Table 2-3 and Sections 9.5, 9.6, and 9.8.

## 5.1.3.3 Follow-up

As of Protocol Amendment 06, tumor scans, survival status follow-ups, and collection of subsequent treatment information will end once the participant has disease progression or treatment discontinuation for any reason, whichever occurs first. Any assessments for monitoring of safety will continue per protocol until the final follow-up visit (FU3). Please refer to Table 2-3.

## **Safety Follow-up**

Upon completion of the Treatment Phase, all participants will enter the Safety Follow-up Phase once the decision is made to discontinue the participant from study treatment (eg, at EOT).

For participants that complete all scheduled weeks of study treatment, EOT visit will be the same as the last scheduled and completed on-treatment visit and the start of Week 1 safety follow-up visit. For participants that do not complete all scheduled weeks of study treatment, EOT visit will be the most recent on-treatment visit (with all available safety and response data; does not need to be repeated) and will be considered the start of Week 1 safety follow-up visit.

Protocol Amendment No.: 06

Date: 13-Aug-2021

After the EOT visit, all participants will be evaluated for any new AEs until 100 days following the last dose of study treatment, as specified in each FRACTION-Gastric Cancer Sub-Protocol. All SAEs must be collected from the date of the participant's written consent until 100 days post discontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. Follow-up visits should occur at Days 30, 60, and 100 ( $\pm$  7 days) after the last dose of study treatment or coinciding with the date of discontinuation ( $\pm$  7 days), if the date of discontinuation is greater than 30 days after the last dose, to monitor for AEs. All participants will be required to complete the 3 clinical safety follow-up visits, regardless of whether they start a new anti-cancer treatment, except for those participants who withdraw consent for study participation or those participants who start retreatment or are re-randomized into Track 2.

## 5.2 Number of Participants

For Sub-Protocols utilizing a Simon-2 stage (optimal) design, up to 54 anti-PD1/PD-L1 or CTLA-4 treatment-naïve participants will be treated per study treatment combination, in Track 1. In Track 2, up to 41 participants will be treated per study treatment combination (see Section 10.1 for details).

For Sub-Protocols not utilizing a Simon-2 stage (optimal) design, a different sample size may be used depending on the statistical considerations for those treatment combinations. In those cases, sample size will be discussed within the individual Sub-Protocols.

## 5.3 End of Study Definition

The start of the study is defined as first visit for first participant screened. End of study is defined as the last visit or scheduled procedure shown in the Schedule of Activities for the last participant. Study completion is defined as the final date on which data for the primary endpoint was or is expected to be collected, if this is not the same.

# 5.4 Scientific Rationale for Study Design

BMS has an extensive portfolio of novel agents that span a variety of targets. To determine which combinations show the most clinical promise and, thus, should be prioritized for future registrational studies, BMS has initiated the FRACTION Program. The FRACTION Program will treat participants with different study treatment options and employ repeat blood sampling, tumor biopsies, and serial assessments to understand markers of response to treatment. These approaches are supported by various precedent studies that use innovative trial designs to quickly assess new agents in participants, with the goal of reducing the time and number of participants required to bring these treatments to those who will benefit from them. For the FRACTION Program, specific study treatment combinations and/or control treatments will be introduced in FRACTION Sub-Protocols for each FRACTION study. Study treatment combinations that have high potential to produce transformational activity in the cancer compared to the control, based on both preclinical and early clinical trials data, will be selected. See Section 3.1 for details.

Protocol Amendment No.: 06

Date: 13-Aug-2021

# 5.4.1 Rationale for Duration of Therapy

The optimal duration of immunotherapy is an important question and continues to be investigated. In Study CA209153, patients with previously treated advanced NSCLC who completed 1 year of nivolumab therapy were randomized to either continue or stop treatment, with the option of retreatment upon progression. Among 163 patients still on treatment at 1 year and without progression, those who were randomized to continue nivolumab had significant improvement in progression-free survival (PFS) compared to those who were randomized to stop treatment, with median PFS (post-randomization) not reached vs 10.3 months, respectively; hazard ratio (HR) = 0.42 (95% CI, 0.25 to 0.71). With a median follow-up of 14.9 months post-randomization, there also was a trend for patients on continued treatment to live longer (OS HR = 0.63 [95% CI: 0.33, 1.20]). Of note, the PFS curves in both groups plateau approximately 1 year after randomization (ie, 2 years after treatment initiation), suggesting that there may be minimal benefit in extending treatment beyond a total of 2 years. <sup>51</sup>

Moreover, accumulating data suggest that 2 years of PD-1 checkpoint inhibitor treatment may be sufficient for long-term benefit. In Study CA209003, a dose-escalation cohort expansion trial evaluating the safety and clinical activity of nivolumab in patients with previously treated advanced solid tumors (including 129 participants with NSCLC) specified a maximum treatment duration of 2 years. Among 16 participants with NSCLC who discontinued nivolumab after completing 2 years of treatment, 12 participants were alive > 5 years and remained progression-free without any subsequent therapy. In the CA209003 NSCLC cohort, the OS curve begins to plateau after 2 years, with an OS rate of 25% at 2 years and 18% at 3 years. These survival outcomes are similar to Phase 3 studies in previously treated NSCLC, in which nivolumab treatment was continued until progression or unacceptable toxicity (2-year OS rates of 23% and 29%, and 3-year OS rates of 16% to 18% for squamous and non-squamous NSCLC, respectively). Sa

Taken together, the data suggest that a shorter duration of nivolumab treatment of only 1 year was associated with increased risk of progression in previously treated patients with NSCLC, suggesting that treatment beyond 1 year is likely needed. Also, treatment beyond 2 years is unlikely to confer additional clinically meaningful benefit, and that the risk of progression after discontinuing treatment at 2 years is low.

Collectively, these data suggest that there is minimal, if any, benefit derived from continuing IO treatment beyond 2 years in advanced tumors. However, even though immunotherapy is well tolerated, patients will be at risk for additional toxicity with longer-term treatment.

#### 5.5 Justification for Dose

Please refer to individual FRACTION-Gastric Cancer Sub-Protocols for their respective dose justifications.

## 6 STUDY POPULATION

For entry into the FRACTION-Gastric Cancer study (per FRACTION-Gastric Cancer Master Protocol), the following criteria must be met prior to dosing on Day 1. For entry into a study

Protocol Amendment No.: 06

Date: 13-Aug-2021

treatment per a FRACTION-Gastric Cancer Sub-Protocol, additional treatment-specific criteria, if applicable, must also be met.

No exceptions will be granted.

#### 6.1 Inclusion Criteria

## 1) Signed Written Informed Consent

- a) Participants must be able to give self-consent and then sign and date an IRB/Independent Ethics Committee (IEC)-approved written informed consent in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not considered part of normal patient care.
- b) Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
- c) Participants must provide consent for mandatory tumor biopsy samples (as detailed in "20" below).

#### 2) Type of Participant and Target Disease Characteristics

- a) All participants must have inoperable, advanced, or metastatic EC, GC or GEJ carcinoma and have histologically confirmed predominant adenocarcinoma and/or squamous carcinoma. The documentation of GEJ involvement can include biopsy, endoscopy, or imaging.
- b) Participants with human epidermal growth factor receptor 2 (HER2) overexpressing tumor who progress after trastuzumab (or are ineligible for or unwilling to be treated with trastuzumab) are eligible to be enrolled.
- c) Prior adjuvant or neoadjuvant chemotherapy, radiotherapy, and/or chemoradiotherapy are permitted, as long as the last administration of the last regimen (whichever was given last) occurred at least 4 weeks prior to randomization.
- d) Participants must have an Eastern Cooperative Oncology Group performance status  $\leq 1$  (see Appendix 7).
- e) Track-specific eligibility criteria
  - i) Track 1: anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment-naïve participants
    - (1). Participants must not have received any anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment prior to this study. Participants previously treated with agents other than anti-PD-1, anti-PD-L1, or anti-CTLA-4 are eligible for Track 1.
    - (2). Participants may have been offered platinum-based chemotherapy for progressive or recurrent disease.
      - a. The platinum-based chemotherapy may have been in the adjuvant, neoadjuvant, or recurrent setting.
    - (3). Not Applicable per Amendment 02.
    - (4). Not Applicable per Amendment 03.

- (5). All participants must consent to the acquisition of fresh pre- and on-treatment tumor biopsies for performance of correlative biomarker studies. Archival specimens may not be substituted for fresh baseline specimens but can be submitted to help understand the evolution of the tumor (ie, PD-L1 expression changes over time) for performance of correlative studies. Participants who either do not consent to a pre-treatment tumor biopsy or do not have accessible lesions are not eligible. An adequate baseline tumor biopsy as determined by a central laboratory pathologist must be obtained prior to randomization. If fresh biopsy is not clinically feasible or safe, the option of archival tissue can be discussed with BMS if the biopsy was obtained within 90 days of study enrollment and there was no intervening systemic anticancer or IO therapy.
- ii) Track 2: anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment-experienced participants
  - (1). Participants must have had progressive or recurrent disease during or after anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment. (Participants treated with any study treatment targeting PD-1, PD-L1, or CTLA-4 will be considered anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment experienced, respectively).
  - (2). Participants may have been offered platinum-based chemotherapy for GC or GEJ.
    - a. The platinum-based chemotherapy may have been in the adjuvant, neoadjuvant, or recurrent setting.
  - (3). Participants who have had prior treatment with any 1 of the agents (or any other agent targeting PD-1, PD-L1, or CTLA-4) in monotherapy or in any combination regimen in a FRACTION-Gastric Cancer Sub-Protocol are eligible for treatment on Track 2.
  - (4). Participants who have had prior combination treatment with the same IO combination agents (or IO agents directed against the same targets) as 1 of the combination regimens in a FRACTION-Gastric Cancer Sub-Protocol are eligible for study treatment on Track 2 but must be randomized to another combination regimen (as outlined in Section 5.1.1 Inclusion Criteria of each FRACTION-Gastric Cancer Sub-Protocol).
  - (5). All participants must consent to the acquisition of fresh pre- and on-treatment tumor biopsies for performance of correlative biomarker studies. Archival specimens may not be substituted for fresh baseline specimens but can be submitted to help understand the evolution of the tumor (ie, PD-L1 expression changes over time) for performance of correlative studies. Participants who either do not consent to a pre-treatment tumor biopsy or do not have accessible lesions are not eligible. An adequate baseline tumor biopsy as determined by a central laboratory pathologist must be obtained prior to randomization. If fresh biopsy is not clinically feasible or safe, the option of archival tissue can be discussed with BMS if the biopsy was obtained within 90 days of study enrollment and there was no intervening systemic anticancer or IO therapy.
- f) At the time of screening, participants must have a life expectancy of at least 3 months following their most recent chemotherapy or immunotherapy for entry into all tracks.

- i) Participants who wish to be re-randomized to a new study treatment combination on Track 2 following progression on a prior study treatment in Tracks 1 or 2 must have a life expectancy of at least 3 months following the last study treatment.
- g) Participants receiving prior palliative radiotherapy to a non-central nervous system (CNS) lesion must have completed that treatment at least 2 weeks prior to the first dose of study treatment.
  - i) Participants with symptomatic tumor lesions at baseline who may require palliative radiotherapy within 4 weeks of the first dose of study treatment are strongly encouraged to receive palliative radiotherapy prior to enrollment, and they must complete that treatment at least 2 weeks prior to the first dose of study treatment.
- h) Participants must have at least 1 lesion with measurable disease, as defined by RECIST v1.1 criteria for solid tumors response assessment (see Appendix 5).
  - i) Participants with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll, provided that the lesion(s) have demonstrated clear progression and can be measured accurately.
- i) Participants with toxicity from any prior anti-cancer treatment must have their toxicity returned to Grade ≤ 1 (NCI CTCAE Version 4.03) or baseline before administration of study treatment.
  - i) Participants with Grade ≥ 2 toxicities attributed to prior anti-cancer treatment that are not expected to resolve and result in long-lasting sequelae, such as neuropathy after a platinum based- treatment, are eligible.
  - ii) Grade >1 alopecia or fatigue is permitted.
- j) Not applicable as per revised protocol 03 Participants must allow a tumor biopsy at the following time points: 1) baseline (prior to study treatment); 2) on-study (Day 28 on-treatment); and 3) EOT, defined as at the time of progression or at the time of a clinically significant event (eg, at EOT for participants with PR or SD or at EOT for participants who discontinue treatment due to an AE), provided that the biopsy is at acceptable clinical risk as judged by the investigator for each study treatment regimen to 1) identify predictive biomarkers for both safety and efficacy of a given combination, 2) define the mechanism of action for a particular combination (pharmacodynamic assessment), and 3) determine the mechanisms of resistance to a particular combination.
  - i) Participants who do not have accessible or suitable lesions are not eligible.
    - (1). Baseline biopsies may be collected from participants with a single measurable lesion (primary or metastatic), as long as it is not an excisional biopsy.
  - ii) For participants whose pretreatment biopsy yields inadequate tissue quantity or quality (as determined by a pathologist in the central laboratory), re-biopsy is permitted.
  - iii) The solid tumor tissue specimen must be a core-needle, biopsy or an excisional or incisional biopsy. Fine-needle biopsies and drainage of pleural effusions with cytospins are not considered adequate for biomarker review and randomization. Biopsies of bone lesions that do not have a soft tissue component or decalcified bone tumor samples are also not acceptable.

- (1). Punch biopsies are acceptable as long as adequate tumor material is provided.
- iv) The biopsy at progression of disease after treatment on any track may function as the pretreatment biopsy for subsequent treatment on Track 2.
- k) Study personnel must ensure that the archival tissue block (preferred) or slides samples, if available, are located and shipped to the central laboratory prior to randomization within 6 weeks of signing the written informed consent, as long as this tissue will not be used for the screening biopsy sample.
- l) Participants must have adequate organ function, as defined by the following:
  - i) White blood cells  $\geq 2,000/\mu L$  (stable off any growth factor after discontinuation within 2 weeks of the first study treatment administration)
  - ii) Neutrophils  $\geq 1,500/\mu L$  (stable off any growth factor after discontinuation within 2 weeks of the first study treatment administration)
  - iii) Platelets  $\geq 100 \times 10^3 / \mu L$  (transfusion to achieve this level is not permitted within 2 weeks of the first study treatment administration)
  - iv) Hemoglobin  $\geq 9.0$  g/dL (transfusion to achieve this level is not permitted within 2 weeks of the first study treatment administration)
  - v) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)  $\leq 3 \times$  institutional upper limit of normal (ULN)
  - vi) Total bilirubin  $\leq 1.5 \times$  institutional ULN (except for participants with Gilbert's syndrome who must have normal direct bilirubin)
  - vii) Serum creatinine ≤ 1.5× institutional ULN or creatinine clearance (CrCl) ≥ 40 mL/min (measured using the Cockcroft-Gault formula below):

Female CrCl =  $\frac{(140 - \text{age in years}) \times \text{weight in kg} \times 0.85}{72 \times \text{serum creatinine in mg/dL}}$ Male CrCl =  $\frac{(140 - \text{age in years}) \times \text{weight in kg} \times 1.00}{72 \times \text{serum creatinine in mg/dL}}$ 

- m) Participants must be able to comply with restrictions and prohibited activities/treatments listed in Section 7.7.1.
- n) Participant re-enrollment: This study permits the re-enrollment of a participant who has discontinued the study as a pretreatment failure (eg, participant has not been treated). If re-enrolled, the participant must be re-consented.
- o) Participants must allow a tumor biopsy at baseline and on study.
  - i) Participants who do not have accessible or suitable lesions are not eligible.
  - ii) For participants whose pretreatment biopsy yields inadequate tissue quantity or quality (as determined by a pathologist in the central laboratory), re-biopsy is permitted.
  - iii) The solid tumor tissue specimen must be a core-needle, biopsy or an excisional or incisional biopsy. Fine-needle biopsies and drainage of pleural effusions with cytospins

are not considered adequate for biomarker review and randomization. Biopsies of bone lesions that do not have a soft tissue component or decalcified bone tumor samples are also not acceptable.

- (1). Punch biopsies are acceptable as long as adequate tumor material is provided.
- iv) The biopsy at progression of disease after treatment on any track may function as the pretreatment biopsy for subsequent treatment on Track 2.

## 3) Age and Reproductive Status

- a) Males and females, ages 18 years or older at the time of consent
- b) Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment. An extension up to 72 hours prior to the start of study treatment is permissible in situations where results cannot be obtained within the standard 24-hour window.
- c) Women must not be breastfeeding.
- d) WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) plus the time required for the study treatment to undergo approximately 5 half-lives, plus the duration of 1 ovulatory cycle (30 days), for a total of 5 months posttreatment completion (see Appendix 4). If the half-life of a study treatment in a FRACTION-Gastric Cancer Sub-Protocol is longer than approximately 5 half-lives of nivolumab, this will be addressed in the FRACTION-Gastric Cancer Sub-Protocol.
  - i) WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements and still must undergo pregnancy testing, as described in this section.
- e) Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception and fetal protection (see Appendix 4) for the duration of treatment with study treatment(s) plus approximately 5 half-lives of the study treatment, plus the duration of sperm turnover (90 days), for a total of 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
  - i) *Not applicable as per revised protocol 03* Azoospermic males are exempt from contraceptive requirements.

Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy and when applicable, the potential of fetal toxicity occurring due to transmission of study drug, present in seminal fluid, to a developing fetus, even if the participant has undergone a successful vasectomy or if the partner is pregnant. Investigators shall advise on the use of highly effective methods of contraception (Appendix 4), which have a failure rate of < 1% when used consistently and correctly.

#### 6.2 Exclusion Criteria

## 1) Medical Conditions

- a) Participants with HER2-positive tumor and previously untreated with trastuzumab are excluded; participants who are ineligible for or unwilling to be treated with trastuzumab are still eligible.
- b) Participants with ascites that cannot be controlled with appropriate interventions.
- c) Participants must not have suspected, known, or progressive CNS metastases; have untreated CNS metastases; or have the CNS as the only site of disease.
  - i) Participants are eligible if CNS metastases are adequately treated and participants neurologically return to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to study entry. In addition, participants must be either off corticosteroids or on a stable or decreasing dose of prednisone ≤ 10 mg daily (or equivalent) for at least 2 weeks prior to study entry.
  - ii) Participants must not have leptomeningeal disease or carcinomatous meningitis.
- d) Participants must not have prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
- e) Participants must not have other active malignancy requiring concurrent intervention.
- f) Participants must not have received a prior organ allograft.
- g) Participants must not have received any anti-cancer treatment (eg, chemotherapy or radiotherapy [except for palliative radiotherapy, which can be received at least 2 weeks prior to study treatment]; biologics; or immunotherapies, including investigational treatments) within 4 weeks prior to the first dose of study treatment administration.
  - i) Participants who have received noncytotoxic anti-cancer therapies (eg, prior use of targeted treatment) and who have completed treatment at least 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study treatment are eligible to enroll. However, if 5 half-lives is shorter than 4 weeks, agreement with the BMS Medical Monitor (or designee) is mandatory.
- h) Participants must not have active, known, or suspected autoimmune disease.
  - i) Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement treatment, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
- i) Participants must not have a condition requiring systemic treatment with either corticosteroids (prednisone > 10 mg daily or equivalent) or other immunosuppressive medications within 14 days of study treatment administration.
  - i) Inhaled or topical steroids and adrenal replacement steroid (prednisone > 10 mg daily or equivalent) are permitted in the absence of active autoimmune disease.

- j) Participants must not have a history of life-threatening toxicity related to prior IO treatment (eg, anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or treatment specifically targeting T-cell co-stimulation or immune checkpoint pathways).
  - i) Participants with toxicities that are unlikely to recur with standard countermeasures (eg, hormone replacement treatment after adrenal crisis) are eligible.
- k) Participants must not have interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
- 1) Participants must not have uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:
  - i) Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  - ii) Uncontrolled angina within the past 3 months
  - iii) Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  - iv) QT interval corrected with Fridericia's formula ≥ 480 ms
  - v) History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, myocarditis, pericarditis, or significant pericardial effusion)
- m) Participants who require daily supplemental oxygen treatment are excluded.
- n) Participants must not have any positive test result for hepatitis B virus or hepatitis C virus (HCV) indicating presence of virus, for example, hepatitis B surface antigen (Australia antigen) positive or hepatitis C antibody (anti-HCV) positive (except if HCV-ribonucleic acid [RNA] negative).
  - i) Participants with a history of resolved hepatitis A virus infection are eligible.
- o) Participants must not have evidence of active infection requiring antibacterial, antifungal, or antiviral treatment  $\leq 7$  days prior to initiation of study treatment.
- p) Participants must not have a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
  - i) Testing for HIV must be performed at sites mandated by local requirements. (For sites in Germany, see Appendix 8.)
- q) Participants must not have known or suspected active tuberculosis.
- r) Participants must not have had any major surgery within 4 weeks of study treatment administration. Participants must have recovered from the effects of a major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
- s) Participants must not have received nononcology vaccines containing live virus for prevention of infectious diseases within 12 weeks prior to the first dose of study treatment.
  - i) The use of inactivated seasonal influenza vaccines (eg, Fluzone<sup>®</sup>) will be permitted on study without restriction.
- t) Participants must not have received packed red blood cell or platelet transfusion within 2 weeks prior to the first dose of study treatment.

u) Participants must not have a known or underlying serious or uncontrolled medical condition that, in the opinion of the investigator or Sponsor, could make the administration of study treatment hazardous to the participants or could adversely affect the ability of the participant to comply with or tolerate the study.

## 2) Allergies and Adverse Drug Reaction

- a) History of any significant treatment allergy (such as anaphylaxis or hepatotoxicity) to prior anti-cancer immune-modulating therapies (eg, checkpoint inhibitors and T-cell co-stimulatory antibodies).
- b) History of allergy or hypersensitivity to study treatment components.

## 3) Other Exclusion Criteria

- a) Prisoners or participants who are involuntarily incarcerated. Note: Under certain specific circumstances, and only in countries where local regulations permit, a person who has been imprisoned may be included or permitted to continue as a participant. Strict conditions apply, and BMS approval is required.
- b) Participants who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

# 6.3 Lifestyle Restrictions

Not applicable. No restrictions are required.

#### 6.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomized. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes date of consent, demography, screen failure details, eligibility criteria, and any serious AEs.

## 6.4.1 Retesting During Screening

Participant Re-enrollment: This study permits the re-enrollment of a participant that has discontinued the study as a pretreatment failure (ie, participant has not been randomized or has not been treated). If re-enrolled, the participant must be re-consented.

Retesting of laboratory parameters and/or other assessments within any single Screening Phase will be permitted (in addition to any parameters that require a confirmatory value).

The most current result prior to randomization is the value by which study inclusion will be assessed, as it represents the participant's most current, clinical state.

Laboratory parameters and/or assessments that are included in Table 2-1, Screening Procedural Outline, may be repeated in an effort to find all possible well-qualified participants. Consultation

Protocol Amendment No.: 06

with the BMS Medical Monitor (or designee) may be needed to identify whether repeat testing of any particular parameter is clinically relevant.

#### 7 TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device intended to be administered to a study participant according to the study randomization or treatment allocation.

Study treatment includes both Investigational [Medicinal] Product (IP/IMP) and Non-IP/Non-IMP and is described in each FRACTION-Gastric Cancer Sub-Protocol.

An IP, also known as IMP in some regions, is defined as a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently from the authorized form, used for an unauthorized indication, or used to gain further information about the authorized form.

Other medications used as support or escape medication for preventive, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as non-IPs.

#### 7.1 Treatments Administered

Other treatments administered as part of the study that are critical to claims of efficacy (eg, background treatment and rescue medications) will be considered study treatment. A table describing the study treatments and dosage information is provided in each FRACTION-Gastric Cancer Sub-Protocol.

## 7.2 Method of Treatment Assignment

This is an open-label study. All participants will be centrally randomized using an IRT. Before the study is initiated, each user will receive log-in information and directions on how to access the IRT.

Specific study treatments are listed in each FRACTION-Gastric Cancer Sub-Protocol. Study treatment will be dispensed at the study visits, as listed in the On-treatment Procedural Outline(s) in each FRACTION-Gastric Cancer Sub-Protocol.

All participants must be assigned a patient identification number (PID) upon providing a signed IRB/IEC-approved written informed consent. During the screening visit, the investigative site will utilize the IRT for enrollment and receive a 5-digit PID designated by BMS that will be unique across all sites. Enrolled participants, including those not dosed, will be assigned sequential PIDs starting with \_\_\_\_\_\_\_\_\_. The PID will ultimately be composed of the site number and participant number. For example, the first participant screened (eg, enrolled) at Site Number 1 will have a PID of \_\_\_\_\_\_\_\_. The following information is required for enrollment:

- Date of obtaining informed consent
- Date of birth

Protocol Amendment No.: 06

930104678 8.0

Approved v 8.0

- Gender at birth
- Anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment experience (see Section 5.1.3.1)

Once enrolled in the IRT, participants who meet all eligibility criteria will be ready to be randomized through the IRT. The following information is required for randomization:

- Participant number
- Date of birth

Randomization participant schedules will be generated and maintained by the IRT vendor. At the conclusion of the trials, BMS will receive copies of all generated participant schedules from the vendor. Because of the nature of the study design, limited early access to the randomization information will be granted to the study team to facilitate early analyses for internal decision making (early termination of study treatment arm, etc).

Each participant who is randomized will be assigned a unique randomization number. This is not the primary identifier for the participant, but is used for the randomization schedule. The primary identifier will be the PID described above, for use on the case report form (CRF) and source documents. A participant being re-randomized in Track 2 will be assigned a different randomization number but will retain the same PID. Randomization numbers will be assigned using a Central Randomization System in the order in which participants qualify for study treatment, not in the order of study enrollment. Randomization ratios within each track will be specified in each FRACTION-Gastric Cancer Sub-Protocol. If, within a given track, study treatment arms from more than 1 FRACTION-Gastric Cancer Sub-Protocol within the FRACTION-Gastric Cancer Master Protocol are simultaneously open to enrollment, then a new participant could be assigned to any of the open study treatment arms. In Track 1, participants will be randomized to newly added study treatment arms/study treatments (through FRACTION-Gastric Cancer Sub-Protocols) in a ratio specified in each new FRACTION-Gastric Cancer Sub-Protocol. New randomization schedules for new FRACTION-Gastric Cancer Sub-Protocols will be generated. If accrual for current FRACTION-Gastric Cancer Sub-Protocols is still ongoing, participants will be allocated to the existing randomization schedule or new randomization schedule based on a pre-specified allocation ratio. Details of allocation ratio will be specified in the new FRACTION-Gastric Cancer Sub-Protocol. In Track 2, participants will be randomized to existing study treatment arm/study treatments and newly added study treatment arm/study treatments with equal probability.

Pre-specified study treatment arm caps (according to Simon 2-stage [optimal] design) will be utilized to control the accrual for each study treatment combination arm under different tracks (Tracks 1 and 2). The cap for the nivolumab in combination with ipilimumab control arm under Track 1 will be set equal to the largest cap among its corresponding experimental arms. In the event that 1 or more participants go off study without being evaluable for response (ie, with no post-baseline tumor measurements and no evidence of clinical progression or death due to disease progression), the enrollment cap for that study treatment arm may be correspondingly raised if

needed to ensure that a sufficient number of evaluable participants are available for decision making according to the Simon 2-stage (optimal) design. If the decision is made to close any study treatment arm for safety concerns, the cap for that study treatment arm will be reduced to the current number of participants already randomized. Accrual will be stopped immediately. Enrollment caps to Track 2 based on new participants or re-randomized participants are described in Section 10.1.2.

Specific instructions for randomization into the Central Randomization System will be provided in a separate manual.

## 7.3 Blinding

This is an open-label study; blinding procedures are not applicable.

# 7.4 Dosage Modification

Specific dosing and treatment regimens for each FRACTION-Gastric Cancer study treatment combination and/or nivolumab in combination with ipilimumab are outlined in each FRACTION-Gastric Cancer Sub-Protocol.

## 7.4.1 Dose Reductions and Delays and Criteria to Resume Dosing

Tumor assessments for all participants should continue as per protocol even if dosing is delayed.

Guidelines for dose reductions and delays due to toxicity and for resuming study treatment for each FRACTION-Gastric Cancer study treatment combination are provided in the FRACTION-Gastric Cancer Sub-Protocols.

# 7.4.2 Treatment Beyond Disease Progression

Not applicable per Protocol Amendment 06.

# 7.4.3 Management Algorithms for IO and Oncology Agents

IO agents are associated with AEs that can differ in severity and duration from AEs caused by other therapeutic classes. Early recognition and management of AEs associated with IO agents may mitigate severe toxicity. Management algorithms have been developed from extensive experience with nivolumab, ipilimumab, and their combination to assist investigators in assessing and managing the following groups of AEs:

- Pulmonary
- Gastrointestinal
- Hepatic
- Endocrinopathies
- Renal
- Skin
- Neurological

The clinical nature of AEs noted with each FRACTION-Gastric Cancer study treatment combination and/or nivolumab in combination with ipilimumab will determine the role of the algorithms above for use in toxicities related to its use in this study.

The management algorithms recommended for utilization for IO and non-IO agents are included in Appendix 6 and in each FRACTION-Gastric Cancer Sub-Protocol.

#### 7.4.4 Treatment of Treatment-related Infusion Reactions

Guidelines for the treatment of study treatment-related infusion reactions for each FRACTION-Gastric Cancer study treatment combination are provided in each FRACTION-Gastric Cancer Sub-Protocol describing that treatment combination.

# 7.5 Preparation/Handling/Storage/Accountability

The IP should be stored in a secure area according to local regulations. It is the responsibility of the investigator to ensure that IP is only dispensed to study participants. The IP must be dispensed only from official study sites by authorized personnel according to local regulations.

The product storage manager should ensure that the study treatment is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study treatment arise, the study treatment should not be dispensed and BMS should be contacted immediately.

Study treatment not supplied by BMS will be stored in accordance with the package insert.

IP documentation (whether supplied by BMS or not) must be maintained that includes all processes required to ensure study treatment is accurately administered. This includes documentation of study treatment storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg, required diluents and administration sets).

For study treatments not provided by BMS and obtained commercially by the site, storage should be in accordance with the product label. Infusion-related supplies (eg, intravenous bags, in-line filters, and 0.9% NaCl solution) will not be supplied by the Sponsor and should be purchased locally if permitted by local regulations.

Storage facilities for controlled substances must be securely locked and substantially constructed, with restricted access to prevent theft or diversion, as applicable by local regulations.

• Further guidance and information for final disposition of unused study treatment are provided in Appendix 2 and the Pharmacy Manual.

# 7.5.1 Retained Samples for Bioavailability / Bioequivalence / Biocomparability

Not applicable.

Protocol Amendment No.: 06

# 7.6 Treatment Compliance

Study treatment will be administered in the clinical facility by trained medical personnel. Treatment compliance will be monitored by treatment accountability, as well as by recording administration of each study treatment in the participants' medical records and CRF.

# 7.7 Concomitant Therapy

#### 7.7.1 Prohibited and/or Restricted Treatments

The following prohibitions and restrictions apply to all FRACTION-Gastric Cancer Sub-Protocols for the FRACTION-Gastric Cancer study. Additional FRACTION-Gastric Cancer Sub-Protocolspecific prohibitions and/or restrictions are outlined in each FRACTION-Gastric Cancer Sub-Protocol.

The following medications are prohibited during the Treatment Phase of the study:

- 1) Immunosuppressive agents (except for those stated in Section 7.7.3) are prohibited unless they are utilized to treat an AE.
- 2) Chronic systemic corticosteroids (prednisone > 10 mg daily or equivalent; except for those stated in Section 7.7.3) are prohibited unless they are utilized to treat an AE.
- 3) Vaccines (except for those stated in Section 7.7.3) are prohibited.
- 4) Any medicinal herbal preparations within 2 weeks prior to the first dose of study treatment are prohibited unless prescribed by a treating physician. Use of marijuana and its derivatives for treatment of symptoms related to cancer treatment are permitted if obtained by medical prescription or if its use (even without a medical prescription) has been legalized locally, as long as no drug-drug interactions are outlined in the specific Sub-Protocol.
- 5) Any concurrent anti-neoplastic treatment (ie, chemotherapy; immunotherapy; extensive, nonpalliative radiation treatment; or standard or investigational agents for treatment of GC/GEJ) is prohibited other than those included in the study treatment combinations.

Any concomitant therapies must be recorded on the CRF from screening to follow-up.

#### 7.7.2 Other Restrictions and Precautions

# 7.7.2.1 Imaging Restriction and Precautions

It is the local imaging facility's responsibility to determine, based on participant attributes (eg, allergy history, diabetic history, and renal status), the appropriate imaging modality and contrast regimen for each participant. Imaging contraindications and contrast risks should be considered in this assessment. Participants with renal insufficiency should be assessed as to whether or not they should receive contrast and, if so, what type and dose of contrast are appropriate. Magnetic resonance imaging (MRI) contrast should not be given to participants with severe renal insufficiency (eg, estimated glomerular filtration rate < 30 mL/min/1.73 m<sup>2</sup>) because of increased risk of nephrogenic systemic fibrosis in this participant population. In these participants, alternative imaging tests or MRI without gadolinium should be considered. In addition, participants are excluded from MRI if they have tattoos, metallic implants, pacemakers,

etc. The ultimate decision to perform MRI in an individual participant in this study rests with the site radiologist, the investigator, and the standard set by the local IRB/IEC.

# 7.7.3 Permitted Therapy

Participants are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course (less than 3 weeks) of corticosteroids prophylaxis (eg, contrast dye allergy) or for treatment of nonautoimmune conditions (eg, delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.

- Inhaled or intranasal corticosteroids (with minimal systemic absorption may be continued if
  the participant is on a stable dose) and adrenal replacement steroid doses of prednisone
  > 10 mg daily or equivalent are permitted in the absence of active autoimmune disease. Nonabsorbed intra-articular steroid injections will be permitted.
- Immunosuppressive agents and the use of systemic corticosteroids are permitted in the context of treating AEs. Participants receiving corticosteroids must be at prednisone < 10 mg daily or equivalent prior to re-initiation of study treatment. Participants may continue to receive hormone replacement treatment.
- The inactivated seasonal influenza vaccine can be given to participants while on treatment without restriction. Vaccines containing live/attenuated virus (e.g., varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella [MMR]) are not permitted while on study treatment and until 100 days post the last dose.
- Non-live COVID-19 vaccination is considered a simple concomitant medication within the study. However, the efficacy and safety of non-live vaccines (including non-live COVID-19 vaccines) in participants receiving investigational agents is unknown.

# 7.7.4 Palliative Local Therapy

Palliative and supportive care for disease-related symptoms may be offered to all participants on the study. Limited radiation treatment or surgery to control isolated lesions is permitted for participants who have investigator-assessed clinical benefit following consultation with the BMS Medical Monitor (or designee).

Participants should not receive study treatment during radiation because the potential for overlapping toxicities with radiotherapy and FRACTION-Gastric Cancer study treatment combinations or nivolumab in combination with ipilimumab is not known. If palliative radiotherapy in short courses and for isolated fields is required to control symptoms not clearly related to disease progression, then study treatment administration should be withheld, if possible, for at least 1 week before radiation and for at least 1 week after its completion. Participants should be closely monitored for any potential toxicity during and after receiving radiotherapy. Prior to resuming study treatment, radio-therapy related- AEs should resolve to Grade ≤ 1 or baseline, and participants must meet relevant eligibility criteria as determined by the BMS Medical Monitor (or designee) in discussion with the investigator. The BMS Medical Monitor (or designee) must be consulted prior to re-initiating study treatment in a participant with a dosing delay lasting > 8 weeks from the previous dose.

Protocol Amendment No.: 06

Details of palliative radiotherapy should be documented in the source records and electronic case report form (eCRF). Details in the source records should include dates of treatment, anatomic site, dose administered and fractionation schedule, and AEs. Symptoms requiring palliative radiotherapy should be evaluated for objective evidence of disease progression. Participants receiving palliative radiation of target lesions will have the evaluation of ORR just prior to radiotherapy, but these participants will no longer be evaluable for the determination of response subsequent to the date palliative radiation occurs.

For participants who need to undergo elective surgery (not tumor related) during the study, it is recommended to hold study treatment(s) for at least 2 weeks before and 2 weeks after surgery, or until the participant recovers from the procedure, whichever is longer. Prior to resuming study treatment, surgically related AEs should resolve to  $\leq$  Grade 1 or baseline, and participants must meet relevant eligibility criteria as determined by the BMS Medical Monitor (or designee) in discussion with the investigator. The BMS Medical Monitor (or designee) must be consulted prior to re-initiating study treatment in a participant with a dosing delay lasting > 8 weeks from the previous dose.

# 7.7.5 Supportive Care Management

Supportive care management for each FRACTION-Gastric Cancer study treatment combination and, as necessary, is outlined in the FRACTION-Gastric Cancer Sub-Protocol describing that treatment combination.

# 7.8 Treatment After the End of the Study

At the end of the study, BMS will not continue to provide BMS-supplied study treatment to participants/investigators unless BMS chooses to extend the study. The investigator should ensure that the participant receives appropriate standard of care to treat the condition under study.

#### 8 DISCONTINUATION CRITERIA

# 8.1 Discontinuation from Study Treatment

Participants must discontinue IP (and non-IP at the discretion of the investigator) for any of the following reasons:

- Participant's request to stop study treatment. Participants who request to discontinue study treatment will remain in the study and must continue to be followed for protocol-specified follow-up procedures as outlined in Section 2. The only exception to this is when a participant specifically withdraws consent for any further contact with him/her or persons previously authorized by participant to provide this information
- Any clinical AE, laboratory abnormality, or intercurrent illness, that, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the participant
- Termination of the study by BMS
- Loss of ability to freely provide consent through imprisonment or involuntarily incarceration for the treatment of either a psychiatric or a physical (eg, infectious disease) illness. (Note: Under specific circumstances and only in countries where local regulations permit, a

participant who has been imprisoned may be permitted to continue as a participant. Strict conditions apply and BMS approval is required.)

- Inability to comply with the protocol
- Pregnancy
- Documented disease progression as defined by RECIST v1.1 (see Appendix 5), unless the participant meets criteria for treatment beyond progression (see Section 7.4.2) or the participant continues study treatment by entering another track or receiving retreatment (see Section 5.1.3.3)
- Clinical deterioration while receiving active study treatment that, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the participant
- Discretion of the investigator
- Protocol-defined reasons for discontinuation (Criteria for permanent discontinuation for each FRACTION-Gastric Cancer study treatment combination and/or nivolumab in combination with ipilimumab are provided in each FRACTION-Gastric Cancer Sub-Protocol.)
- End of study

Refer to Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol for data to be collected at the time of study treatment discontinuation and follow-up and for any further evaluations that can be completed.

In the case of pregnancy, the investigator must immediately notify the BMS Medical Monitor (or designee) of this event. In most cases, the study treatment will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for participant safety). Please notify the BMS Medical Monitor (or designee) within 24 hours of awareness of the pregnancy. If the investigator determines a possible favorable benefit/risk ratio that warrants continuation of study treatment, a discussion between the investigator and the BMS Medical Monitor (or designee) must occur.

All participants who discontinue study treatment should comply with protocol-specified follow-up procedures as outlined in Section 2. The only exception to this requirement is when a participant withdraws consent for all study procedures, including posttreatment study follow-up, or loses the ability to consent freely (ie, is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or a physical illness).

If study treatment is discontinued prior to the participant's completion of the study, the reason for the discontinuation must be documented in the participant's medical records and entered on the appropriate CRF page.

Additional study treatment-specific discontinuation criteria are provided in each FRACTION-Gastric Cancer Sub-Protocol.

#### 8.1.1 Permanent Discontinuation

Criteria for permanent discontinuation for each FRACTION-Gastric Cancer study treatment combination are provided in the FRACTION-Gastric Cancer Sub-Protocol describing that treatment combination.

# 8.1.2 Study Treatment Combination Arm Discontinuation Criteria

In the event that 20% or more of study participants in a novel FRACTION-Gastric Cancer study treatment combination arm of a given track, at any given time, meet any of the toxicity criteria for permanent discontinuation (as described in Section 8.1.1), then consideration will be given to discontinue that FRACTION-Gastric Cancer study treatment combination arm in that track. This will include early side effects seen with combination agents and longer-term effects such as endocrinopathies. This action will be taken in consultation with the SMB and will consider other pertinent facts in coming to a decision, including the toxicity profile of that combination seen outside FRACTION-Gastric Cancer, participant benefit as measured by anti-tumor response, and comparison to nivolumab in combination with ipilimumab.

Discontinuation of a study treatment combination arm in a given track for any reason will not lead to discontinuation for that combination in all tracks. Safety of all open-label study treatment combination arms in other tracks that contain the same agent (or agents) will be assessed by SMB and the Sponsor. In the event of serious, unexpected, or life-threatening emergent toxicities, relevant study treatment combination arms may then be modified to maintain the safety of participants. Decisions on such steps and the re-initiation of any study treatment combination arms that had been stopped would be made by SMB in consultation with the Sponsor and relevant authorities (eg, IRB/IEC).

# 8.1.3 Post Study Treatment Study Follow-up

In this study, PFSR is a key endpoint of the study. Post-study follow-up is of critical importance and is essential to preserving participant safety and the integrity of the study. Participants who discontinue study treatment must continue to be followed (in this study or a rollover study) for safety (Section 5).

# 8.2 Discontinuation from the Study

Participants who request to discontinue study treatment will remain in the study and must continue to be followed up for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him/her or persons previously authorized by participant to provide this information.

- Participants should notify the investigator of the decision to withdraw consent from future follow-up in writing, whenever possible.
- The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is from further treatment with study treatment only or also from study procedures and/or posttreatment study follow-up, and entered onto the appropriate CRF page.
- In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

# 8.3 Lost to Follow-up

- All reasonable efforts must be made to locate participants to determine and report their ongoing status. This includes follow-up with persons authorized by the participant.
- Lost to follow-up is defined by the inability to reach the participant after a minimum of 3 documented phone calls, faxes, or emails, as well as lack of response by participant to 1 registered mail letter. All attempts should be documented in the participant's medical records.
- If it is determined that the participant has died, the site will use permissible local methods to obtain date and cause of death.
- If investigator's use of third-party representative to assist in the follow-up portion of the study has been included in the participant's informed consent, then the investigator may use a Sponsor-retained third-party representative to assist site staff with obtaining participant's contact information or other public vital status data necessary to complete the follow-up portion of the study.
- The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information.
- If, after all attempts, the participant remains lost to follow-up, then the last known alive date as determined by the investigator should be reported and documented in the participant's medical records.

#### 9 STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and timing are summarized in the Schedule of Activities in Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol.
- Protocol waivers or exemptions are not allowed.
- All immediate safety concerns must be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study treatment.
- Adherence to the study design requirements, including those specified in the Schedule of Activities in Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria before randomization. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (eg, blood count) and obtained before signing of informed consent may be utilized for screening or baseline purposes provided that the procedure meets the protocol-defined criteria and has been performed within the timeframe defined in the Schedule of Activities in Section 2 and the Ontreatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol.

# 9.1 Efficacy Assessments

Disease assessment with contrast-enhanced computed tomography (CT)/MRI scans acquired on dedicated CT/MRI equipment is preferred for this study. CT or MRI of the abdomen, chest, pelvis, and all known sites of disease should be performed for tumor assessments.

CT scans should be acquired with 5-mm slices with no intervening gap (contiguous). Should a participant have a contraindication for CT intravenous contrast, a contrast-enhanced MRI of the chest, abdomen, pelvis, and other known sites of disease may be obtained. MRIs should be acquired with slice thickness of 5 mm with no gap (contiguous). Every attempt should be made to image each participant using an identical acquisition protocol on the same scanner for all imaging time points.

MRI or CT brain scans during on-study treatment and follow-up periods are required only if there is a history of brain metastasis or clinically indicated for symptoms that suggest CNS involvement. Surveillance MRI should be performed per standard of care (approximately every 12 weeks or sooner). Participants with a history of bone metastasis should have a bone scan, if clinically indicated.

Assessments will be performed at baseline and at the time points described in each FRACTION-Gastric Cancer Sub-Protocol, up to and including Week 24 during the Treatment Phase or until disease progression per RECIST v1.1 criteria (see Appendix 5) or confirmed disease progression for participants treated beyond progression (defined as an additional 10% increase in tumor burden volume with a minimum 5 mm absolute increase from time of initial PD assessment [an increase in the sum of diameters of all target lesions and/or the diameters of new measurable lesions compared to the time of initial PD]), discontinuation of study treatment, or withdrawal from the study. Please refer to Section 2 for timing of assessments. Tumor assessments at other time points may be performed if the investigator is concerned about tumor progression. Assessment of response will be outlined for each combination therapy in the specific FRACTION-Gastric Cancer Sub-Protocol. Assessments of PR and CR must be confirmed at least 4 weeks after initial response. Assessment of tumor response will be reported by the investigator for appropriate populations of participants, as defined by RECIST v1.1 criteria (see Appendix 5) for participants with solid tumors. Same modality/scanner should be used for all assessments.

Changes in tumor measurements and tumor responses will be assessed by the investigator using RECIST v1.1 criteria.<sup>54</sup> Investigators will also report the number and size of new lesions that appear while on study. The time point of tumor assessments will be reported on the CRF based on the investigator's assessment using RECIST v1.1 criteria. (See Appendix 5 and Section 7.4.2 for specifics of RECIST v1.1 criteria to be utilized in this study.)

Tumor assessments will be submitted to a third party radiology vendor on an ongoing basis; participant management is not dependent on third-party review of tumor assessments.

As a participant's response to prior therapy is an important part of medical history, additional details regarding the previous therapy, including but not limited to best response to therapy, timing of progression on prior therapy, method of how the progression was measured, existence of

confirmation scan to document progression and detailed information such as other clinical evidence (eg, increased pain requiring palliative radiotherapy) to support progression, response/progression dates, and reason for discontinuation will be collected in this trial.

# 9.1.1 Imaging Assessment for the Study

Central assessments are not planned for this study; however, copies of all scans will be stored for possible future central analysis, if determined to be necessary by BMS. At the Sponsor's discretion, scans may be collected centrally to be reviewed by independent radiologists.

#### 9.2 Adverse Events

The definitions of an AE or SAE can be found in Appendix 3.

AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, that are considered related to the study treatment or the study, or that caused the participant to discontinue before completing the study.

Contacts for SAE reporting are specified in Appendix 3.

## 9.2.1 Time Period and Frequency for Collecting AE and SAE Information

The collection of nonserious AE information should begin at initiation of study treatment and continue until 100 days following the last dose of study treatment and at the time points specified in the Schedule of Activities (see Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol). Nonserious AE information should also be collected from the start of a placebo lead-in period or other observational period intended to establish a baseline status for the participants.

Sections 5.6.1 and 5.6.2 in the IBs represent the Reference Safety Information to determine expectedness of SAEs for expedited reporting. Following the participant's written consent to participate in the study, all SAEs, whether related or not related to study treatment, must be collected, including those thought to be associated with protocol-specified procedures.

All SAEs must be collected that occur during the screening period and within 100 days of discontinuation of dosing. If applicable, SAEs must be collected that relate to any later protocol-specified procedure (eg, a follow-up skin biopsy). Participants who are randomized and never treated with study treatment must have SAEs collected for 30 days from the date of randomization.

The investigator must report any SAE that occurs after these time periods and that is believed to be related to study treatment or protocol-specified procedure.

- Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the appropriate section of the eCRF section.
- All SAEs will be recorded and reported to the Sponsor or designee within 24 hours, as indicated in Appendix 3.

• The investigator will submit any updated SAE data to the Sponsor within 24 hours of this being available.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the investigator must promptly notify the Sponsor.

The method of evaluating and assessing causality of AEs and SAEs and the procedures for completing and reporting/transmitting SAE reports are provided in Appendix 3.

Every AE must be assessed by the investigator with regard to whether it is considered immune mediated. For events which are potentially immune mediated, additional information will be collected on the participant's CRF.

Immune-mediated AEs are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. Immune-mediated AEs can include events with an alternate etiology that were exacerbated by the induction of autoimmunity. Information supporting the assessment will be collected on the participant's CRF.

# 9.2.2 Method of Detecting AEs and SAEs

AEs can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a participant. (In order to prevent reporting bias, participants should not be questioned regarding the specific occurrence of one or more AEs.)

# 9.2.3 Follow-up of AEs and SAEs

- Nonserious AEs should be followed to resolution or stabilization or reported as SAEs if they become serious (see Appendix 3).
- Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study treatment and for those present at the end of study treatment as appropriate.
- All identified nonserious AEs must be recorded and described on the nonserious AE page of the CRF (paper or electronic). Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs and nonserious AEs of special interest (as defined in each FRACTION-Gastric Cancer Sub-Protocol) will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the participant is lost to follow-up (as defined in Section 8.3).

Further information on follow-up procedures is given in Appendix 3.

Protocol Amendment No.: 06

# 9.2.4 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of SAEs is essential so that legal obligations and ethical responsibilities toward the safety of participants and the safety of a product under clinical investigation are met.
- An investigator who receives an investigator safety report describing SAEs or other specific safety information (eg, summary or listing of SAEs) from the Sponsor will file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

The Sponsor or designee will be reporting AEs to regulatory authorities and ethics committees according to local applicable laws including European Directive 2001/20/EC and Food and Drug Administration Code of Federal Regulations 21 CFR Parts 312 and 320. A Suspected, Unexpected Serious Adverse Reaction (SUSAR) is a subset of SAEs and will be reported to the appropriate regulatory authorities and investigators following local and global guidelines and requirements.

## 9.2.5 Pregnancy

If, following initiation of the study treatment, it is subsequently discovered that a participant is pregnant or may have been pregnant at the time of study exposure, including during at least 5 half-lives- after product administration, the investigator must immediately notify the BMS Medical Monitor (or designee) of this event and complete and forward a Pregnancy Surveillance Form to BMS Medical Monitor (or designee) within 24 hours of awareness of the event and in accordance with SAE reporting procedures described in Appendix 3.

In most cases, the study treatment will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for participant safety). Please call the BMS Medical Monitor (or designee) within 24 hours of awareness of the pregnancy.

Follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome and, where applicable, offspring information must be reported on the Pregnancy Surveillance Form.

Any pregnancy that occurs in a female partner of a male study participant should be reported to the BMS (or designee). In order for the BMS (or designee) to collect any pregnancy surveillance information from the female partner, the female partner must sign an informed consent form for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form.

In cases where a study drug can be present in seminal fluid, at exposures sufficient to potentially cause fetal toxicity, and if any sexual activity (eg, vaginal, anal, oral) has occurred between a male participant and a pregnant WOCBP partner(s), the information should be reported to the Sponsor or designee, even if the male participant has undergone a successful vasectomy. In order for Sponsor or designee to collect any pregnancy surveillance information from the female partner, the female partner(s) must sign an informed consent form for disclosure of this information. Information on the pregnancy will be collected on the Pregnancy Surveillance Form.

Protocol Amendment No.: 06

# 9.2.6 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the nonserious AE CRF page or SAE Report Form electronic, as appropriate. Paper forms are only intended as a back-up option when the electronic system is not functioning.

- Any laboratory test result that is clinically significant or meets the definition of an SAE
- Any laboratory test result abnormality that required the participant to have study treatment discontinued or interrupted
- Any laboratory test result abnormality that required the participant to receive specific corrective therapy

It is expected that wherever possible, the clinical rather than laboratory term would be used by the reporting investigator (eg, anemia versus low hemoglobin value).

# 9.2.7 Potential Drug Induced Liver Injury

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential drug-induced liver injury (p-DILI) event. All occurrences of p-DILIs, meeting the defined criteria, must be reported as SAEs (see Section 9.2 and Appendix 3 for reporting details).

p-DILI is defined as follows:

- Aminotransferase (AT) (ALT or AST) elevation  $> 3 \times ULN$  AND
- Total bilirubin  $> 2 \times ULN$ , without initial findings of cholestasis (elevated serum alkaline phosphatase)

**AND** 

• No other immediately apparent possible causes of AT elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, preexisting chronic or acute liver disease, or the administration of other treatment(s) known to be hepatotoxic or cancer metastases.

The key responsibilities for investigators during p-DILI assessment include the following: (i) early detection, medical evaluation (including the exclusion of other potential causes), and rapid laboratory confirmation of liver-related abnormalities and (ii) BMS notification of p-DILI cases via SAE forms. Following the gathering and assessment of relevant clinical information, BMS is responsible for the following: (iii) timely evaluation and triaging of p-DILI cases, (iv) expedited reporting of p-DILI cases, and (v) expanded review of p-DILI cases, including a detailed assessment of all available clinical information, investigations, and biochemical data.

Investigators are expected to monitor ongoing routine and ad hoc hepatic laboratory test results to rapidly determine whether a participant meets p-DILI criteria. They are expected to promptly notify BMS of all p-DILI cases. p-DILI cases may be identified by abnormal liver biochemistry values, whether or not they are accompanied by liver-related signs and/or symptoms. In both cases, expedited confirmation with repeat laboratory testing should occur within 3 business days using a

Hepatic Laboratory Panel (ALT, AST, total bilirubin, and alkaline phosphatase). Any participant with an abnormal Hepatic Laboratory Panel that meets p-DILI criteria is a candidate for study treatment discontinuation. Any confirmed p-DILI events must be reported (along with a description of the clinical findings) to BMS as an SAE within 24 hours of confirmation.

An extensive clinical history, examination, and appropriate investigations should be obtained to exclude cholestatic and other apparent causes that may explain the observed abnormalities in liver function and/or hepatic signs and symptoms. Other apparent causes include, nonexhaustively and by way of example only, infectious diseases (such as active hepatitis A, B, and C), congenital diseases (such as Gilbert's syndrome), neoplastic diseases (such as hepatocellular carcinoma), autoimmune diseases (such as primary biliary cirrhosis), and the use of concomitant hepatotoxic medications (such as antibiotics, oral contraceptive pill, and herbal medicines). All investigations to exclude potential causes of liver function abnormalities or hepatic signs and/or symptoms should be guided by relevant factors such as the participant's age, gender, clinical history, and signs and symptoms.

## 9.2.8 Other Safety Considerations

Any significant worsening noted during interim or final physical examinations, ECG, X-ray filming, and any other potential safety assessment required or not required by protocol should also be recorded as a nonserious or serious AE, as appropriate, and reported accordingly.

## 9.3 Overdose

An overdose is defined as the accidental or intentional administration of any dose of a product that is considered both excessive and medically important. See Appendix 3 for reporting overdose.

# 9.4 Safety

Planned time points for all safety assessments are listed in the Schedule of Activities in Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol.

## 9.4.1 Clinical Safety Laboratory Assessments

Investigators must document their review of each laboratory safety report.

A local laboratory will perform the analyses and will provide reference ranges for these tests. The clinical laboratory assessments are indicated in Table 9.4.1-1.

Results of clinical laboratory tests performed on Day -1 must be available prior to dosing.

Results of all laboratory tests required by this protocol must be provided to BMS, recorded either on the laboratory pages of the CRF or by another mechanism, as agreed upon between the investigator and BMS (eg, provided electronically). If the units of a test result differ from those printed on the CRF, the recorded laboratory values must specify the correct units. Any abnormal laboratory test result considered clinically significant by the investigator must be recorded on the appropriate AE page of the CRF (see Section 9.2.6).

Protocol Amendment No.: 06 Date: 13-Aug-2021

## Table 9.4.1-1: Clinical Laboratory Assessments

#### Hematology

CBC with differential including platelets

#### **Serum Chemistry**

AST Total protein
ALT Albumin

Total bilirubin Sodium

Direct bilirubin Potassium

Alkaline phosphatase Chloride

LDH Carbon dioxide or bicarbonate

Creatinine Calcium

BUN or urea Phosphorus

Uric acid (screening only) Magnesium

Glucose Creatine kinase

Amylase CrCl (screening only)

Lipase C-reactive protein

Gamma-glutamyl transferase

#### Urinalysis

Protein Leukocyte esterase
Glucose Specific gravity

Blood pH

Microscopic examination of the sediment if blood, protein, or leukocyte esterase are positive on the dipstick

#### Serology

Serum for hepatitis A (IgG and IgM) antibody, serum for hepatitis C antibody or hepatitis C RNA (if hepatitis C antibody is positive, reflex to hepatitis C RNA), HBsAg, and HIV-1 and HIV-2 antibodies (testing for HIV-1 and HIV-2 antibodies must be performed at the sites mandated by local requirements.)

#### Other Analyses

Pregnancy test (WOCBP only)

TSH with reflex to free T3 and free T4, as applicable

FSH, if needed to document postmenopausal status, as defined in Appendix 4

Abbreviations: BUN = blood urea nitrogen; CBC = complete blood count; FSH = follicle stimulating hormone; HBsAg = hepatitis B surface antigen; IgG = immunoglobin G; IgM = immunoglobin M; LDH = lactate dehydrogenase; T3 = triiodothyronine; T4 = thyroxine; TSH = thyroid-stimulating hormone.

Protocol Amendment No.: 06

# 9.4.2 Imaging Safety Assessment

Any incidental findings of potential clinical relevance that are not directly associated with the objectives of the protocol should be evaluated and handled by the study investigator as per standard medical/clinical judgment.

### 9.5 Pharmacokinetic

Separate detailed instructions for the collection, processing, handling, labeling, storage, and shipment of PK samples will be provided in the Laboratory Procedures Manual.

The details pertaining to the timing of PK sample collection for Tracks 1 and 2, on treatment and follow-up, are provided in each FRACTION-Gastric Cancer Sub-Protocol.

The serum samples will be analyzed for study treatments. In addition, selected serum samples may be analyzed by an exploratory method that measures study treatment for technology exploration purposes; exploratory results will not be reported.

Upon implementation of Protocol Amendment 06, PK sample collection is no longer necessary for any participant who is on study treatment.

Please refer to Table 2-3.

# 9.6 Pharmacodynamics

Pharmacodynamic measures (in the form of biomarker assessments) may be assessed for associations with clinical outcomes.

The sample subtypes and testing plans associated with each are described in Section 9.8. Complete instructions on the collection, processing, handling, and shipment of all samples described herein will be provided in a separate Laboratory Procedures Manual.

Upon implementation of Protocol Amendment 06, samples for pharmacodynamic assessments are no longer necessary for any participant who is on study treatment.

Please refer to Table 2-3.

# 9.7 Pharmacogenomics

Not applicable.

#### 9.8 Biomarkers

Planned time points for all biomarker assessments are listed in the Schedule of Activities in Section 2 and the On-treatment Procedural Outline(s) specific to each FRACTION-Gastric Cancer Sub-Protocol.

Upon implementation of Protocol Amendment 06, samples for biomarker assessments are no longer necessary for any participant who is on study treatment.

Please refer to Table 2-3.

Protocol Amendment No.: 06











Approved v 8.0 930104678 8.0



# 9.8.5 Immunogenicity Assessments

Separate detailed instructions for the collection, processing, handling, labeling, storage, and shipment of immunogenicity samples will be provided in the Laboratory Procedures Manual.

The details pertaining to the timing of immunogenicity sample collection for the On-treatment Phase and Follow-up are provided in each FRACTION-Gastric Cancer Sub-Protocol.

The serum samples will be banked for analyses of ADAs by validated immunoassays. In addition, selected serum samples may be analyzed by an exploratory method that detects ADAs for technology exploration purposes; exploratory results will not be reported. Serum samples designated for PK may also be used for immunogenicity analysis, if required (eg, insufficient volume for complete immunogenicity assessment or to follow up on suspected immunogenicity-related AE).



Protocol Amendment No.: 06

#### 9.8.10 Other Assessments

Not applicable.

## 9.9 Medical Resource Utilization and Health Economics

# 9.9.1 Patient-reported Outcomes

The effects of GC and its treatment on health status and quality of life will be assessed using the 3-level version of EQ-5D self-report questionnaire (EQ-5D-3L) and Functional Assessment of Cancer Therapy-Gastric (FACT-Ga) Gastric Cancer Subscale (GaCS), and/or Esophagus Cancer Subscale (ECS) from the Functional Assessment of Cancer Therapy-Esophageal (FACT-E). 58,59,60 Participants will be asked to complete the assessments during on-study clinic visits and/or at designated visits during the Safety and Survival Follow-up Phases. The questionnaires will be provided in the participant's preferred language (if available) or in English and may be administered by telephone during the Survival Follow-up Phase. A standardized script in the participant's preferred language (if available) will be used to facilitate telephone administration of the EQ-5D-3L. Section 2 and the On-treatment Procedural Outline(s) in each FRACTION-Gastric Cancer Sub-Protocol provide information regarding the timing of patient-reported outcomes assessments.

Participants' reports of general health, functional status, and utility for health will be measured using the EQ-5D-3L. The EQ-5D-3L is a standardized instrument used to measure self-reports of health status and functioning. The instrument's descriptive system consists of 5 dimensions, which are mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels, reflecting "no health problems," "moderate health problems," and "extreme health problems." A dimension for which there are no problems is said to be at Level 1, while a dimension for which there are extreme problems is said to be at Level 3. Thus, the vectors 11111 and 33333 represent the best health state and the worst health state, respectively, described by the EQ-5D-3L. Altogether, the instrument describes 3<sup>5</sup> or 243 health states. Empirically derived weights can be applied to an individual's responses to the EQ-5D-3L descriptive system to generate an index measuring the value to society of his or her current health. Such preference-weighting systems have been developed for Japan, United Kingdom, US, Spain, Germany, and numerous other populations. In addition, the EQ-5D-3L includes a visual analog scale that allows respondents to rate their own current health on a 101-point scale ranging from "best imaginable" to "worst imaginable" health.

In addition to the EQ-5D (which all participants will complete), participants will also complete one or more disease-specific symptom subscales based on their cancer type:

- Participants with GC cancer will complete the Functional Assessment of Cancer Therapy-Gastric (FACT-Ga) Gastric Cancer Subscale (GaCS)
- Participants with EC will complete the Esophagus Cancer Subscale (ECS) from the Functional Assessment of Cancer Therapy-Esophageal (FACT-E).
- Participants with GEJ will complete items from both the GaCS and ECS subscales.
The FACT-Ga is a validated, cancer-targeted measure of disease-related symptoms, functioning, and well-being. Nineteen of the FACT-Ga questionnaire's items comprise the disease-specific GaCS, which assesses GC symptoms and impacts relating to pain, reflux, dysphagia, eating difficulties, tiredness, weakness, interference, and difficulty planning. Each GaCS item is rated on a 5-point scale ranging from 0 (not at all) to 4 (very much). A summary score is derived by aggregating responses for the 19 items, with higher scores indicating less symptom burden.

The FACT-E is a validated, cancer-targeted measure of disease-related symptoms, functioning, and well-being. Seventeen of the FACT-E questionnaire's items comprise the disease-specific ECS, which assesses esophageal cancer symptoms and impacts relating to swallowing, eating, dry mouth, trouble breathing, communicating with others, appetite, coughing, pain and weight loss. Each ECS item is rated on a 5-point scale ranging from 0 (not at all) to 4 (very much). A summary score is derived by aggregating responses for the 17 items, with higher scores indicating less symptom burden.

#### 10 STATISTICAL CONSIDERATIONS

## 10.1 Sample Size Determination

Sample sizes are guided by Simon 2-stage (optimal) designs. Because of the different participant populations (anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment-naïve versus anti-PD-1, anti-PD-L1, or anti-CTLA-4 treatment experienced) and existing options under each track, different criteria are applied to determine the number of participants for each stage and the strength of the efficacy signal that would recommend proceeding to the next stage. Details are described in subsequent sections and in Table 10.1-1. Any additional statistical considerations unique to the new treatment combinations will be described in the new sub-protocols.

For sample size calculation and for simplicity of description, recommendations for stopping or progressing to the next stage are based on the number of objective responses observed. However, since best overall response (BOR) does not necessarily capture the full extent of clinical benefit and since response can be delayed or of short duration, BMS will also review other aspects of clinical benefit that may better predict OS benefit, such as DOR and PFSR, as well as the relative performance of different study treatment combination arms, before making a final determination.

Enrollment will be continued after reaching the indicated number of participants at Stage 1 while the initial efficacy evaluation is ongoing. This will allow additional participants to enroll to account for unexpected trial impact, such as response nonevaluable participants due to early dropout, design parameter change (eg., historical rate update), etc.

Although the sample size calculations are based on efficacy considerations, safety will also be continuously assessed and will be taken into account in the decision to continue or terminate a study treatment arm. In Track 2, 41 participants per study treatment arm in Stages 1 and 2 combined will result in 88% probability of detecting an AE that has a true rate of 5%. More participants per study treatment arm in Stages 1 and 2 combined will result in a higher probability of detecting an AE that has a true rate of 5%.

| <b>Table 10.1-1:</b> | Simon 2-stage (Optimal) Design Considerations |
|----------------------|-----------------------------------------------|
|----------------------|-----------------------------------------------|

| | Historical | | Stage 1 Responders/Stage 1 n Stage | | onders/Total n | Error a séa d'un roviélle | E-mandad maridh |
|---|---|---|---|---|---|---|---|
| Track | ORR/<br>Target ORR | Consider<br>Futility | Go to Stage 2 | Consider<br>Futility | Consider<br>Efficacy | Expected n with<br>Historical ORR | Expected n with<br>Target ORR |
| 1 | 20%/40% | ≤ 4/19 | ≥ 5/19 | ≤ 15/54 | ≥ 16/54 | 30.4 | 51.6 |
| 2 | 5%/20% | ≤ 1/21 | ≥ 2/21 | ≤ 4/41 | ≥ 5/41 | 26.6 | 39.8 |

Note: Numbers of responses serve as a guideline; however, the totality of efficacy data will be considered when making decisions to terminate or continue an arm.

The Track 1 Simon 2-stage (optimal) design assumes a historical response rate of 20% and a target response rate of 40%, based on the observed response rate of approximately 24% for the nivolumab in combination with ipilimumab and approximately 12% for nivolumab monotherapy participants in Study CA209032. A false positive rate of 5% and power of 90% are used.

Because there is very little data available on participants with prior anti-PD-1, anti-PD-L1, or anti CTLA-4 treatment, the Track 2 design is not based on an observed historical response rate. Rather, the assumption is made that a response rate below 5% would not be worth further study and that a target response rate of 20% would be worth pursuing in this population. A false positive rate of 5% and power of 90% are used.

With regard to sample size, participants who are re-randomized to a different study treatment in Track 2 will be counted once for each randomization; participants who are retreated within the same study treatment arm will only be counted once.

Protocol Amendment No.: 06

Date: 13-Aug-2021

Approved v8.0 930104678 8.0

## 10.1.1 Track 1 - Anti-PD-1, Anti-PD-L1, and Anti-CTLA-4 Treatment-naïve Participants

As shown in Table 10.1-1, a minimum of 19 participants in each study treatment combination arm will be treated in Stage 1 for an initial evaluation of efficacy. If the total number of responses observed in Stage 1 is  $\leq 4/19$ , the study treatment combination arm would likely not be considered efficacious; otherwise, enrollment to Stage 2 will continue, and an additional 35 participants will be treated. If the total number of responses at the end of Stage 2 is  $\leq 15/54$ , the study treatment combination arm will be terminated for futility; if there are more than 15 responses observed at the end of Stage 2, the study treatment combination arm may be carried on for further treatment development. The totality of efficacy data and response profile for each combination arm will be considered when making decisions to terminate or continue an arm.

The operating characteristics of this Simon 2-stage (optimal) design are provided in Figure 10.1.1-1. With the stopping boundaries as shown in Table 10.1-1, if the study treatment combination arm has an ORR no better than the historical control at 20%, then there is a 95% overall chance of stopping for futility, with a 67% chance of stopping at Stage 1; there is a 5% false positive rate. If the study treatment combination arm has an ORR equal to the target of 40%, then there is a 90% chance of declaring efficacy after Stage 2, whereas if the true ORR is 25%, 30%, or 35%, the power would be 21%, 49%, or 75%, respectively.

Figure 10.1.1-1: Operating Characteristics of Track 1 Simon 2-stage (Optimal) Design (Power = 90%, Alpha = 5%)



Abbreviation: prob = probability.

If 16 responses are observed at the end of Stage 2 (Declare Efficacy), then the 90% confidence interval (CI) for ORR will be (19%, 42%). The CI is calculated using the Clopper-Pearson method.

As stated in Section 10.1, the number of responses given here is used for sample size calculation and for simplicity of description. Before making a decision to terminate or continue an arm, BMS will also review the totality of all available data, which includes other aspects of efficacy that may help predict OS benefit, such as DOR and PFSR; clinical safety information; and biomarker data, as well as the relative performance of other treatment arms.

## 10.1.2 Track 2 - Anti-PD-1, Anti-PD-L1, or Anti-CTLA-4 Treatment-experienced Participants

For each study treatment combination arm under Track 2, the Simon 2-stage (optimal) design will be used. Initially, 21 participants per study treatment combination arm will be treated in Stage 1 and preliminary efficacy will be assessed when those participants are evaluable. If 1 or fewer responses are observed in Stage 1, the study treatment combination arm would likely not be considered efficacious; otherwise, Stage 2 will be initiated and enroll an additional 20 participants, for a total of 41 participants per study treatment combination arm. The totality of efficacy data and response profile for each combination will be considered when making decisions to terminate or continue an arm.

The operating characteristics of this Simon 2-stage (optimal) design are provided in Figure 10.1.2-1. With the stopping boundaries as shown in Table 10.1-1, if the study treatment combination arm has an ORR no better than 5%, then there is a 95% overall chance of stopping for futility, with a 72% chance of stopping at Stage 1; there is a 5% false positive rate. If the study treatment combination arm has an ORR equal to the target of 20%, then it has a 90% chance of declaring efficacy after Stage 2.

Stage 1 Stage 2 **Efficacy Stop ORR = 20%** (Prob. 90%) ≥ 5 Responses ≥ 2 Responses 20 Additional 21 Participants **Participants** ≤1 Responses ≤ 4 Responses Futility **Futility** Stop Stop **ORR = 5%** (Prob. (Prob. 72%)

Figure 10.1.2-1: Operating Characteristics of Track 2 Simon 2-stage (Optimal) Design (Power =90%, Alpha = 5%)

Abbreviation: prob = probability.

If 5 responses are observed at the end of Stage 2 (Declare Efficacy), then the 90% CI for ORR will be (5%, 24%). The CI is calculated using the Clopper-Pearson method.

As stated in Section 10.1, the number of responses given here is used for sample size calculation and for simplicity of description. Before making a decision to terminate or continue an arm, BMS will also review the totality of all available data, which includes other aspects of efficacy that may help predict OS benefit, such as DOR and PFSR; clinical safety information; and biomarker data, as well as the relative performance of other treatment arms.

Both participants previously treated in any track (re-randomized participants) and new participants who meet eligibility criteria are permitted to enter Track 2. Some slots in Track 2 will be reserved for re-randomized participants to ensure that both types of participants are enrolled in Track 2. At the initiation of the study, recruitment of re-randomized participants will be limited to 11 participants per Track 2 study treatment combination arm in Stage 1. In Stage 2, recruitment of additional re-randomized participants will be limited to 12 participants out of the 27 additional participants. The limited number of re-randomized participants may be re-adjusted depending on the enrollment rates, the rate of progression in Tracks 1 and 2, and the number of currently open study treatment arms in Track 2.



## 10.2 Populations for Analyses

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Enrolled | All participants who sign informed consent |
| Randomized | All participants who are randomized to any study treatment arm of any track in this study |
| Treated | All participants who are randomized and take at least 1 dose of study treatment |
| PK | All treated participants who have evaluable concentration time data |
| Immunogenicity | All treated participants who have available immunogenicity assessment data |
| Biomarker | All treated participants who have available biomarker data |

Protocol Amendment No.: 06

| Population | Description |
|---|---|
| Response-evaluable | All treated participants with measurable disease and 1 of the following: 1) at least 1 postbaseline tumor measurement, 2) clinical progression, or 3) death |

## 10.3 Statistical Analyses

The statistical analysis plan will be developed and finalized before database lock. Below is a summary of planned statistical analyses of the primary and secondary endpoints.

## 10.3.1 Efficacy Analyses

The primary efficacy analyses will be performed on treated population for the final analysis. Efficacy analyses based on the response-evaluable population may be performed for interim analyses, when the minimum follow-up period is less than sufficient to warrant adequate interpretation of the result. Details on censoring scheme on time-to-event endpoints such as DOR, PFS, and OS will be described in the SAP.

| Endpoint | Statistical Analysis Methods |
|---|---|
| ORR BOR for a participant will be assessed per RECIST v1.1 by investigator. | Estimate of ORR and corresponding 2-sided exact 95% CI will be derived using the Clopper-Pearson method by study treatment under each track. |
| Median DOR DOR for a participant with a BOR of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression per RECIST v1.1 or death, whichever occurs first. | Median DOR using the Kaplan-Meier method and corresponding 2-sided 95% CI will be derived using Brookmeyer and Crowley methodology (using log-log transformation) by study treatment under each track. |
| PFSR at 24 weeks PFS for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first. | Estimate by the Kaplan-Meier method and corresponding 95% CI will be derived based on Greenwood formula by study treatment under each track. |
| OS rate at certain time points OS for a participant is defined as the time from the first dosing date to the date of death due to any cause. | Estimate by the Kaplan-Meier method and corresponding 95% CI will be derived based on Greenwood formula by study treatment under each track. |

Treatments under each track for different populations will be analyzed independently. There is no intention to combine the same study treatment across tracks for efficacy analyses.

Efficacy from retreatment will be assessed and analyzed separately from the initial treatment.

Participants re-randomized into Track 2 will be combined with participants originally randomized into Track 2 for efficacy analysis.

Specific analyses to be performed for each track are shown in Table 10.3.1-1.

Protocol Amendment No.: 06

Date: 13-Aug-2021 78

| <b>Table 10.3.1-1:</b> | <b>Analyses Planned for Each Track</b> |
|------------------------|----------------------------------------|
|------------------------|----------------------------------------|

| Track | | ORR | DOR | PFSR | os |
|---------|------------------------------------|-----|-----|------|----|
| Track 1 | End of Simon Stages 1 and 2 | X | X | X | X |
| Track 2 | End of Simon Stages 1 and 2 | X | X | X | X |
| | Early Termination at Simon Stage 1 | | | X | X |

#### Track 1 - Anti-PD-1, Anti-PD-L1, and Anti-CTLA-4 Treatment-naïve Participants

The following additional analyses will be performed for Track 1 anti-PD-1, anti-PD-L1, and anti-CTLA-4 treatment-naïve participants combined at end of Stage 2. These efficacy analyses will be performed when the study treatment arms have been fully enrolled and followed up for at least 6 months. A descriptive odds ratio and estimate of the difference in ORRs, along with corresponding 2-sided 95% CIs, will be provided to evaluate differences between the 2 randomized study treatment arms (FRACTION-Gastric Cancer study treatment combination arm and nivolumab in combination with ipilimumab control arm). Additionally, for each study treatment arm, the ORR and corresponding 95% CIs will be calculated using Clopper-Pearson method. A descriptive hazard ratio and corresponding 2-sided 95% CI of PFS and OS will be estimated in a Cox proportional hazards model using study treatment as a single covariate to evaluate difference between the 2 study treatment arms (experimental and control arms). The PFS and OS curves for each study treatment arm will be estimated. Two-sided 95% CIs for median PFS and OS will be computed. PFSR at 24 weeks and survival rates at certain time points (eg, 2 years) will be estimated. Associated 2-sided 95% CIs will be calculated.

## 10.3.2 Safety Analyses

All safety analyses will be performed on the treated population.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Incidence of AEs, SAEs, and AEs leading to discontinuation and deaths AEs will be graded according to CTCAE Version 4.03. | Frequency distribution of treated participants with AE using the worst CTC grade on treatment. Participants will be counted once at the PT level, once at the SOC level, and once in the "Total subject" row at their worst CTC grade, regardless of SOC or PT. |
| Laboratory abnormalities Laboratory values will be graded according to CTCAE Version 4.03. | Laboratory shift table using worst CTC grade on treatment per participant. |

Abbreviations: CTC = Common Terminology Criteria; PT = preferred term; SOC = system organ class.

Same treatments under different tracks with different populations may be combined for safety analyses.

### 10.3.3 Other Analyses

Not applicable.

Protocol Amendment No.: 06

Date: 13-Aug-2021 79

## 10.3.3.1 Pharmacokinetic Analyses

The concentration-time data obtained in this study may be combined with data from other studies in the clinical development program to develop a population PK model. This model may be used to evaluate the effects of intrinsic and extrinsic covariates on the PK of each component of each FRACTION-Gastric Cancer study treatment combination and/or nivolumab in combination with ipilimumab and to determine measures of individual exposure (such as steady-state peak, trough, and time-averaged concentration). Model-determined exposures may be used for exposure-response-analyses of selected efficacy and safety endpoints. Results of population PK and exposure-response analyses will be reported separately.

## 10.3.3.2 Immunogenicity Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Incidence of ADA to individual component of study treatment combination arm | Frequency distribution of baseline ADA-positive participants and ADA-positive |
| Baseline ADA-positive participant is defined as a participant | participants after initiation of the study |
| who has an ADA-detected sample at baseline. <sup>a</sup> An | treatment |
| ADA-positive participant is a participant with at least | |
| 1 ADA-positive sample relative to baseline after initiation of | |
| the study treatment. | |

<sup>&</sup>lt;sup>a</sup> Baseline sample is the last sample before initiation of the study treatment.

## 10.3.3.3 Exploratory Biomarker Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Summary measures of change (or % change) from baseline in various biomarkers | Summary statistics by planned study day and treatment under each track; plots of the time course of biomarkers |

If there is indication of meaningful pattern over time, further analysis (eg, by linear mixed model) may be performed to characterize the relationship. Methods such as, but not limited to, logistic regression will be used to explore possible associations between biomarker measures and clinical outcomes. Additional details will be provided in the statistical analysis plan. Exploratory biomarker/pharmacodynamic analysis may be presented separately from the main clinical study report.

### 10.3.3.4 Outcomes Research Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Summary measures of EQ-5D-3L index and VAS scores and GaCS and/or ECS scores with corresponding change from baseline for each score | Summary statistics by planned study day and treatment under each track |
| EQ-5D-3L index scores will be derived using the United Kingdom weighting algorithm. | |
| Questionnaire completion rate | Summary statistics by planned study day and |
| Defined as the proportion of questionnaires actually received out of the expected number | treatment under each track |
| Proportion of participants reporting no, moderate, or severe problems in each of the 5 EQ-5D-3L dimensions | Summary statistics by planned study day and treatment under each track |
| Proportion will be based on the number of participants assessed at each assessment time point. | |

VAS = visual analog scale.

## 10.3.4 Interim Analyses

Data from individual study treatment arms under each track of this study may emerge at different times; timely decisions (including early termination) for each individual study treatment under different tracks are needed. Database lock and analysis for certain FRACTION-Gastric Cancer study treatment combination arms will be performed when all participants in these study treatment combination arms (under each track) have completed treatment and with sufficient follow-up. Potential interim analyses for each study treatment combination arm under each track at the end of Stage 1 (6 months after the first treatment date of the last participant within that arm) will be performed. These interim analyses will be performed independent of each other.

The SMB will have access to interim reports of safety and will provide advice to the Sponsor regarding study treatment arm termination due to safety concerns.

The statistical analysis plan will further describe the planned interim analyses.

Additional interim analyses may also be performed for administrative purposes or publications. No formal inferences requiring any adjustment to statistical significance level will be performed.

#### 11 REFERENCES

- Mellman I, Coukos G, Dranoff G. Cancer immunotherapy comes of age. Nature 2011;29:480-9.
- Pennock GK, Chow LQM. The evolving role of immune checkpoint inhibitors in cancer treatment. The Oncologist 2015;20:812-22.
- Schaer DA, Hirschhorn-Cymerman D, Wolchok JD. Targeting tumor-necrosis factor receptor pathways for tumor immunotherapy. J Immunother Cancer 2014;2:7.
- Watts TH. TNF/TNFR family members in costimulation of T cell responses. Annu Rev Immunol 2005;23:23-68.
- Vinay DS, Kwon BS. Immunotherapy of cancer with 4-1BB. Mol Cancer Ther 2012;11:1062-70.
- Ascierto PA, Simeone E, Sznol M, et al. Clinical experiences with anti-CD137 and anti-PD-1 therapeutic antibodies. Semin Oncol 2010;37(5):508-16.
- Gough MJ, Crittenden MR, Sarff MC, et al. Adjuvant therapy with agonistic antibodies to CD134 (OX40) increases local control after surgical or radiation therapy of cancer in mice. J Immunother 2010;33:798-809.
- <sup>8</sup> Curti BD, Kovacsovics-Bankowski M, Morris N, et al. OX40 is a potent immune-stimulating target in late-stage cancer patients. Cancer Res 2013;73:7189-98.
- Ohen AD, Schaer DA, Liu C, et al. Agonist anti-GITR monoclonal antibody induces melanoma tumor immunity in mice by altering regulatory T cell stability and intra-tumor accumulation. PLoS One 2010;5:e10436.
- Rosenzweig M, Ponte J, Apostolou I, et al. Development of TRX518, an aglycosyl humanized monoclonal antibody (Mab) agonist of huGITR [abstract]. J Clin Oncol 2010;28:e13028.
- He L-Z, Thomas L, Weidlick J, et al. Development of a human anti-CD27 antibody with efficacy in lymphoma and leukemia models by two distinct mechanisms [abstract]. Blood 2011;118:2861.
- Ansell SM, Northfelt DW, Flinn I, et al. Phase I evaluation of an agonist anti-CD27 human antibody (CDX-1127) in patients with advanced hematologic malignancies. J Clin Oncol 2014;32(5s):( abstr 3024).
- Wolchok JD, Kluger HM, Callahan MK, et al. Safety and clinical activity of nivolumab (anti-PD-1, BMS-936558, ONO-4538) in combination with ipilimumab in patients (pts) with advanced melanoma (MEL). J Clin Oncol 2013:31(suppl, abstr 9012).

- Sznol M, Kluger HM, Callahan MK, et al. Survival, response duration, and activity by BRAF mutation (MT) status of nivolumab (NIVO, anti-PD-1, BMS-936558, ONO-4538) and ipilimumab (IPI) concurrent therapy in advanced melanoma (MEL). J Clin Oncol 2014;32(suppl, abstr LBA9003).
- Hellmann MD, Gettinger SN, Goldman JW, et al. CheckMate 012: Safety and efficacy of first-line (1L) nivolumab (nivo; N) and ipilimumab (ipi; I) in advanced (adv) NSCLC. J Clin Oncol 2016;34(suppl,; abstr 3001).
- Escudier B, et al. CheckMate 214: Efficacy and safety of nivolumab + ipilimumab (N+I) v sunitinib (S) for treatment-naive advanced or metastatic renal cell carcinoma (mRCC), including IMDC risk and PD-L1 expression subgroups. ESMO 2017; abstract LBA5.
- Chen S, Lee LF, Fisher TS, et al. Combination of 4-1BB agonist and PD-1 antagonist promotes antitumor effector/memory CD8 T cells in a poorly immunogenic tumor model. Cancer Immunol Res 2015;3(2):149-60.
- Kim ES, Herbst RS, Wistuba II, et al. The BATTLE Trial: personalizing therapy for lung cancer. Cancer Discov 2011;1(1):44-53.
- Esserman LJ, Berry DA, Cheang MCU, et al. Chemotherapy response and recurrence-free survival in neoadjuvant breast cancer depends on biomarker profiles: results from the I-SPY 1 TRIAL (CALGB 150007/150012; ACRIN 6657). Breast Cancer Res Treat 2012;132:1049-62.
- Herbst RS, Gandara DR, Hirsch FR, et al. Lung Master Protocol (Lung-MAP)-A biomarker-driven protocol for accelerating development of therapies for squamous cell lung cancer: SWOG S1400. Clin Cancer Res 2015;21(7):1514-24.
- American Society of Clinical Oncology (ASCO). Targeted Agent and Profiling Utilization Registry Study (TAPUR). [cited 2015 Sep 11.] Available from URL: http://www.asco.org/practice-research/targeted-agent-and-profiling-utilization-registry-study.
- Ferlay J, Soerjomataram I, Dikshit R, et al. Cancer incidence and mortality worldwide: Sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer 2015;136:E359-E86.
- Edgren G, Adami HO, Weiderpass E, Nyren O: A global assessment of the oesophageal adenocarcinoma epidemic. Gut 2013; 62: 1406–1414
- <sup>24</sup> GLOBOCAN 2012: Estimated Cancer Incidence, Mortality and prevalence Worldwide in 2012 http://globocan.iarc.fr.
- NCCN guideline Gastric cancer (Ver 3.0, 2015). http://www.nccn.org/professionals/physician\_gls/f\_guidelines\_nojava.asp. Accessed: 18-Mar-2016.
- Waddell T, Verheij M, Allum W, et al. Gastric cancer†: ESMO-ESSO-ESTRO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol (2013) 24 (suppl 6):vi57-vi63.
- Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2010 (ver. 3).Gastric Cancer 2011;14:113-23.

- Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, et al. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet (London, England). 2010;376(9742):687–97
- Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, et al. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014;15(11):1224–35
- Fuchs CS, Tabernero J, Tomášek J, Chau I, Melichar B, Safran H, Tehfe MA, Filip D, Topuzov E, Schlittler L, et al. Biomarker analyses in REGARD gastric/GEJ carcinoma patients treated with VEGFR2-targeted antibody ramucirumab. Br J Cancer. 2016;115(8):974–82
- Ohtsu A, Shah MA, Cutsem EV, et al. Bevacizumab in Combination With Chemotherapy As First-Line Therapy in Advanced Gastric Cancer: A Randomized, Double-Blind, Placebo-Controlled Phase III Study. J Clin Oncol 2011;29:3968-76.
- <sup>32</sup> Cunningham D, Starling N, Rao S, et al. Capecitabine and Oxaliplatin for Advanced Esophagogastric Cancer. N Engl J Med 2008;358:36-46.
- Yamada Y, Higuchi K, Nishikawa K, et al. Phase III study comparing oxaliplatin plus S-1 with cisplatin plus S-1 in chemotherapy-naïve patients with advanced gastric cancer. Annals of Oncology 2015;26:141-48.
- Janjigian YY, et al CheckMate-032 Study: Efficacy and Safety of Nivolumab and Nivolumab Plus Ipilimumab in Patients With Metastatic Esophagogastric Cancer. J Clin Oncol. 2018 Aug 15:JCO2017766212. doi: 10.1200/JCO.2017.76.6212. [Epub ahead of print]
- Brahmer J, Reckamp KL, Baas P, et al. Nivolumab versus Docetaxel in Advanced Squamous Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35.
- Larkin J, Chiarion-Sileni V, Gonzalez R, et al. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med 2015;373:23-34.
- Motzer RJ, Escudier B, McDermott DF, et al. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13.
- Opdivo (nivolumab) US Prescribing Information. [cited 2016 Mar 18]. Accessed from URL http://packageinserts.bms.com/pi/pi opdivo.pdf.Bristol-Myers Squibb, 2016.
- Summary of Product Characteristics (SmPC), Nivolumab. http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_-Product Information/human/003985/WC500189765.pdf. Accessed: 18-Mar-2016.
- Yervoy (Ipilimumab) US Prescribing Information. [cited 2016 Mar 18]. Accessed from URL: http://packageinserts.bms.com/pi/pi yervoy.pdf. Bristol-Myers Squibb 2016.

- Ipilimumab Summary of Product Characteristics [cited 2016 Mar 18]. Available from URL: http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_\_Product\_Information/human/002213/WC500109299.pdf.
- <sup>42</sup> Curran MA, Montalvo W, Yagita H, et al. PD-1 and CTLA-4 combination blockade expands infiltrating T cells and reduces regulatory T and myeloid cells within B16 melanoma tumors. Proc Natl Acad Sci U S A 2010;107: 4275-80.
- Wu C, Zhu Y, Jiang J et al. Immunohistochemical localization of programmed death-1 ligand-1 (PD-L1) in gastric carcinoma and its clinical significance. Acta Histochem.2006;108(1):19-24.
- Ohigashi Y, Sho M, Yamada Y et al. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005;11(8):2947-53.
- Janjigian YY, Ott PA, Calvo E, et al. Nivolumab ± ipilimumab in pts with advanced (adv)/metastatic chemotherapy-refractory (CTx-R) gastric (G), esophageal (E), or gastroesophageal junction (GEJ) cancer: CheckMate 032 study. J Clin Oncol. 2017;35(suppl 15):4014-4.
- Bang YJ, et al. Relationship between PD-L1 expression and clinical outcomes in patients with advanced gastric cancer treated with the anti-PD-1 monoclonal antibody pembrolizumab (MK 3475) in KEYNOTE-012.ASCO 2015, abstract 4001.
- <sup>47</sup> Chung HC, Arkenau HT, Wyrwicz L, et al. Avelumab (MSB0010718C), an anti-PD-L1 antibody, in patients with advanced gastric or gastroesophageal junction cancer: a Phase Ib trial. ESMO 2015, abstract. 2364.
- Kang YK, Boku N, Satoh T, et al. Nivolumab in patients with advanced gastric or gastrooesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebocontrolled, phase 3 trial. Lancet 2017;S0140-6736(17)31827-5.
- Keytruda (pembrolizumab) US prescribing information. [cited 2016 Nov 9]. Accessed from URL http://www.merck.com/product/usa/pi circulars/k/keytruda/keytruda pi.pdf, 2017.
- Fuchs CS, Doi T, Jang RW-J, et al. KEYNOTE-059 cohort 1: Efficacy and safety of pembrolizumab (pembro) monotherapy in patients with previously treated advanced gastric cancer. J Clin Oncol 2017:35(suppl, abstr 4003).
- Spigel DR, et al. Randomized results of continuous vs 1-year fixed-duration in patients with advanced non-small cell lung cancer. Oral presentation at the European Society of Medical Oncology Annual Meeting. 2017 Sep 8-12; Madrid, Spain. Abstract 1297O.
- Brahmer J, et al. Five-year follow-up from the CA209-003 study of nivolumab in previously treated advanced non-small cell lung cancer: clinical characteristics of long-term survivors. Oral presentation presented at: American Association for Cancer Research (AACR) Annual Meeting; April 1-5, 2017; Washington, DC, USA.

- Felip E, et al. Three-year follow-up from Checkmate 017/057: Nivolumab versus docetaxel in patients with previously treated advacned non-small cell lung cancer (NSCLC). Poster discussion presentation at the European Society of Medical Oncology Annual Meeting. 2017 Sep 8-12; Madrid, Spain. Poster 1301PD.
- Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (Version 1.1). Eur J Cancer 2009;45:228-47.



- Brooks RG. EuroQol: the current state of play. Health Policy 1996;37(1):53-72.
- Garland SN et al. Prospective Evaluation of the Reliability, Validity, and Minimally Important Difference of the Functional Assessment of Cancer Therapy-Gastric (FACT-Ga) Quality-of-Life Instrument. Cancer. 2011;117:1302–12.
- Darling G, Eton DT, Sulman J, et al. Validation of the Functional Assessment of Cancer Therapy Esophageal Cancer Subscale. Cancer 2006;107(4):854-63.

## 12 APPENDICES

Protocol Amendment No.: 06

Date: 13-Aug-2021 87

## APPENDIX 1 ABBREVIATIONS AND TRADEMARKS

| Term | Definition |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse event |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| AT | aminotransferase |
| BATTLE | Biomarker-integrated Approaches of Targeted Therapy for Lung cancer Elimination |
| BMS | Bristol-Myers Squibb Company |
| BOR | best overall response |
| BUN | blood urea nitrogen |
| CD | cluster of differentiation |
| CI | confidence interval |
| COVID-19 | coronavirus disease 2019 |
| CNS | central nervous system |
| CR | complete response |
| CrCl | creatinine clearance |
| CRF | case report form |
| CT | computed tomography |
| CTC | Common Terminology Criteria |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTLA-4 | cytotoxic T-lymphocyte antigen 4 |
| dMMR | mismatch repair deficient |
| DOR | duration of response |
| EC | esophageal cancer |
| ECG | electrocardiogram |

Protocol Amendment No.: 06

**ECOG** 

eCRF

Date: 13-Aug-2021

Eastern Cooperative Oncology Group

electronic case report form

| Term | Definition |
|---|---|
| ЕОТ | end of treatment |
| EQ-5D-3L | 3-level version of EQ-5D self-report questionnaire |
| FACT-Ga | Functional Assessment of Cancer Therapy-Gastric |
| FRACTION | Fast Real-time Assessment of Combination Therapy in Immuno-ONcology |
| FSH | follicle stimulating hormone |
| FU | follow-up |
| GaCS | Gastric Cancer Subscale |
| GC | gastric cancer |
| GEJ | gastroesophageal junction |
| GITR | glucocorticoid-induced tumor necrosis factor receptor-related |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HER2 | human epidermal growth factor receptor 2 |
| HIV | human immunodeficiency virus |
| HR | hazard ratio |
| IB | Investigator's Brochure |
| IEC | Independent Ethics Committee |
| IFNγ | interferon gamma |
| IHC | immunohistochemical/immunohistochemistry |
| IMP | investigational medicinal product |
| IO | immuno-oncology |
| IP | investigational product |
| IRB | Institutional Review Board |
| IRC | Independent Review Committee |
| IRT | Interactive Response Technology |
| LAG-3 | lymphocyte activation gene 3 |
| LDH | lactate dehydrogenase |

| Term | Definition |
|--------|-------------------------------------------------|
| MRI | magnetic resonance imaging |
| MSI-H | microsatellite instability-high |
| NCI | National Cancer Institute |
| NK | natural killer |
| NSCLC | non-small cell lung cancer |
| ORR | objective response rate |
| OS | overall survival |
| PD | progressive disease |
| PD-1 | programmed death-1 |
| p-DILI | potential drug-induced liver injury |
| PD-L1 | programmed death-ligand 1 |
| PD-L2 | programmed death-ligand 2 |
| PFS | progression-free survival |
| PFSR | progression-free survival rate |
| PID | patient identification number |
| PK | pharmacokinetic(s) |
| PR | partial response |
| prob | probability |
| PT | preferred term |
| QTcF | QT interval corrected with Fridericia's formula |
| Q2W | every 2 weeks |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | stable disease |
| SMB | Safety Monitoring Board |

| Term | Definition |
|--------|------------------------------------------------|
| SOC | system organ class |
| SUSAR | suspected, unexpected serious adverse reaction |
| Т3 | triiodothyronine |
| T4 | thyroxine |
| TNFRsf | tumor necrosis factor receptor super family |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| US | United States |
| VAS | visual analog scale |
| WOCBP | women of child-bearing potential |

#### APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS

The term 'Participant' is used in the protocol to refer to a person who has consented to participate in the clinical research study. The term 'Subject' used in the electronic case report form (eCRF) is intended to refer to a person (Participant) who has consented to participate in the clinical research study.

# REGULATORY AND ETHICAL CONSIDERATIONS GOOD CLINICAL PRACTICE

This study will be conducted in accordance with:

- Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines, Good Clinical Practice (GCP),
- as defined by the International Council on Harmonisation (ICH)
- in accordance with the ethical principles underlying European Union Directive 2001/20/EC
- United States Code of Federal Regulations, Title 21, Part 50 (21CFR50)
- applicable local requirements.

The study will be conducted in compliance with the protocol. The protocol and any amendments and the participant informed consent will receive approval/favorable opinion by Institutional Review Board/Independent Ethics Committee (IRB/IEC), and regulatory authorities according to applicable local regulations prior to initiation of the study.

All potential serious breaches must be reported to the Sponsor or designee immediately. A potential serious breach is defined as a Quality Issue (eg, protocol, deviation, etc) that is likely to affect, to a significant degree, one or more of the following: (1) the physical, safety or mental integrity of one or more subjects/participants; (2) the scientific value of the trial (eg, reliability and robustness of generated data). Items (1) or (2) can be associated with either GCP Regulation(s) or Trial protocol(s).)

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

## INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, consent form, participant recruitment materials (eg, advertisements), and any other written information to be provided to subjects/participants. The investigator or Bristol-Meyers Squibb (BMS) should also provide the IRB/IEC with a copy of the Investigator Brochure or product labeling information to be provided to subjects/participants and any updates.

Protocol Amendment No.: 06

The investigator, Sponsor or designee should provide the IRB/IEC with reports, updates and other information (eg, expedited safety reports, amendments, and administrative letters) according to regulatory requirements or institution procedures.

#### COMPLIANCE WITH THE PROTOCOL AND PROTOCOL REVISIONS

The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion of an amendment from the IRB/IEC (and if applicable, also by local health authority) except where necessary to eliminate an immediate hazard(s) to study subjects/participants.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining relevant approval/favorable opinion(s) the deviation or change will be submitted, as soon as possible to:

- IRB/IEC
- Regulatory Authority(ies), if applicable by local regulations (per national requirements)

Documentation of approval/favorable opinion signed by the chairperson or designee of the IRB(s)/IEC(s) and if applicable, also by local health authority must be sent to BMS.

If an amendment substantially alters the study design or increases the potential risk to the participant: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from subjects/participants currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new subjects/participants prior to enrollment.

If the revision is done via an administrative letter, investigators must inform their IRB(s)/IEC(s).

#### FINANCIAL DISCLOSURE

Investigators and sub-Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### **INFORMED CONSENT PROCESS**

Investigators must ensure that subjects/participants are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

In situations where consent cannot be given by subjects/participants, their legally acceptable representatives (as per country guidelines) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the participant volunteers to participate.

Protocol Amendment No.: 06

Sponsor or designee will provide the investigator with an appropriate (ie, Global or Local) sample informed consent form which will include all elements required by ICH, GCP, and applicable regulatory requirements. The sample informed consent form will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

#### Investigators must:

- Provide a copy of the consent form and written information about the study in the language in which the participant is most proficient prior to clinical study participation. The language must be non-technical and easily understood.
- Allow time necessary for participant or participant's legally acceptable representative to inquire about the details of the study.
- Obtain an informed consent signed and personally dated by the participant or the participant's legally acceptable representative and by the person who conducted the informed consent discussion.
- Obtain the IRB/IEC's written approval/favorable opinion of the written informed consent form and any other information to be provided to the subjects/participants, prior to the beginning of the study, and after any revisions are completed for new information.

If informed consent is initially given by a participant's legally acceptable representative or legal guardian, and the participant subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the participant.

Revise the informed consent whenever important new information becomes available that is relevant to the participant's consent. The investigator, or a person designated by the investigator, should fully inform the participant or the participant's legally acceptable representative or legal guardian, of all pertinent aspects of the study and of any new information relevant to the participant's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify subjects/participants must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the subjects'/participants' signed informed consent form and, in the United States, the subjects'/participants' signed Health Insurance Portability and Accountability Act Authorization.

The consent form must also include a statement that BMS and regulatory authorities have direct access to participant records.

The rights, safety, and well-being of the study subjects/participants are the most important considerations and should prevail over interests of science and society.

For the Fast Real-time Assessment of Combination Therapies in Immuno-ONcology (FRACTION) Program, participants should receive consent forms that include relevant information for all treatments to which they are eligible for enrollment; participants will not receive consent forms that include data relevant to agents within the FRACTION Program that are not within the Sub-Protocol for which they are screened. Informed consents to Sub-Protocols that

Protocol Amendment No.: 06

are closed, terminated early, or in any way no longer in effect will not be provided to new participants as an eligible treatment consent. Participants in any follow-up phase for a Sub-Protocol that is closed or terminated will receive pertinent updated safety and risk information if it becomes known. Participants in any follow-up phase may receive revised informed consent via mail and follow-up phone call by the investigator site.

### **SOURCE DOCUMENTS**

The Investigator is responsible for ensuring that the source data are accurate, legible, contemporaneous, original and attributable, whether the data are hand-written on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved, or transmitted electronically via computerized systems (and/or any other kind of electronic devices) as part of regulated clinical trial activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records (EMRs/EHRs), adverse event tracking/reporting, protocol required assessments, and/or drug accountability records).

When paper records from such systems are used in place of electronic format to perform regulated activities, such paper records should be certified copies. A certified copy consists of a copy of original information that has been verified, as indicated by a dated signature, as an exact copy having all of the same attributes and information as the original.

#### STUDY TREATMENT RECORDS

Records for study treatments (whether supplied by BMS, its vendors, or the site) must substantiate study treatment integrity and traceability from receipt, preparation, administration, and through destruction or return. Records must be made available for review at the request of BMS/designee or a Health Authority.

| If | Then |
|---|---|
| Supplied by BMS (or its vendors): | Records or logs must comply with applicable regulations and guidelines and should include: amount received and placed in storage area amount currently in storage area label identification number or batch number amount dispensed to and returned by each participant, including unique participant identifiers amount transferred to another area/site for dispensing or storage nonstudy disposition (eg, lost, wasted) amount destroyed at study site, if applicable amount returned to BMS retain samples for bioavailability/bioequivalence/biocomparability, if applicable dates and initials of person responsible for Investigational Product dispensing/accountability, as per the Delegation |
| Sourced by gite and not guardied by | of Authority Form. The investigator or designed against responsibility. |
| Sourced by site, and not supplied by BMS or its vendors (examples include IP sourced from the sites stock or commercial supply, or a specialty pharmacy) | The investigator or designee accepts responsibility for documenting traceability and study treatment integrity in accordance with requirements applicable under law and the standard operating procedures (SOPs)/standards of the sourcing pharmacy. |

BMS or designee will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

#### **CASE REPORT FORMS**

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for adverse events (AEs) and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the Sponsor or designee electronic data capture tool, electronic CRFs will be prepared for all data collection fields except for fields specific to serious adverse events (SAEs) and pregnancy, which will be reported on the electronic SAE form and Pregnancy Surveillance

Protocol Amendment No.: 06

Date: 13-Aug-2021 96

form, respectively. If electronic SAE form is not available, a paper SAE form can be used. Spaces may be left blank only in those circumstances permitted by study-specific CRF completion guidelines provided by Sponsor or designee.

The confidentiality of records that could identify subjects/participants must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF, SAE/pregnancy CRFs, must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a subinvestigator and who is delegated this task on the Delegation of Authority Form. Subinvestigators in Japan may not be delegated the CRF approval task. For electronic CRFs, review and approval/signature is completed electronically through the BMS electronic data capture tool. The investigator must retain a copy of the CRFs including records of the changes and corrections.

Each individual electronically signing electronic CRFs must meet Sponsor or designee training requirements and must only access the BMS electronic data capture tool using the unique user account provided by Sponsor or designee. User accounts are not to be shared or reassigned to other individuals.

#### MONITORING

Monitoring details describing strategy, including definition of study critical data items and processes (eg, risk-based initiatives in operations and quality such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the monitoring plan.

Representatives of BMS must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable. Certain CRF pages and/or electronic files may serve as the source documents.

In addition, the study may be evaluated by Sponsor or designee internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to Sponsor or designee.

#### RECORDS RETENTION

The investigator (or head of the study site in Japan) must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by BMS or designee, whichever is longer. The

Protocol Amendment No.: 06

Date: 13-Aug-2021 97

investigator (or head of the study site in Japan) must contact BMS prior to destroying any records associated with the study.

BMS or designee will notify the investigator (or head of the study site in Japan) when the study records are no longer needed.

If the investigator withdraws from the study (eg, relocation, retirement), the records shall be transferred to a mutually agreed upon designee (eg, another investigator, study site, IRB). Notice of such transfer will be given in writing to BMS or designee.

#### **RETURN OF STUDY TREATMENT**

For this study, study treatments (those supplied by BMS, a vendor or sourced by the investigator) such as partially used study treatment containers, vials and syringes may be destroyed on site.

| If | Then |
|---|---|
| Study treatments supplied by BMS (including its vendors) | Any unused study treatments supplied by BMS can only be destroyed after being inspected and reconciled by the responsible Study Monitor unless study treatments containers must be immediately destroyed as required for safety, or to meet local regulations (eg, cytotoxics or biologics). |
| | If study treatments will be returned, the return will be arranged by the responsible Study Monitor. |
| Study treatments sourced by site, not supplied<br>by BMS (or its vendors) (examples include<br>study treatments sourced from the sites stock<br>or commercial supply, or a specialty<br>pharmacy) | responsibility to dispose of all containers according to the institutional guidelines and |

It is the investigator's or designee's responsibility to arrange for disposal, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The following minimal standards must be met:

- On-site disposal practices must not expose humans to risks from the drug.
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances.
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's SOPs and a copy provided to BMS upon request.
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing the containers. The

method of disposal, i.e., incinerator, licensed sanitary landfill, or licensed waste disposal vendor must be documented.

• Accountability and disposal records are complete, up-to-date, and available for the Monitor to review throughout the clinical trial period.

It is the investigator's or designee's responsibility to arrange for disposal of all empty containers.

If conditions for destruction cannot be met the responsible Study Monitor will make arrangements for return of study treatments provided by BMS (or its vendors). Destruction of non-study treatments sourced by the site, not supplied by BMS, is solely the responsibility of the investigator or designee.

#### **DISSEMINATION OF CLINICAL STUDY DATA**

In order to benefit potential study participants, patients, healthcare providers and researchers, and to help BMS honor its commitments to study participants, BMS will make information about clinical research studies and a summary of their results available to the public as per regulatory and BMS requirements. BMS will post study information on local, national, or regional databases in compliance with national and international standards for disclosure. BMS may also voluntarily disclose information to applicable databases.

#### **CLINICAL STUDY REPORT**

A Signatory Investigator must be selected to sign the clinical study report.

For each CSR related to this protocol, the Signatory Investigator will be selected as appropriate based on the following criteria:

- Participant recruitment (eg, among the top quartile of enrollers)
- Involvement in trial design
- Other criteria (as determined by the study team)

#### SCIENTIFIC PUBLICATIONS

The data collected during this study are confidential and proprietary to Sponsor or designee. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the clinical trial agreement (CTAg) governing Study site or Investigator participation in the study. These requirements include, but are not limited to, submitting proposed publications to Sponsor or designee at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTAg.

Scientific Publications (such as abstracts, congress podium presentations and posters, and manuscripts) of the study results will be a collaborative effort between the study Sponsor and the external authors. No public presentation or publication of any interim results may be made by any

Protocol Amendment No.: 06

principal investigator, sub-investigator or any other member of the study staff without the prior written consent of the Sponsor.

Authorship of publications at BMS is aligned with the criteria of the International Committee of Medical Journal Editors (ICMJE, www.icmje.org). Authorship selection is based upon significant contributions to the study (ie, ICMJE criterion #1). Authors must meet all 4 ICMJE criteria for authorship:

- 1) Substantial intellectual contribution to the conception or design of the work; or the acquisition of data (ie, evaluable subjects with quality data), analysis, or interpretation of data for the work (eg, problem solving, advice, evaluation, insights and conclusion); AND
- 2) Drafting the work or revising it critically for important intellectual content; AND
- 3) Final approval of the version to be published; AND
- 4) Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

Those who make the most significant contributions, as defined above, will be considered by BMS for authorship of the primary publication. Sub-investigators will generally not be considered for authorship in the primary publication. Geographic representation will also be considered.

Authors will be listed by order of significant contributions (highest to lowest), with the exception of the last author. Authors in first and last position have provided the most significant contributions to the work.

For secondary analyses and related publications, author list and author order may vary from primary to reflect additional contributions.

#### **APPENDIX 3**

ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW UP AND REPORTINGADVERSE EVENTS

#### **Adverse Event Definition:**

An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.

## **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or results from other safety assessments (eg, ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator. Note that abnormal lab tests or other safety assessments should only be reported as AEs if the final diagnosis is not available. Once the final diagnosis is known, the reported term should be updated to be the diagnosis.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose, as a verbatim term (as reported by the investigator), should not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae and should specify "intentional overdose" as the verbatim term

#### **Events NOT Meeting the AE Definition**

- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).

#### **DEFINITION OF SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met.

Protocol Amendment No.: 06

#### SERIOUS ADVERSE EVENTS

Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:

Results in death

Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)

Requires inpatient hospitalization or causes prolongation of existing hospitalization (see NOTE below)

NOTE:

The following hospitalizations are not considered SAEs in BMS clinical studies:

- a visit to the emergency room or other hospital department < 24 hours, that does not result in admission (unless considered an important medical or life-threatening event)
- elective surgery, planned prior to signing consent
- admissions as per protocol for a planned medical/surgical procedure
- routine health assessment requiring admission for baseline/trending of health status (e.g., routine colonoscopy)
- medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases
- admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (e.g., lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason)
- admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols)

Results in persistent or significant disability/incapacity

Is a congenital anomaly/birth defect

Is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [e.g., medical, surgical] to prevent one of the other serious outcomes listed in the definition above.) Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.) Potential drug induced liver injury (DILI) is also considered an important medical event. (See Section 9.2.7 for the definition of potential DILI.)

Pregnancy and potential drug induced liver injury (DILI) must follow the same transmission timing and processes to BMS as used for SAEs (see section 9.2.5 for reporting pregnancies).

Protocol Amendment No.: 06

#### **EVALUATING AES AND SAES**

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to Sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to Sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send a SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of AEs and SAEs

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports must include the same investigator term(s) initially reported.)

If an ongoing SAE changes in its intensity or relationship to study treatment or if new information becomes available, the SAE report must be updated and submitted within 24 hours to BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs must be followed to resolution or stabilization.

#### REPORTING OF SAES TO SPONSOR OR DESIGNEE

- SAEs, whether related or not related to study treatment, and pregnancies must be reported to BMS (or designee) immediately within 24 hours of awareness of the event.
- SAEs must be recorded on the SAE Report Form.
  - The required method for SAE data reporting is through the eCRF.
  - The paper SAE Report Form is only intended as a back-up option when the electronic data capture (EDC) system is unavailable/not functioning for transmission of the eCRF to BMS (or designee).
    - ♦ In this case, the paper form is transmitted via email or confirmed facsimile (fax) transmission
    - When paper forms are used, the original paper forms are to remain on site
- Pregnancies must be recorded on a paper Pregnancy Surveillance Form and transmitted via email or confirmed facsimile (fax) transmission

SAE Email Address: Refer to Contact Information list.

SAE Facsimile Number: Refer to Contact Information list.

**SAE Telephone Contact** (required for SAE and pregnancy reporting): Refer to Contact Information list

## APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION

#### **DEFINITIONS**

#### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

## Women in the following categories are not considered WOCBP:

- Premenarchal
- Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

- Postmenopausal female
  - A postmenopausal state is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.

Note: Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The durations of the washout periods below are suggested guidelines and the investigators should use their judgement in checking serum FSH levels.

- 1 week minimum for vaginal hormonal products (rings, creams, gels)
- 4 week minimum for transdermal products
- 8 week minimum for oral products

Other parenteral products may require washout periods as long as 6 months. If the serum FSH level is > 40 mIU/mL at any time during the washout period, the woman can be considered postmenopausal.

Protocol Amendment No.: 06

#### **End of Relevant Systemic Exposure**

End of relevant systemic exposure is the time point where the Investigational Medicinal Product (IMP) or any active major metabolites has decreased to a concentration that is no longer considered to be relevant for human teratogenicity or fetotoxicity. This should be evaluated in context of safety margins from the no-observed adverse effect level or the time required for 5 half-lives of the IMP to pass.

## CONTRACEPTION GUIDANCE FOR FEMALE PARTICIPANTS OF CHILD BEARING POTENTIAL

One of the highly effective methods of contraception listed below is required during study duration and until the end of relevant systemic exposure, defined as approximately 5 half-lives after the end of study treatment, plus 30 days.

Local laws and regulations may require use of alternative and/or additional contraception methods.

## **Highly Effective Contraceptive Methods That Are User Dependent**

Failure rate of <1% per year when used consistently and correctly.<sup>a</sup>

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation and/or implantation (These methods of contraception cannot be used by WOCBP participants in studies where hormonal contraception is prohibited)<sup>b</sup>
  - oral (birth control pills)
  - intravaginal (vaginal birth control suppositories, rings, creams, gels)
  - transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - oral
  - injectable

#### **Highly Effective Methods That Are User Independent**

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation and/or implantation (This method of contraception cannot be used by WOCBP participants in studies where hormonal contraception is prohibited)<sup>b</sup>
- Intrauterine device (IUD)<sup>c</sup>
- Intrauterine hormone-releasing system (IUS) (This method of contraception cannot be used by WOCBP participants in studies where hormonal contraception is prohibited) <sup>b,c</sup>
- Bilateral tubal occlusion
- Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment.

Protocol Amendment No.: 06

The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- It is not necessary to use any other method of contraception when complete abstinence is elected.
- WOCBP participants who choose complete abstinence must continue to have pregnancy tests, as specified in Section 2.
- Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP participants chooses to forego complete abstinence

#### NOTES:

- <sup>a</sup> Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.
- Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. Hormonal contraception is permissible only when there is sufficient evidence that the IMP and other study medications will not alter hormonal exposures such that contraception would be ineffective or result in increased exposures that could be potentially hazardous. In this case, alternative methods of contraception should be utilized.
- <sup>c</sup> Intrauterine devices and intrauterine hormone releasing systems are acceptable methods of contraception in the absence of definitive drug interaction studies when hormone exposures from intrauterine devices do not alter contraception effectiveness

#### Less Than Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of >1% per year when used consistently and correctly.

- Male or female condom with or without spermicide. Male and female condoms cannot be used simultaneously
- Diaphragm with spermicide
- Cervical cap with spermicide
- Vaginal Sponge with spermicide
- Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mechanism of action (This method of contraception cannot be used by WOCBP participants in studies where hormonal contraception is prohibited)

## **Unacceptable Methods of Contraception**

- Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- Withdrawal(coitus interruptus).
- Spermicide only
- Lactation amenorrhea method (LAM)

## CONTRACEPTION GUIDANCE FOR MALE PARTICIPANTS WITH PARTNER(S) OF CHILD BEARING POTENTIAL

Male participants with female partners of childbearing potential are eligible to participate if they agree to the following during the treatment and until the end of relevant systemic exposure.

• Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.

Protocol Amendment No.: 06
- Male participants are required to use a condom for study duration and until the end of relevant systemic exposure defined as approximately 5 half-lives after the end of treatment plus an additional 90 days.
- Female partners of males participating in the study to consider use of effective methods of contraception until the end of relevant systemic exposure, defined as approximately 5 half-lives after the end of treatment plus an additional 90 days in the male participant.
- Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration during the treatment and until approximately 5 half-lives plus an additional 90 days after the end of treatment.
- Refrain from donating sperm for the duration of the study treatment and for approximately 5 half-lives plus an additional 90 days after the end of treatment.

#### **COLLECTION OF PREGNANCY INFORMATION**

Guidance for collection of Pregnancy Information and outcome of pregnancy on the Pregnancy Surveillance Form is provided in Section 9.2.5 and the Appendix for Adverse Events and Serious Adverse Events Definitions and procedures for Evaluating, Follow-up and Reporting.

#### APPENDIX 5 RECIST v1.1

# 1 ASSESSMENT OF OVERALL TUMOR BURDEN AND MEASURABLE DISEASE

To assess objective response or future progression, it is necessary to estimate the *overall tumor burden at baseline* and use this as a comparator for subsequent measurements. Measurable disease is defined by the presence of at least one measurable tumor lesion. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness.

At baseline, tumor lesions/lymph nodes will be categorized measurable or non-measurable as follows:

#### 1.1 Measurable lesions

Measurable lesions must be accurately measured in at least one dimension (longest diameter in the plane of the measurement to be recorded) with a minimum size of:

- 10 mm by CT/MRI scan (CT/MRI scan slice thickness no greater than 5 mm)
- 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable)
- 20 mm by chest x-ray
- *Malignant lymph nodes*: To be considered pathologically enlarged *and* measurable, a lymph node must be ≥15 mm in *short* axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the *short* axis will be measured and followed.

#### 1.2 Non-measurable lesions

- All other lesions, including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\ge 10$  to < 15 mm short axis), as well as truly non-measurable lesions.
- Lesions considered truly non-measurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that in not measurable by reproducible imaging techniques.

## 1.3 Special considerations regarding lesion measurability

#### 1.3.1 Bone lesions

- Bone scan, PET scan or plain films are *not* considered adequate imaging techniques to measure bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with *identifiable soft tissue components*, that can be evaluated by cross sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the *soft tissue component* meets the definition of measurability described above.
- Blastic bone lesions are non-measurable.

### 1.3.2 Cystic lesions

- Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.
- 'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same subject, these are preferred for selection as target lesions.

## 1.3.3 Lesions with prior local treatment

Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion.

#### 1.4 Specifications by methods of measurements

#### 1.4.1 Measurement of lesions

All measurements should be recorded in metric notation (mm). All baseline evaluations should be performed as close as possible to the treatment start and never more than 28 days before the beginning of the treatment.

#### 1.4.2 Method of assessment

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging based evaluation should always be done rather than clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam.

#### 1.4.2.1 CT/MRI scan

CT/MRI is the best currently available and reproducible method to measure lesions selected for response assessment. Measurability of lesions on CT/MRI scan is based on the assumption that CT/MRI slice thickness is 5 mm or less. When CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness.

## 1.4.2.2 Chest X-ray

Chest CT is preferred over chest X-ray, particularly when progression is an important endpoint, since CT is more sensitive than X-ray, particularly in identifying new lesions. However, lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

#### 1.4.2.3 Clinical lesions

Clinical lesions will only be considered measurable when they are superficial and  $\geq 10$  mm diameter as assessed using calipers. For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is suggested. As previously noted, when lesions can be evaluated by both clinical exam and imaging, imaging evaluation should be undertaken since it is more objective and may also be reviewed at the end of the study.

Protocol Amendment No.: 06

#### 1.4.2.4 Ultrasound

Ultrasound is *not* useful in assessment of lesion size and should not be used as a method of measurement. If new lesions are identified by ultrasound in the course of the study, confirmation by CT or MRI is advised.

### 1.4.2.5 Endoscopy, laparoscopy

The utilization of these techniques for objective tumor evaluation is *not* advised.

#### 1.4.2.6 Tumor markers

Tumor markers *alone* cannot be used to assess objective tumor response.

# 2 BASELINE DOCUMENTATION OF 'TARGET' AND 'NON-TARGET' LESIONS

#### 2.1 Target lesions

When more than one measurable lesion is present at baseline all lesions up to a maximum of 5 lesions total (and a maximum of 2 lesions per organ) representative of all involved organs should be identified as *target lesions* and will be recorded and measured at baseline.

Target lesions should be selected on the basis of their **size** (lesions with the longest diameter), be representative of all involved organs, and should lend themselves to *reproducible repeated measurements*.

A *sum of the diameters* (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the *baseline sum diameters*. If lymph nodes are to be included in the sum, then as noted below, only the *short* axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the disease.

#### 2.1.1 Lymph nodes

**Lymph nodes** merit special mention since they are normal anatomical structures which may be visible by imaging even if not involved by tumor. Pathological nodes which are defined as measurable and may be identified as target lesions must meet the criterion of a **short axis of** ≥15 mm by CT scan. Only the *short* axis of these nodes will contribute to the baseline sum. Nodes that have a short axis <10 mm are considered non-pathological and should not be recorded or followed.

### 2.2 Non-target lesions

All other lesions (or sites of disease) including pathological lymph nodes should be identified as *non-target lesions* and should also be recorded at baseline. Measurements are not required and these lesions should be followed as 'present', 'absent', or in rare cases 'unequivocal progression'. In addition, it is possible to record multiple non-target lesions involving the same organ as a single item on the case record form (e.g. 'multiple enlarged pelvic lymph nodes' or 'multiple liver metastases').

#### 3 TUMOR RESPONSE EVALUATION

#### 3.1 Evaluation of target lesions

<u>Complete Response (CR)</u>: **Disappearance of all target lesions.** Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

<u>Partial Response (PR)</u>: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

<u>Progressive Disease (PD):</u> At least a **20% increase in the sum of diameters of target lesions, taking as reference the** *smallest sum on study* **(this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an <b>absolute increase of at least 5 mm**. (*Note:* the appearance of one or more new lesions is also considered progression).

<u>Stable Disease (SD):</u> Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

## 3.1.1 Special notes on the assessment of target lesions

### **3.1.1.1** Lymph nodes

Lymph nodes identified as target lesions should always have the actual short axis measurement recorded and should be measured in the same anatomical plane as the baseline examination, even if the nodes regress to below 10 mm on study. This means that when lymph nodes are included as target lesions, the 'sum' of lesions may not be zero even if complete response criteria are met, since a normal lymph node is defined as having a short axis of < 10 mm.

## 3.1.1.2 Target lesions that become 'too small to measure'

All lesions (nodal and non-nodal) recorded at baseline should have their actual measurements recorded at each subsequent evaluation, even when very small (e.g. 2 mm). If the radiologist is able to provide an actual measurement, that should be recorded, even if it is below 5 mm.

However, when such a lesion becomes difficult to assign an exact measure to then:

- if it is the opinion of the radiologist that the lesion has likely disappeared, the measurement should be recorded as 0 mm.
- if the lesion is believed to be present and is faintly seen but too small to measure, a default value of 5 mm should be assigned (note: in case of a lymph node believed to be present and faintly seen but too small to measure, a default value of 5 mm should be assigned in this circumstance as well). This default value is derived from the 5 mm CT slice thickness (but should not be changed with varying CT slice thickness).

## 3.1.1.3 Target lesions that split or coalesce on treatment

- When non-nodal lesions 'fragment', the longest diameters of the fragmented portions should be added together to calculate the target lesion sum.
- As lesions coalesce, a plane between them may be maintained that would aid in obtaining maximal diameter measurements of each individual lesion. If the lesions have truly coalesced

such that they are no longer separable, the vector of the longest diameter in this instance should be the maximal longest diameter for the 'coalesced lesion'.

## 3.2 Evaluation of non-target lesions

While some non-target lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol.

<u>Complete Response (CR):</u> Disappearance of all non-target lesions. All lymph nodes must be non-pathological in size (<10 mm short axis).

Non-CR/Non-PD: Persistence of one or more non-target lesion(s) above the normal limits.

<u>Progressive Disease (PD):</u> *Unequivocal progression* of existing non-target lesions. (*Note:* the appearance of one or more new lesions is also considered progression).

### 3.2.1 Special notes on assessment of non-target lesions

The concept of progression of non-target disease requires additional explanation as follows:

## 3.2.1.1 When the subject also has measurable disease

- To achieve 'unequivocal progression' on the basis of the non-target disease, there must be an overall level of substantial worsening in non-target disease such that, even in presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy.
- A modest 'increase' in the size of one or more non-target lesions is usually not sufficient to quality for unequivocal progression status.

## 3.2.1.2 When the subject has only non-measurable disease

- To achieve 'unequivocal progression' on the basis of the non-target disease, there must be an overall level of substantial worsening such that the overall tumor burden has increased sufficiently to merit discontinuation of therapy.
- A modest 'increase' in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status.
- Because worsening in non-target disease cannot be easily quantified (by definition: if all lesions are non-measurable) a useful test that can be applied when assessing subjects for unequivocal progression is to consider if the increase in overall disease burden based on the change in non-measurable disease is comparable in magnitude to the increase that would be required to declare PD for measurable disease: i.e. an increase in tumor burden representing an additional 73% increase in 'volume' (which is equivalent to a 20% increase diameter in a measurable lesion). Examples include an increase in a pleural effusion from 'trace' to 'large', an increase in lymphangitic disease from localized to widespread, or may be described in protocols as 'sufficient to require a change in therapy'.
- If 'unequivocal progression' is seen, the subject should be considered to have had overall PD at that point.

Protocol Amendment No.: 06

#### 3.2.1.3 Tumor markers

Tumor markers *alone* cannot be used to assess objective tumor responses. If markers are initially above the upper normal limit, however, they must normalize in order for a subject to be considered as having attained a complete response.

#### 3.3 New lesions

The appearance of new malignant lesions denotes disease progression. The finding of a new lesion should be unequivocal: i.e. not attributable to differences in scanning technique, change in imaging modality or findings thought to represent something other than tumor (for example, some 'new' bone lesions may be simply healing or flare of pre-existing lesions). This is particularly important when the subject's baseline lesions show partial or complete response. For example, necrosis of a liver lesion may be reported on a CT scan report as a 'new' cystic lesion, which it is not.

A lesion identified on a follow-up study in an anatomical location that was *not* scanned at baseline is considered a new lesion and will indicate disease progression. An example of this is the subject who has visceral disease at baseline and while on study has a CT or MRI brain scan ordered which reveals metastases. The subject's brain metastases are considered to be evidence of PD even if he/she did not have brain imaging at baseline.

If a new lesion is equivocal, for example because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. *If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.* 

### 3.3.1 FDG-PET evaluation

While FDG-PET response assessments need additional study, it is sometimes reasonable to incorporate the use of the qualitative assessment of FDG-PET scanning to complement CT scanning in assessment of progression (particularly possible 'new' disease). New lesions on the basis of FDG-PET imaging can be identified according to the following algorithm:

- Negative FDG-PET at baseline, with a positive FDG-PET at follow-up is a sign of PD based on a new lesion.
- No FDG-PET at baseline and a positive FDG-PET at follow-up:
  - If the positive FDG-PET at follow-up corresponds to a new site of disease confirmed by CT, this is PD.
  - If the positive FDG-PET at follow-up is not confirmed as a new site of disease on CT, additional follow-up CT scans are needed to determine if there is truly progression occurring at that site (if so, the date of PD will be the date of the initial positive FDG-PET scan).
  - If the positive FDG-PET at follow-up corresponds to a pre-existing site of disease on CT that is not progressing on the basis of the anatomic images, this is not PD.

#### 4 RESPONSE CRITERIA

#### 4.1 Time point response

A response assessment should occur at each time point specified in the protocol.

For subjects who have **measurable disease** at baseline <u>Table 1</u> provides a summary of the overall response status calculation at each time point.

Table 1. Time point response: subjects with target (+/- non-target) disease.

| Target lesions | Non-target lesions | New lesions | Overall response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, NE =not evaluable.

## 4.1.1 Missing assessments and not evaluable designation

When no imaging/measurement is done at all at a particular time point, the subject is **not evaluable** (NE) at that time point. If only a subset of lesion measurements are made at an assessment, the case is also considered NE at that time point, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not have changed the assigned time point response.

#### 4.1.2 Confirmation scans

• Verification of Response: Confirmation of PR and CR is required at least 4 weeks later to ensure responses identified are not the result of measurement error. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by consecutive repeat assessments that should be performed no less than 28 days after the criteria for response are first met. For this study, the next scheduled tumor assessment can meet this requirement.

## 4.2 Best overall response: All timepoints

The *best overall response* is determined once all the data for the subject is known. It is the best response recorded from the start of the study treatment until the objectively documented progression per RECIST v1.1 or subsequent anticancer therapy, whichever occurs first (taking into

Protocol Amendment No.: 06

account any requirement for confirmation). The subject's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions.

Best response is defined as the best response across all time points with subsequent confirmation. Complete or partial responses may be claimed only if the criteria for each are met at a subsequent time point as specified in the protocol (generally 4 weeks later).

In this circumstance, the best overall response can be interpreted as specified in <u>Table 2</u>. When SD is believed to be best response, it must meet the protocol specified minimum time from baseline. Measurements must have met the SD criteria at least once after study entry at a minimum interval (in general not less than 6 weeks).

| Table 2. Best overall response when confirmation of CR and PR <i>IS</i> required | | |
|---|---|---|
| Overall response | Overall response | BEST overall response |
| First time point | Subsequent time point | |
| CR | CR | CR |
| CR | PR | SD, PD or PR <sup>a</sup> |
| CR | SD | SD provided minimum criteria for SD duration met, otherwise, PD |
| CR | PD | SD provided minimum criteria for SD duration met, otherwise, PD |
| CR | NE | SD provided minimum criteria for SD duration met, otherwise NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD provided minimum criteria for SD duration met, otherwise, PD |
| PR | NE | SD provided minimum criteria for SD duration met, otherwise NE |
| NE | NE | NE |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, NE = not evaluable.

Protocol Amendment No.: 06 Date: 13-Aug-2021

<sup>&</sup>lt;sup>a</sup> If a CR is truly met at first time point, then any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, makes the disease PD at that point (since disease must have reappeared after CR). Best response would depend on whether minimum duration for SD was met. However, sometimes 'CR' may be claimed

when subsequent scans suggest small lesions were likely still present and in fact the subject had PR, not CR at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

### 4.3 Duration of response

## 4.3.1 Duration of overall response

The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).

The duration of overall complete response is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

#### 4.3.2 Duration of stable disease

Stable disease is measured from the start of the treatment (in randomized trials, from date of randomization) until the criteria for progression are met, taking as reference the smallest sum on study (if the baseline sum is the smallest, this is the reference for calculation of PD).

Protocol Amendment No.: 06

#### APPENDIX 6 NIVOLUMAB MANAGEMENT ALGORITHMS

These general guidelines constitute guidance to the Investigator and may be supplemented by discussions with the Medical Monitor representing the Sponsor. The guidance applies to all immuno-oncology agents and regimens.

A general principle is that differential diagnoses should be diligently evaluated according to standard medical practice. Non-inflammatory etiologies should be considered and appropriately treated.

Corticosteroids are a primary therapy for immuno-oncology drug-related adverse events. The oral equivalent of the recommended IV doses may be considered for ambulatory patients with low-grade toxicity. The lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

Consultation with a medical or surgical specialist, especially prior to an invasive diagnostic or therapeutic procedure, is recommended.

The frequency and severity of the related adverse events covered by these algorithms will depend on the immuno-oncology agent or regimen being used. The frequency and severity of the related adverse events covered by these algorithms will depend on the immuno-oncology agent or regimen being used.

## **GI Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause is identified, treat accordingly and continue I-O therapy. Opiates/narcotics may mask symptoms of perforation. Infliximab should not be used in cases of perforation or sepsis.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

27-Jun-2019

Protocol Amendment No.: 06

## Renal Adverse Event Management Algorithm

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

930104678 8.0

27-Jun-2019

Protocol Amendment No.: 06 Date: 13-Aug-2021

Approved v8.0

## **Pulmonary Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy. Evaluate with imaging and pulmonary consultation.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids

27-Jun-2019

Protocol Amendment No.: 06

## **Hepatic Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy. Consider imaging for obstruction.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

27-Jun-2019

Protocol Amendment No.: 06 Date: 13-Aug-2021

Approved v8.0 930104678 8.0

<sup>\*</sup>The recommended starting dose for grade 4 hepatitis is 2 mg/kg/day methylprednisolone IV.

## **Endocrinopathy Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy. Consider visual field testing, endocrinology consultation, and imaging.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

27-Jun-2019

Protocol Amendment No.: 06

## **Skin Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

Alf SJS/TEN is suspected, withhold I-O therapy and refer patient for specialized care for assessment and treatment. If SJS or TEN is diagnosed, permanently discontinue I-O therapy.

27-Jun-2019

Protocol Amendment No.: 06

<sup>\*</sup>Refer to NCI CTCAE v4 for term-specific grading criteria.

## **Neurological Adverse Event Management Algorithm**

Rule out non-inflammatory causes. If non-inflammatory cause, treat accordingly and continue I-O therapy.



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (e.g. prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

27-Jun-2019

Protocol Amendment No.: 06 Date: 13-Aug-2021

Approved v8.0 930104678 8.0

## **Myocarditis Adverse Event Management Algorithm**



Patients on IV steroids may be switched to an equivalent dose of oral corticosteroids (eg, prednisone) at start of tapering or earlier, once sustained clinical improvement is observed. Lower bioavailability of oral corticosteroids should be taken into account when switching to the equivalent dose of oral corticosteroids.

Prophylactic antibiotics should be considered in the setting of ongoing immunosuppression.

ATG = anti-thymocyte globulin; BNP = B-type natriuretic peptide; ECG = electrocardiogram; IV = intravenous; MRI = magnetic resonance imaging

27-Jun-2019

Protocol Amendment No.: 06

## APPENDIX 7 ECOG PERFORMANCE STATUS

| STATUS | SCALES | | STATUS |
|---|---|---|---|
| | KARNOFSKY | ZUBROD-ECOG-<br>WHO | |
| Normal, no complaints | 100 | 0 | Normal activity |
| Able to carry on normal activities Minor signs or symptoms of disease | 90 | 1 | Symptoms, but fully ambulatory |
| Normal activity with effort | 80 | | |
| Cares for self. Unable to carry on normal activity or to do active work | 70 | 2 | Symptomatic, but in bed < 50% of the day. |
| Requires occasional assistance,<br>but able to care for most of his<br>needs | 60 | | |
| Requires considerable assistance and frequent medical care | 50 | 3 | Needs to be in bed > 50% of the day, but not bedridden |
| Disabled. Requires special care and assistance | 40 | | |
| Severely disabled. Hospitalization indicated though death non imminent | 30 | 4 | Unable to get out of bed |
| Very sick. Hospitalization necessary. Active supportive treatment necessary | 20 | | |
| Moribund | 10 | | |
| Dead | 0 | 5 | Dead |

From: Minna JD, Higgins GA and Glatstein EJ. Cancer of the lung. In: DeVita V, Hellman S, Rosenberg S (Eds.). Cancer: Principles and Practice of Oncology, Lippincott, Philadelphia, 1984, p. 536.

## APPENDIX 8 COUNTRY SPECIFIC REQUIREMENTS

# <u>Countries: Germany, et al. Where Exclusion of HIV Positive Participants Is Locally Mandated</u>

| | Country-specific language |
|---|---|
| Section 2 Flow Chart/Time<br>and Events Schedule, Table 2-<br>1: Screening Assessments-<br>Laboratory Tests | Add "HIV" to the list of laboratory tests |
| Section 6.2 Exclusion Criteria, Exclusion criterion p, i)a | "Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)"to be replaced with "Positive test for HIV". |

## APPENDIX 9 REVISED PROTOCOL SUMMARY OF CHANGE HISTORY

## Overall Rationale for the Revised Protocol 05, 13-Sep-2019

The FRACTION-Gastric Cancer Master Protocol (CA018003) was updated to include the myocarditis adverse event management algorithm in Appendix 6: Nivolumab Management Algorithms.

| Section Number<br>& Title | Description of Change | Brief Rationale |
|---|---|---|
| Title Page | Medical Monitor/Study Director information was updated | Administrative information was updated. |
| Synopsis | The synopsis was updated to align with the protocol changes. | The synopsis was updated to align with the protocol changes. |
| Section 2 Schedule of<br>Activities Table 2-3<br>Follow-up Procedural<br>Outline | The Note associated with Procedure Patient-reported Outcomes Assessment was updated to include the use of the Esophagus Cancer Subscale. | - |
| Section 4 Objectives<br>and Endpoints Table<br>4-1 Objectives and | Exploratory objective "To evaluate disease-related symptom improvement, as measured by the GaCS of the FACT-Ga in treated participants" was updated to include ECS of the FACT-E. | With the addition of participants with esophageal cancer, the Esophagus Cancer |
| Endpoints | The corresponding endpoint was updated to include ECS scores. | Subscale (ECS) from the Functional Assessment of |
| Section 9.9.1 Patient-reported Outcomes | This section was updated to include Esophagus Cancer Subscale (ECS) from the Functional Assessment of Cancer Therapy-Esophageal (FACT-E). A description of when each assessment is used, was added. A description of the FACT-E assessment was added. | Cancer Therapy-<br>Esophageal (FACT-E)<br>patient-reported outcome<br>assessment was added |
| Section 10.3.3.4<br>Outcomes Research<br>Analyses | ECS scores were added to the endpoint "Summary measures of EQ-5D-3L index and VAS scores and GaCS with corresponding change from baseline for each score." | |
| Section 5.2 Number of<br>Participants | A clarification was made that the number of participants is appropriate for Sub-Protocols using a Simon-2 stage (optimal) design. For Sub-Protocols not utilizing a Simon-2 stage design, a different sample size may be used depending on the statistical considerations for those treatment combinations. In those cases, sample size will be discussed within the individual Sub-Protocols. | This information was updated to provide clarification. |
| Section 5.4.1<br>Rationale for Duration<br>of Therapy | The following statement was removed: "Therefore, in FRACTION-Gastric Cancer Sub-Protocol A, treatment with BMS-986217 and nivolumab will be extended for up to 2 years." | This statement was removed because this Master Protocol is not specific to Sub-protocol A. |

Protocol Amendment No.: 06

| SUMMARY OF KEY CHANGES FOR REVISED PROTOCOL 05 | | |
|---|---|---|
| Section Number<br>& Title | Description of Change | Brief Rationale |
| Appendix 6 | Nivolumab Management Algorithms were updated to include the myocarditis adverse event management algorithm. | BMS has updated the management algorithms associated with nivolumab. These new algorithms replace the previous algorithms. |
| All | Typographical errors corrected. | Minor, therefore have not been summarized. |

## Overall Rationale for the Revised Protocol 04, 03-May-2019

The FRACTION-Gastric Master Protocol was revised to add information about the approval of pembrolizumab for the treatment of patients with MSI-H/dMMR cancers with no satisfactory alternative treatment options. It was also updated to clarify pretreatment tumor biopsy collection timing and assessment of adequacy.

| Summary of Key Changes of Revised Protocol 04 | | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| Section 2 Schedule of<br>Activities,<br>Table 2-1 Screening<br>Procedural Outline | In the note associated with "Mandatory Pretreatment Tumor Biopsy," collection timing was updated from "prior to first dose of study treatment" to "prior to randomization." It was clarified that the adequacy of the tumor tissue must be confirmed by the central laboratory prior to randomization. | Collection timing and assessment of pretreatment tumor biopsies was updated to clarify the information for study sites. |
| Section 3.2.1<br>FRACTION-Gastric<br>Cancer | An update was made to indicate that pembrolizumab is an Anti-PD-1 antibody. The following information was also added: "pembrolizumab is also approved (accelerated approval) for the treatment of patients with MSI-H/dMMR cancers with no satisfactory alternative treatment options." | This update was made to explicitly describe anti-PD-1 as an SOC option for MSI-H cancers in lack of satisfactory treatment alternatives. |
| Section 5.1.3.1 Screening | The sentence "Fresh biopsy must be confirmed received by the central lab before randomization" (per Administrative Letter 02) was removed and replaced with "An adequate baseline tumor biopsy (as determined by a central laboratory pathologist) must be obtained prior to randomization." | Tissue quality is critical for<br>biomarker analysis. Local<br>laboratory confirmation has led<br>to inconsistent tissue quality<br>and missing biomarker data. |
| Section 6.1 Inclusion<br>Criteria | Inclusion Criteria 2) e) i) 5) and Inclusion Criteria 2) e) ii) 5) were updated: The sentences "Fresh biopsy must be confirmed received by central lab before randomization. The biopsy sample must meet the minimum quality requirements and H&E assessment is to be performed primarily at the central laboratory." were removed and replaced with "An adequate baseline tumor biopsy as determined by a central laboratory pathologist must be obtained prior to randomization." | Assessment of pretreatment tumor biopsies was updated to clarify the information for study sites. |
| Section 6.1 Inclusion<br>Criteria | Inclusion Criteria 2) j) ii) and Inclusion Criteria 2) o) ii) were updated to remove the option to have a local pathologist assess the adequacy of the biopsy tissue quantity and quality. | Tissue quality is critical for biomarker analysis. Local laboratory confirmation has led to inconsistent tissue quality and missing biomarker data. |
| Section 6.2 Exclusion<br>Criteria | The following information in bold was added to exclusion criteria 3) a): "Under certain specific circumstances, and only in countries where local regulations permit, a person who has been imprisoned may be included or permitted to continue as a participant. | This update was made to align with the BMS protocol model document standards. |
| Section 7.7.3 Permitted<br>Therapy | Language was updated to indicate that vaccines containing live/attenuated virus are not permitted while on study treatment and until 100 days after | This update was made to align with the program-wide standard for nivolumab. |

Protocol Amendment No.: 06

| Summary of Key Changes of Revised Protocol 04 | | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| | the last dose. The option to discuss the use of live vaccines with the BMS medical monitor (or designee) was removed. | |
| Section 8.1 Discontinuation from Study Treatment | The following note was added to the description of participants who are imprisoned or involuntarily incarcerated: "Under specific circumstances and only in countries where local regulations permit, a participant who has been imprisoned may be permitted to continue as a participant. Strict conditions apply and BMS approval is required." | This update was made to align with the current version of the BMS Protocol Model Document. |
| Appendix 02: Study<br>Governance<br>Considerations | Language was updated to indicate that "subject" also refers to "participant." The definition of serious breach was updated. A section describing "scientific publications" was added. Additional minor clarifications were made. | Updates were made to align with the current version of the BMS Protocol Model Document. |

## Overall Rationale for the Revised Protocol 03, 05-Feb-2019

The FRACTION-Gastric Master Protocol was revised to expand indication to esophageal cancer based on the results of CheckMate-032 clinical study. Added clarification on timing and eligibility for efficacy assessment scans at FU1 and FU3.

Sections in synopsis have been updated to align with the protocol section changes listed below.

| Summary of Key Changes of Revised Protocol 03 | | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| Section 2, Schedule of Activities; Table 2-1: Screening Procedural Outline; Table 2-2: Baseline for Re-randomization Procedural Outline | In Table 2-1, Notes for Utilize IRT were modified and time to randomization is now up to 7 days. In Table 2-1 and Table 2-2, 12-lead ECG Notes now reads as: ECGs should be recorded after the participant has been supine for at least 5 minutes. Record QTcF. If ECG abnormality is noted, a repeat ECG must be performed. | Compliance with current IRT manual. The bolded phrase was added at the end. The requirement to perform and evaluate ECG was further reinforced with the need to perform repeat ECG in case of abnormal findings. |
| Section 2, Schedule of<br>Activities; Table 2-3:<br>Follow-up Procedural<br>Outline;<br>Section 9.1 Efficacy<br>Assessments | In Table 2-3, Tumor Response Assessment Notes now reads as: All participants should receive scans at FU1 except for participants who started subsequent therapy or participants with PD who have already been treated beyond progression. Scans at FU3 and every 12 weeks (±14 days) will only be collected for participants with CR, PR, SD, or NE at treatment discontinuation. Section 9.1 now includes same language for consistency with Table 2-3. | Clarification on timing and eligibility for scans at FU1 and FU3 |
| Section 3.2 Background;<br>Section 4 Objectives and<br>Endpoints, Table 4-1:<br>Objectives and Endpoints;<br>Section 11 References | Background and Table 4-1 were revised to include esophageal cancer (EC). New references are added to support EC indication. | Revised to expand indication to EC based on the results of CheckMate-032 clinical study that demonstrated clinical efficacy of nivolumab + ipilimumab combination in esophagogastric cancers. |
| Section 6.1 Inclusion Criteria; 2) Type of Participant and Target Disease Characteristics | Criteria 2) a) modified to be read as: All participants must have inoperable, advanced, or metastatic EC, GC or GEJ carcinoma and have histologically confirmed predominant adenocarcinoma and/or squamous carcinoma. | Criteria has been modified and revised to expand indication to EC |

Protocol Amendment No.: 06

| Summary of Key Cha | Summary of Key Changes of Revised Protocol 03 | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| | Criteria 2) e) i) (5) and Criteria 2) e) ii) (4) has been updated to be read as: All subjects must consent to the acquisition of fresh pre- and on-treatment tumor biopsies for performance of correlative biomarker studies. Archival specimens may not be substituted for fresh baseline specimens but can be submitted to help understand the evolution of the tumor (ie, PD-L1 expression changes over time) for performance of correlative studies. Subjects who either do not consent to a pre-treatment tumor biopsy or do not have accessible lesions are not eligible. Fresh biopsy must be confirmed received by central lab before randomization. The biopsy sample must meet the minimum quality requirements and H&E assessment is to be performed primarily at the central laboratory. If fresh biopsy is not clinically feasible or safe, the option of archival tissue can be discussed with BMS if the biopsy was obtained within 90 days of study enrollment and there was no intervening systemic anticancer or IO therapy. | Biopsy requirements has been updated in order to: 1. To reflect PD-L1 testing is no longer a stratification factor and PD-L1 results are therefore not relevant in screening phase 2. Ensuring tissue quality remains crucial, and this was clarified 3. Option of using archival tissue was introduced with specific requirements to allow optimal correlative analyses |
| Section 6.1 Inclusion<br>Criteria, 3) Age and<br>Reproductive Status; | Criteria 3) e) and Section 9.2.5 has been modified to add the text to address fetal protection. | Required by POL-009087<br>(Women Of Child Bearing<br>Potential and Clinical Trials |
| Section 9.2.5 Pregnancy | to add the text to address fetal protection. | Policy) |
| Section 6.1 Inclusion<br>Criteria, Criteria 2) j) and<br>Criteria 3) e) i) | These criteria are not applicable after the implementation of this revised protocol and "Not applicable as per revised protocol 03" has been added in the front of both criterias. | Criteria 2) j) has been revised for tumor biopsy and is now added as a new criteria 2) o). Criteria 3) e) i) is not applicable since there is no fetal tox information available and it is required for azoospermic males to follow contraception guidelines. |
| Section 7.7.1 Prohibited and/or Restricted Treatments | Added to 4th bullet that use of marijuana and its derivatives are permitted for treatment of symptoms related to cancer treatment. | Marijuana has become legalized in many geographic regions and is increasingly being used for cancer patients. Multiple institutions have requested the use of marijuana |

Protocol Amendment No.: 06

| Summary of Key Changes of Revised Protocol 03 | | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| | | in the protocol as patients are legally utilizing marijuana for multiple purposes, including but not limited to pain, poor/loss of appetite, anxiety, anorexia, and nausea. |
| Section 9.1 Efficacy<br>Assessments | Added "As participant's response to prior therapy is an important part of medical history, additional details regarding the previous therapy, including but not limited to best response to therapy, timing of progression on prior therapy, method of how the progression was measured, existence of confirmation scan to document progression and detailed information such as other clinical evidence (eg, increased pain requiring palliative radiotherapy) to support progression, response/progression dates, and reason for discontinuation will be collected in this trial." | Addition of collection of details of progressive disease in relation to participant's prior therapy. |
| | Text under third paragraph was modified regarding brain metastasis and clarification was added. | Text has been modified to add clarification that participants with a history of brain metastasis or symptoms should have a surveillance MRI study per standard care. |
| Section 9.3 Overdose | Last statement was updated | Modified text to be consistent with revised language in Appendix 3. |
| Appendix 3 Adverse Events and Serious Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting; Appendix 4 Contraception Guidance for Female Participants of Child Bearing Potential; Appendix 6 Management Algorithms | Mentioned appendices have been updated | Modifications have been made to align with the most current protocol appendix model document |
| All | Minor rewording/re-formatting for clarification. | For clarity and consistency within the document. |

Protocol Amendment No.: 06

## Overall Rationale for the Revised Protocol 02, 14-Dec-2017

The FRACTION-Gastric Master Protocol was revised to allow participants with complete response, partial response, or stable disease to continue treatment for up to a total duration of 2 years. Additionally, PD-L1 status was removed as a stratification factor.

| Summary of key changes of Revised Protocol 02 | | |
|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 2, Schedule of Activities; Table 2-2, Baseline for Re-randomization Procedural Outline; Section 3.1.1.2, Specific Attributes of the FRACTION Program Design; Section 5.1, Overall Design; Section 5.1.1, FRACTION-Gastric Cancer Tracks 1 and 2 Design; Figure 5.1.1-1, Tracks 1 and 2 Study Design Schematic; Section 5.1.3.2, Treatment; Section 5.1.3.3, Follow-up; Section 5.4.1, Rationale for Duration of Therapy | Participants will receive treatment of up to 2 years total duration. | Emerging data suggest that patients may derive clinical benefit beyond 6 months of immunotherapy. Therefore, patients will continue on study treatment for up to 2 years and re-treatment is not permitted. |
| Table 2-1, Screening Procedural Outline;<br>Section 5.1.3.1, Screening; Section 6.1,<br>Inclusion Criteria "2.e.i.5" and "2.e.ii.1"; | Changes made to reflect<br>that PD-L1 status will no<br>longer be a stratification<br>factor, and therefore,<br>results will no longer be<br>needed before<br>randomization | Expression of PD-L1 on tumor is not required for clinical benefit based on a randomized clinical trial in gastric cancer (ATTRACTION 2). Therefore, PD-L1 will not be used as a stratification factor. |
| Table 2-1, Screening Procedural Outline | Duration of randomization prior to first dose extended Data to be collected on toxicities from treatment with prior immunotherapies | 1. To allow patients to complete all the post-randomization procedures required for a sub-protocol, duration between randomization and start of treatment can be extended to allow for completion of study-related tests. 2. For patients previously treated with PD-1/PD-L1/CTLA-4, enrolling directly into Track 2, we will collect additional data on details of adverse events with prior immunotherapies. |
| Section 10.1.1, Track 1 - Anti-PD-1, Anti-PD-L1, and Anti-CTLA-4 Treatment-naïve Participants; Section 10.1.2, Track 2 - Anti-PD-1, Anti-PD-L1, and Anti-CTLA-4 Treatment-experienced Participants; | Number of participants<br>updated | Updated based on removal of prospective stratification of PD-L1 |
| Table 2-3, Follow-up Procedural Outline | ECOG Performance<br>Status assessment added<br>at Follow-up visits 2 and<br>3 | Collect performance status during follow-up. |

Protocol Amendment No.: 06

| Summary of key changes of Revised Protocol 02 | | |
|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 3.1, Study Rationale; Section 3.1.1.1,<br>Rationale for the FRACTION Program;<br>Section 3.2.1, FRACTION-Gastric Cancer | Included updates from recent clinical studies | |
| Throughout | Minor rewording/re-<br>formatting for<br>clarification | |